

# Clinical Trial of the Edwards Aortic Bioprosthesis, Model 11000

NCT01651052

May 8, 2012



# Clinical Trial of the Edwards Pericardial Aortic Bioprosthesis, Model 11000

# CLINICAL PROTOCOL (Clinical Investigational Plan)

Clinical Trial Number: 2010-03 Revision: C Effective Date: May 8, 2012

## **Trial Sponsor:**

Edwards Lifesciences LLC One Edwards Way Irvine, CA 92614 USA

PROPRIETARY DATA: This document and the information contained herein may not be reproduced, used or disclosed without written permission from Edwards Lifesciences LLC

Edwards Lifesciences, Edwards, the stylized E logo, Carpentier-Edwards, Magna Ease, PERIMOUNT, PERIMOUNT Magna, and ThermaFix are trademarks of Edwards Lifesciences Corporation.



## 1 PROTOCOL SIGNATURE PAGE

| Trial Title: | Clinical Trial of the Edwards Pericardial Aortic Bioprosthesis,<br>Model 11000 |
|---|---|
| Protocol Number: | 2010-03 |
| Version Number: | Rev. C |
| Date: | 8 MAY 2012 |

I have read this protocol and agree to participate in the clinical investigation of the Model 11000 sponsored by Edwards Lifesciences, LLC. I agree to conduct this investigation according to the requirements of the trial protocol and in accordance with Good Clinical Practice, applicable State and U.S. Federal regulations and conditions imposed by the reviewing Institutional Review Board/Ethics Committee/Research Ethics Board. I agree to supervise all sub-investigators at my site as well as the use of all of the investigational devices at my institution and to ensure appropriate informed consent is obtained from all subjects prior to inclusion in this trial.

| INVESTIGATOR NAME | INVESTIGATOR TITLE |
|------------------------|--------------------|
| INVESTIGATOR SIGNATURE | DATE |
| SPONSOR NAME | SPONSOR TITLE |
| SPONSOR SIGNATURE | DATE |



## 2 TRIAL CONTACT PERSONNEL

## 2.1 SPONSOR CONTACT





## 2.2 TRIAL CONTACT







## **Table of Contents**

| 1 | PF | ROTOC | OL SIGNATURE PAGE | 2 |
|----|------------|---------|--------------------------------------|----|
| 2 | TF | RIAL CO | NTACT PERSONNEL | 3 |
| | 2.1<br>2.2 | | OR CONTACTONTACT | |
| 3 | PF | ROTOC | OL SYNOPSIS | 7 |
| 4 | | | ATIONS | |
| 5 | | | JCTION | |
| • | | | | |
| | 5.1<br>5.2 | | UCTION AND BACKGROUND | |
| | | | Indication for use | |
| | | | Prior Testing | |
| | | | Prior clinical studies | |
| 6 | В | ENEFITS | S AND RISKS | 13 |
| | 6.1 | BENEFI | TS | 13 |
| | 6.2 | RISKS | | 13 |
| 7 | CI | ΙΝΙζΔΙ | TRIAL DESIGN | 14 |
| • | | | | |
| | 7.1 | | CATION | |
| | 7.2 | | SE | |
| | 7.3 | | INTS | |
| | | | Safety endpoints | |
| | - | | Performance endpoints | |
| | | | Other Data | |
| 8 | SI | JBJECT | POPULATION | 15 |
| | 8.1 | DEMOG | GRAPHIC AND CLINICAL CHARACTERISTICS | 15 |
| | 8.2 | INCLUS | ION CRITERIA | 16 |
| | 8.3 | Exclus | ION CRITERIA | 16 |
| | 8.4 | WITHD | RAWAL CRITERIA AND PROCEDURES | 17 |
| 9 | ST | TATISTI | CAL METHODS | 18 |
| | 9.1 | SAMPLI | E SIZE | 18 |
| | 9.2 | ANALYS | SIS POPULATION | 18 |
| | 9.3 | SAFETY | ANALYSIS | 18 |
| | 9.4 | PERFOR | RMANCE ANALYSIS | 18 |
| | 9.5 | OTHER | DATA | 19 |
| | 9.6 | MISSIN | G DATA | 19 |
| 10 | T | RIAL PR | OCEDURES | 19 |
| | 10.1 | Bas | ELINE EVALUATION | 20 |
| | | 0.1.1 | Subject screening | |
| | | 0.1.2 | Informed consent | |
| | | 0.1.3 | Baseline assessment | |
| | 10.2 | | GICAL PROCEDURE | |
| | 10 | 0.2.1 | Procedure preparation | |
| | | 0.2.2 | Model 11000 Implanting Procedure | |

## Clinical Trial Number: 2010-03

| | 10.2. | 3 Implant Assessment | 21 |
|----|--------|-----------------------------------------------|-----|
| | 10.3 | SUBJECT ENROLLMENT | 21 |
| | 10.4 | POST-PROCEDURE | 22 |
| | 10.4. | 1 Post-procedure care | 22 |
| | 10.4.2 | | |
| | 10.4. | 3 Follow-up assessments | 22 |
| | 10.5 | ECHOCARDIOGRAM | |
| | 10.6 | DEVICE REMOVAL / EXPLANT | |
| | 10.7 | MISSED SUBJECT VISITS | |
| | 10.8 | TRIAL SUBJECT EXIT | |
| | 10.9 | CLINICAL TRIAL TERMINATION | 24 |
| 11 | ADVE | ERSE EVENTS | .24 |
| | 11.1 | REPORTING PROCEDURE | 24 |
| | 11.2 | ADVERSE EVENT DEFINITIONS | |
| | 11.2. | | |
| | 11.2. | | |
| | 11.2. | ** | |
| | 11.2.4 | | |
| | 11.2. | 5 Unanticipated serious adverse device effect | 25 |
| | 11.3 | DEATHS AND EXPLANTS | |
| | 11.3. | | |
| | 11.4 | CLINICAL EVENTS COMMITTEE | 26 |
| 12 | TDIAL | L AND DATA MANAGEMENT | 20 |
| 14 | INIAL | | |
| | 12.1 | TRIAL CORE LABS | |
| | 12.1. | | |
| | 12.2 | DEVICE SHIPMENTS | |
| | 12.3 | INVENTORY AND ACCOUNTABILITY RECORDS | |
| | 12.4 | DEVICE STORAGE | |
| | 12.5 | DEVICE RETURN | |
| | 12.6 | PROTOCOL DEVIATIONS | |
| | 12.6. | | |
| | | Training | |
| | 12.7. | | |
| | 12.7.2 | | |
| | | MONITORING | |
| | 12.8. | | |
| | 12.8.2 | | |
| | 12.9 | DOCUMENTATION REQUIREMENTS | |
| | 12.9. | | |
| | 12.9.2 | | |
| | 12.9. | | |
| | 12.9.4 | | |
| | 12.10 | PROTOCOL AMENDMENTS | |
| | 12.11 | AUDITS AND INSPECTIONS | 30 |
| 13 | ETHIC | CAL AND REGULATORY CONSIDERATIONS | .30 |
| | 13.1 | APPLICABLE REGULATIONS AND GUIDELINES | 30 |
| | 13.2 | DATA PROTECTION AND SUBJECT CONFIDENTIALITY | 31 |
| | 13.3 | INFORMED CONSENT AND REVIEW COMMITTEES | 31 |

## Clinical Trial Number: 2010-03

| 13.4 | Investigator responsibilities | . 31 |
|---------|---------------------------------------|------|
| 13.4 | l.1 General duties | . 31 |
| 13.4 | 1.2 Investigator records | . 32 |
| 13.4 | 1.3 Investigator reports | . 32 |
| 13.5 | TRIAL SPONSOR RESPONSIBILITIES | . 32 |
| 13.5 | 5.1 General duties | . 32 |
| 13.5 | 5.2 Selection of investigators | . 33 |
| 13.5 | i.3 Monitoring the clinical trial | . 33 |
| 13.5 | i.4 Sponsor records | . 33 |
| 13.5 | 5.5 Sponsor reports | . 33 |
| 13.6 | PUBLICATION POLICY | . 33 |
| 14 REFE | ERENCES | 34 |
| 15 APPI | ENDICES | 34 |
| 15.1 | ADVERSE EVENT (CODES AND DEFINITIONS) | . 35 |
| 15.2 | SAMPLE INFORMED CONSENT FORM | |
| 15.3 | CASE REPORT FORMS | . 37 |
| 15.4 | PROTOCOL DEVIATION CODES | . 38 |
| 15.5 | DEVICE DEFICIENCY CODES | . 39 |
| 15.6 | ECHO MANUAL | . 40 |
| 15.7 | EQ-5D QUESTIONNAIRE | . 41 |
| 15.8 | SF-12 v2 Questionnaire | . 42 |



# 3 PROTOCOL SYNOPSIS

| Trial Number: | 2010-03 |
|---|---|
| Title: | Clinical trial of the Edwards Pericardial Aortic Bioprosthesis, Model 11000 |
| Trial Sponsor: | Edwards Lifesciences LLC<br>One Edwards Way, Irvine, CA 92614 USA |
| Krakow Principal Investigator: | |
| Warsaw Principal<br>Investigator: | |
| Trial<br>Purpose: | The purpose of this observational trial is to gather further clinical data to confirm the safety and performance of the Edwards Pericardial Aortic Bioprosthesis, Model 11000 in this trial population. |
| Trial Device: | Edwards Pericardial Aortic Bioprosthesis, Model 11000. An identical valve model, Model 11000A, has labeling that bears the CE marking of conformity under EC Design-Examination Certificate No. 2103732DE04 and CE Marking of Conformity Certificate No. 2103732CE04. |
| Intended Use: | The Model 11000 valve is intended for subjects who require replacement of their native or prosthetic aortic valve. |
| Trial Design: This is a prospective, non-randomized, non-controlled, observed clinical trial. Up to 200 subjects will be enrolled at up to 6 participating trial site subject is consented for a period of 5 years. All subjects will be as clinically at the following intervals: Baseline, Implant, discharmonths, and annually to 5 years. | |
| Population: | Adult subjects diagnosed with aortic valve disease requiring replacement of the native or prosthetic aortic valve. |
| Enrollment<br>Criteria: | <ul> <li>Is 18 years or older</li> <li>Provides written informed consent prior to trial procedures</li> <li>Diagnosed with aortic valve disease requiring a planned replacement as indicated in the preoperative evaluation</li> <li>Scheduled to undergo planned aortic valve replacement with or without concomitant bypass surgery</li> <li>Geographically stable and agrees to attend all follow-up assessments at the hospital of surgical services for up to 5 years</li> </ul> |



#### **Exclusion Criteria**

- Requires emergency surgery<sup>1</sup>
- Has prior mitral, tricuspid or pulmonic valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain in situ
- Requires multiple valve replacement/repair
- Requires a surgical procedure outside of the cardiac area (e.g. vascular bypass)
- Has aneurysm of the aortic root and/or ascending aorta requiring surgical intervention
- Has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months to the scheduled aortic valve replacement (AVR) surgery
- Has renal insufficiency as determined by creatinine (S-Cr) level ≥ 2.5 mg/dL or end-stage renal disease requiring chronic dialysis at screening visit
- Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to AVR surgery
- Has acute myocardial infarction (MI) within 30 days prior to AVR surgery
- Has presence of non-cardiac disease limiting life expectancy to less than 12 months
- Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM)
- Diagnosed with hyperparathyroidism
- Exhibits left ventricular ejection fraction ≤ 30% as validated by diagnostic procedure within 30 days prior to AVR surgery
- Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
- Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 60 days prior to AVR surgery
- Documented leukopenia (WBC < 3.5x 10³/μL), acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L), thrombocytopenia (platelet count < 50x10³/μL) or history of bleeding diathesis or coagulopathy</li>
- Diagnosed with myxomatous disease/connective tissue disorders (e.g. Marfan's Syndrome)
- Has prior organ transplant
- Current or recent participation (within 6 weeks prior to surgery) in an investigational drug or device trial
- Was previously implanted with trial device<sup>2</sup>

Emergent surgery – surgery is carried out on the referral day before the beginning of the next working day.

Note: Previously implanted means that the index aortic valve replacement procedure was completed. The procedure is complete when the surgeon takes the subject off cardiopulmonary bypass and restarts the heart.



| | <ul> <li>Pregnant (female subject of childbearing potential only), lactating or planning to become pregnant during the duration of participation in trial</li> <li>Currently incarcerated or unable to give voluntary informed consent</li> <li>Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant</li> </ul> |
|---|---|
| Trial Endpoints: | Safety Endpoints: Descriptive information of early rates and late linearized rates of the following: Structural valve deterioration Thromboembolism All bleeding/hemorrhage Major bleeding/hemorrhage All paravalvular leak Major paravalvular leak Non-structural valve dysfunction Endocarditis Hemolysis All cause mortality Trial valve-related mortality Explant Performance Endpoints: Clinically acceptable hemodynamic performance confirmed by core lab evaluation of echocardiography New York Heart Association (NYHA) functional class compared to baseline Change in Quality of Life questionnaires EQ-5D (EuroQol) and Short Form 12 version 2 (SF-12v2) from baseline/screening to 1-year |
| Other data: | Blood Data |



# 4 ABBREVIATIONS

| ACC | American College of Cardiology | | |
|---|---|---|---|
| | American College of Cardiology | | Instructions for the |
| AE | Adverse Event | IFU | Instructions for Use |
| AHA | American Heart Association | INR | International Normalized Ratio |
| AS | Aortic Stenosis | IRB | Institutional Review Board |
| ASD | Atrial Septal Defect | ISO | International Standardization Organization |
| AVR | Aortic Valve Replacement | LVOT | Left Ventricular Outflow Tract |
| CABG | Coronary Artery Bypass Graft | MI | Myocardial Infarction |
| CBC | Complete Blood Count | MOF | Multi-system Organ Failure |
| CEC | Clinical Events Committee | MR | Magnetic Resonance |
| CFR | Code of Federal Regulations | NSVD | Nonstructural Valve Dysfunction |
| CO/CI | Cardiac Output/Cardiac Index | NYHA | New York Heart Association |
| CRF | Case Report Form | OPC | Objective Performance Criteria |
| CV | Critical Value | PFO | Patent Foramen Ovale |
| CVA | Cerebrovascular Accident | PMA | Premarket Approval |
| DIC | Disseminated Intravascular Coagulation | POD | Postoperative Day |
| EC | Ethics Committee | PT | Prothrombin Time |
| eCRF | Electronic Case Report Form | PTFE | Polytetrafluoroethylene |
| ECG | Electrocardiogram | PTT | Partial Thromboplastin Time |
| EDC | Electronic Data Capture | PVL | Paravalvular Leak |
| EOA | Effective Orifice Area | QOL | Quality of Life |
| EQ-5D | EuroQol health questionnaire | RBC | Red Blood Cell |
| FDA | Food and Drug Administration | REB | Research Ethics Board |
| <b>FMEA</b> | Failure Modes and Effects Analysis | RGA | Returned Good Authorization |
| GCP | Good Clinical Practice | SAE | Serious Adverse Effect |
| GLP | Good Laboratory Practices | SAR | Specific Absorption Rate |
| HGB | Hemoglobin | SAVR | Surgical Aortic Valve Replacement |
| HIPAA | Health Insurance Portability & Accountability Act | SF-12 | Short Form 12 health questionnaire |
| HCT | Hematocrit | SVD | Structural Valve Deterioration |
| HIT | Heparin Induced Thrombocytopenia | TAD | Tissue Annulus Diameter |
| носм | Hypertrophic Obstructive Cardiomyopathy | TEE | Transesophageal Echocardiography |
| ICF | Informed Consent Form | TIA | Transient Ischemic Attack |
| ICU | Intensive Care Unit | UADE | Unanticipated Adverse Device Effect |
| ID | Identification | WBC | White Blood Cell |
| IDE | Investigational Device Exemption | | |



#### 5 INTRODUCTION

#### 5.1 INTRODUCTION AND BACKGROUND

Valvular heart disease is a life-threatening disease that afflicts millions of people worldwide and leads to approximately 250,000 valve repairs and/or replacements each year. The number of subjects requiring aortic valve replacement (AVR) is increasing due to prolonged life expectancy. Many subjects are asymptomatic until the disease is well advanced and, once diagnosed, have poor prognosis depending on the severity of valve calcification and history of cardiac events. Diseased heart valves can be treated by medication, surgical repair or surgical replacement.

#### 5.1.1.1 AORTIC HEART DISEASE

Aortic valvular heart disease includes conditions involving any of the following – obstructions of the aortic heart valve or stenosis; leakage of the aortic valve, known as regurgitation, incompetence, or insufficiency, and combinations of the two, sometimes referred to as mixed disease or combined lesions. Valvular heart disease may be caused by any number of factors, including congenital abnormalities, infection by various micro-organisms, degenerative calcification and rheumatic heart disease. When subjects become symptomatic, angina, syncope, and congestive heart failure (CHF) are the primary clinical signs observed. Studies report that among symptomatic subjects with medically treated moderate-to-severe AS, mortality rates after the onset of symptoms are approximately 25% at one year and 50% at two years. Other studies show that subjects with symptomatic AS have a life expectancy between 2 – 4 years. Neither aortic stenosis nor aortic insufficiency can be effectively treated medically; however, the symptoms of aortic valve disease can be managed medically.

## 5.1.1.2 TREATMENT OF AORTIC VALVULAR HEART DISEASE

Aortic stenosis and insufficiency can be treated by surgical intervention, including balloon valvuloplasty, valve repair, and valve replacement. Balloon valvuloplasty, a treatment option for aortic stenosis, utilizes a balloon-tipped catheter to stretch open the narrowed valve. Valvuloplasty is predominately used to treat children or adults who are poor surgical candidates. Valve repair techniques include annuloplasty for dilated valve disease, patching leaflet perforations, resected vegetations, or tears, and leaflet extension.<sup>3,4</sup> Aortic valve repair for stenosis does not show good clinical results.<sup>5</sup> Replacement of the aortic valve is indicated for symptomatic subjects and asymptomatic subjects with left ventricular dysfunction.

#### 5.1.1.3 BIOPROSTHETIC HEART VALVES

Bioprosthetic heart valves are indicated for use in subjects suffering from valvular heart disease. These tissue valves are used particularly in those subjects for whom long-term anticoagulation therapy is contraindicated or who may be difficult to maintain on anticoagulation therapy.

### 5.2 DEVICE DESCRIPTION

Refer to the *Instructions for Use* in the Clinical Investigator's Brochure (CIB) for a complete description of the device.



The Edwards pericardial aortic bioprosthesis, Model 11000, is a trileaflet bioprosthesis comprised of bovine pericardium that has been preserved in a buffered glutaraldehyde solution and mounted on a flexible frame. It is available in sizes 19, 21, 23, 25, 27, and 29 mm. The bioprosthesis is stored in non-liquid packaging.

The frame is designed to be compliant at the orifice as well as at the commissures. The compliance of the commissure supports is intended to reduce the loading shock at the valve commissures and free margin of the leaflets. The compliance of the orifice is intended to reduce the stress on the leaflets. The compliant orifice concept is based on the physiology and mechanics of natural heart valves and reported experience with implantation of unstented homografts.

The lightweight wireform is made of a corrosion-resistant cobalt-chromium alloy, chosen because of its superior efficiency and fatigue-resistant characteristics, and is covered with a woven polyester fabric.

A thin cobalt-chromium alloy/polyester film laminate band surrounds the base of the wireform frame providing structural support for the orifice. A silicone-rubber sewing ring covered with a porous, seamless polytetrafluoroethylene (PTFE) cloth attached to the wireform frame, which facilitates tissue ingrowth and encapsulation. The aortic sewing ring has been scalloped to conform to the natural aortic root. The compliant nature of the sewing ring facilitates coaptation between the bioprosthesis and an often irregular or calcific tissue bed.

To facilitate implantation in patients with small aortic roots, the Model 11000A has a low profile height. The sewing ring has three, equally spaced black silk suture markers at the cusp centers to aid in bioprosthesis orientation and suture placement.

#### The Model 11000 bioprosthesis does not require rinsing prior to implantation.

A holder is attached to the bioprosthesis by means of sutures to facilitate handling and suturing the bioprosthesis during implantation. The holder is easily detached by the surgeon.

Edwards Pericardial Aortic Bioprosthesis, Model 11000. An identical valve model, Model 11000A, has labeling that bears the CE marking of conformity under EC Design-Examination Certificate No. 2103732DE04 and CE Marking of Conformity Certificate No. 2103732CE04.

#### 5.2.1 INDICATION FOR USE

The Model 11000 is intended for patients who require replacement of their native or prosthetic aortic valve.

Refer to the *Instructions for Use* in the Clinical Investigator's Brochure (CIB) for contraindications, procedure steps, and cautions.

#### 5.2.2 PRIOR TESTING

A Clinical Investigator's Brochure (CIB) is prepared for the Model 11000; please refer to this document for pre-clinical testing.

## 5.2.3 PRIOR CLINICAL STUDIES

Twenty (20) subjects are implanted with the Model 11000 Pericardial Bioprosthesis under Version A of this ongoing clinical trial.



A summary of prior clinical studies on similar pericardial valves are included in the Clinical Investigator's Brochure.

#### 6 BENEFITS AND RISKS

#### 6.1 BENEFITS

The benefits of the Model 11000 are assumed the same as other bioprosthetic valves including improved valvular function, acute alleviation of symptoms related to aortic stenosis or insufficiency, and/or improved morbidity and mortality. The additional benefits of this valve are not yet proven.

The anticipated additional benefits of aortic valve, Model 11000 are to eliminate the need for rinsing the index valve prior to implant, less exposure to the risks of glutaraldehyde, and elimination of hazardous waste requiring special disposal.

#### 6.2 RISKS

As with all prosthetic heart valves, serious complications, sometimes leading to death may be associated with the use of tissue valves. Complications due to individual subject reaction to an implanted device, or to physical or chemical changes in the components, particularly those of biological origin, may occur at varying intervals (hours or days) necessitating reoperation and replacement of the prosthetic device. Some or all of the risks listed below could require a reoperation or explant, and/or they may lead to permanent disability or death.

# Known/potential risks associated with stented bioprosthetic heart valves include but not limited to:

- Angina
- Bleeding diatheses (coagulopathy) related to anticoagulant therapy
- Cardiac arrhythmias
- Cardiac failure
- Coronary ostial blockage
- Endocarditis
- Hemolysis/Hemolytic anemia
- Hemorrhage
- Immunological response
- Leaflet entrapment (impingement)
- Myocardial infarction
- Nonstructural valve dysfunction
- Paravalvular/Perivalvular leak

- Malfunctions of valve due to distortion at implant, fracture of wireform, physical and or chemical deterioration of valve components
- Patient prosthetic mismatch (PPM)
- Regurgitation/insufficiency
- Stenosis
- Thromboembolism/stroke
- Tissue deterioration including infection, calcification, thickening, perforation, degeneration, suture abrasion, instrument trauma, and or leaflet detachment
- Transient ischemic attack (TIA)
- Valve pannus
- Valve thrombosis



## Potential risks associated with aortic valve replacement surgery include but not limited to:

- Allergic reaction
- Annular dissection
- Aortic dissection
- Arterial dissection
- Bleeding, anticoagulant related
- Bleeding, procedural
- Bleeding, post-procedural
- Cardiac arrest
- Cardiogenic shock
- Disseminated intravascular coagulation (DIC)
- Esophageal rupture
- Heart failure
- Hematoma
- Heparin induced thrombocytopenia (HITs)
- Hypotension
- Hypertension

- Hypoxemia
- Infection, local or wound
- Infection, systemic (septicemia)
- Myocardial infarction
- Multi-system organ failure (MOF)
- Pericardial effusion
- Pericardial tamponade
- Pleural effusion
- Pulmonary edema
- Pneumonia
- Renal dysfunction
- Respiratory failure
- Thromboembolism
  - Venous, peripheral or central
  - Arterial, peripheral or central
  - Pulmonary, thrombus or other

Risks associated with Model 11000 are anticipated to be the same as those listed above for other aortic bioprosthetic valves and valve replacement surgery. Based on pre-clinical testing, there are no new risks anticipated with the Model 11000 tissue process or sterilization method.

There may be other unknown risks. All safety events will be collected and reviewed throughout the entire trial and follow-up period. Investigators will be notified of any additional risks identified that could affect the health, safety or welfare of the trial subjects.

#### 7 CLINICAL TRIAL DESIGN

This is a prospective, non-randomized, non-controlled, observational clinical trial. Up to 200 subjects will be enrolled at up to 6 participating trial sites. Each subject is consented for a period of 5 years. All subjects will be assessed clinically at the following intervals: Baseline, Implant, discharge, 3 months and annually to 5 years.

#### 7.1 JUSTIFICATION

This trial is designed to confirm that the performance observed in pre-clinical testing also is observed in the human population.

#### 7.2 PURPOSE

The purpose of this observational trial is to gather further clinical data to confirm the safety and performance of the Edwards Pericardial Aortic Bioprosthesis, Model 11000 in this trial population.



#### 7.3 ENDPOINTS

#### 7.3.1 SAFETY ENDPOINTS

Descriptive information of early rates and late linearized rates of the following:

- Structural valve deterioration
- Thromboembolism
- All bleeding/hemorrhage
- Major bleeding/hemorrhage
- All paravalvular leak
- Major paravalvular leak

- Non-structural valve dysfunction
- Endocarditis
- Hemolysis
- All cause mortality
- Trial valve-related mortality
- Explant

#### 7.3.2 Performance endpoints

The following performance endpoints will be assessed at each scheduled follow-up visit:

- Clinically acceptable hemodynamic performance confirmed by core lab evaluation of echocardiography
- New York Heart Association (NYHA) functional class compared to baseline
- Change in Quality of Life questionnaires EQ-5D (EuroQol) and Short Form 12 version 2 (SF-12v2) from baseline/screening to 1-year

#### 7.3.3 OTHER DATA

The following blood data also will be collected at baseline, 3 months, and at each annual visit:

Complete blood count (CBC): including White Blood Cell Count (WBC), Red Blood Cell Count (RBC), Hemoglobin (Hgb), Hematocrit (HCT), and platelet count (PLT), and plasma free hemoglobin.

Serum creatinine will be collected at baseline only.

Coagulation profile will be collected at baseline, discharge, 3 months, and at the 1, 3, and 5 year follow-up visits.

## 8 SUBJECT POPULATION

## 8.1 DEMOGRAPHIC AND CLINICAL CHARACTERISTICS

Adult subjects diagnosed with aortic valve disease and scheduled to undergo aortic valve replacement are eligible for participation in the clinical trial.

#### 8.2 INCLUSION CRITERIA

The principal investigator at the trial site has the responsibility of screening potential subjects to determine if the patients meet all the inclusion criteria. The following are requirements for entry into the clinical trial:

- Is 18 years or older
- Provides written informed consent prior to trial procedures
- Diagnosed with aortic valve disease requiring a planned replacement as indicated in the preoperative evaluation
- Scheduled to undergo planned aortic valve replacement with or without concomitant bypass surgery
- Geographically stable and agrees to attend all follow-up assessments at the hospital of surgical services for up to 5 years

#### 8.3 EXCLUSION CRITERIA

The principal investigator at the trial site must exclude subjects if any of the exclusion criteria are present. The following are the criteria for exclusion from participating in the clinical trial:

- Requires emergency surgery<sup>3</sup>
- Has prior mitral, tricuspid or pulmonic valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain in situ
- Requires multiple valve replacement/repair
- Requires a surgical procedure outside of the cardiac area (e.g. vascular bypass)
- Has aneurysm of the aortic root and/or ascending aorta requiring surgical intervention
- Has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months to the scheduled aortic valve replacement (AVR) surgery
- Has renal insufficiency as determined by creatinine (S-Cr) level ≥ 2.5 mg/dL or end-stage renal disease requiring chronic dialysis at screening visit
- Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to AVR surgery
- Has acute myocardial infarction (MI) within 30 days prior to AVR surgery
- · Has presence of non-cardiac disease limiting life expectancy to less than 12 months
- Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM)
- Diagnosed with hyperparathyroidism
- Exhibits left ventricular ejection fraction ≤ 30% as validated by diagnostic procedure within 30 days prior to AVR surgery
- Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
- Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 60 days prior to AVR surgery

<sup>&</sup>lt;sup>3</sup> Emergent surgery – surgery is carried out on the referral day before the beginning of the next working day.



- Documented leukopenia (WBC < 3.5x 10<sup>3</sup>/μL), acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L), thrombocytopenia (platelet count < 50x10<sup>3</sup>/μL) or history of bleeding diathesis or coagulopathy
- Diagnosed with myxomatous disease/connective tissue disorders (e.g. Marfan's Syndrome)
- Has prior organ transplant
- Current or recent participation (within 6 weeks prior to surgery) in an investigational drug or device trial
- Was previously implanted with trial device<sup>4</sup>
- Pregnant (female subject of childbearing potential only), lactating or planning to become pregnant during the duration of participation in trial
- Currently incarcerated or unable to give voluntary informed consent
- Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant

#### 8.4 WITHDRAWAL CRITERIA AND PROCEDURES

Subjects may voluntarily withdraw consent at any time during the clinical trial with no loss of benefit or penalty. Subjects will be exempt from follow-up after withdrawing from the clinical trial. For subjects consented but have withdrawn, the trial site must retain the subject's informed consent and all documents pertaining to the subject prior to the subject's withdrawal.

The Investigator may withdraw any subject due to any of the following conditions:

- Participation in the clinical trial may be contrary to the subject's current medical treatment, based on new information or changes in the subject's medical condition.
- Any anatomical findings that would determine subject not suitable for implant with the Edwards aortic valve, Model 11000, which are discovered, intra-operatively. These may include findings such as:
  - The position of the coronary ostia relative to the Edwards aortic valve, Model 11000 would result in obstruction of blood flow,
  - the subject is hemodynamically unstable during the procedure requiring the procedure to be aborted prior to implanting the trial device,
  - c. A device is not available in the correct size for the subject;

The Investigator will document the withdrawal of trial subjects and notify the Trial Sponsor within five (5) working days. Additional subjects will be screened to replace those subjects who are withdrawn by the Investigator during the surgical procedure prior to implant.

Edwards will inform the Investigator of any new information about the trial that may affect the health, safety or welfare of the subjects or that may influence subject's decision to continue participating in the trial.

<sup>&</sup>lt;sup>4</sup> Note: Previously implanted means that the index aortic valve replacement procedure was completed. The procedure is complete when the surgeon takes the subject off cardiopulmonary bypass and restarts the heart.



## 9 STATISTICAL METHODS

#### 9.1 SAMPLE SIZE

Up to 200 subjects will be enrolled in the trial at up to 6 participating sites.

#### 9.2 ANALYSIS POPULATION

The analyses of safety data will include all enrolled subjects. Subjects are considered enrolled in the clinical trial after meeting the enrollment criteria, signing the informed consent and the surgeon determines that the index valve can be implanted.

The analyses of performance data will include the index valve population, defined as all subjects that are enrolled into the trial and that are implanted with the index valve.

#### 9.3 SAFETY ANALYSIS

Early adverse events within 30 days of procedure will be reported as the number of events divided by the number of enrolled subjects. Linearized rates will be used to summarize adverse events for the late (>30 days) post-operative period. The linearized rates will be calculated as the number of late events divided by the total number of late-subject years.

Percentages for the early events and linearized rates for the late events also will be calculated for all other complications observed in the trial.

Actuarial rates based on the method of Kaplan-Meier will be calculated for each of the safety endpoints at each of the follow-up time points.

#### 9.4 PERFORMANCE ANALYSIS

## Hemodynamic Variables

Valvular regurgitation will be summarized by the number and percentage of subjects in each level of regurgitation. Other hemodynamic parameters will be summarized by N, mean, and standard deviation. These summaries will be summarized at baseline and each applicable follow-up visit for all subjects in the investigational valve population, and will be stratified by valve size.

#### NYHA Class

A comparison of preoperative and postoperative NYHA functional class (presented as the percentage of subjects in each class at baseline, at each follow-up time-point, and as the percentage of subjects at each follow-up time-point who improved, worsened, or did not change in class) will be presented. This comparison will be based on the investigational valve population. Additionally, a cross-tabulation of baseline vs. 1-year NYHA Class will be presented for all subjects in the investigational valve population with both baseline and 1-year NYHA data.

## Quality of Life

The number, mean and standard deviation for the Quality of Life (EQ-5D) summary measurement will be presented at the pre-procedure and at the 1-year post procedure follow-up visit. In addition, the number and mean for the change from pre-procedure to the 1-year post procedure follow-up visit will be calculated and presented.



The number, mean, and standard deviation for the SF-12 physical and mental health summary measures (PCS-12 and MCS-12, respectively) will be calculated at the pre-procedure and at the 1-year pos procedure follow-up visit. In addition, the number and mean for the change from pre-procedure to the 1-year follow-up in PCS-12 and MCS-12 will be presented.

#### 9.5 OTHER DATA

The mean and standard deviation of blood data will be calculated and presented.

#### 9.6 MISSING DATA

All analyses will apply to any available valid data. No data imputation will be performed for missing data.

## 10 TRIAL PROCEDURES

Table 3 summarizes all procedures to be conducted during the trial.

1, 3, 5 2 & 4 Trial Procedure Baseline Implant Discharge 3 months year years Written Informed Consent Х Pregnancy Test Х Medical History Х Medical Evaluation Х Х Х Х Х Height Х Weight Х Х Х 12-lead ECG Х Х Х Х Х NYHA Х Х Х Х Medications Х Х Х Х Х Adverse Events Х Х Х Х Х χ² Echocardiography (TTE) Х X Χ Х Echocardiography<sup>3</sup> (TEE) Х Auscultation χ<sup>2</sup> Quality of Life (EQ-5D and SF-12v2)4 Х Х **Blood tests** Complete Blood Count<sup>5</sup> Х X Х Х X Plasma free hemoglobin Х Х Х Х Х Serum Creatinine Х Coagulation Profile Х Х Х

**Table 3: Summary of Trial Assessments** 

#### Procedure table notes:

- 1 TTE will be the standard echo assessment for the aortic valve
- 2 If murmur heard then echo required
- 3 TEE intra-operatively and within 1 hour (from cross clamp removal) to confirm placement of the device and confirm initial function
- 4 Quality of Life only required at Baseline and at 1-year post-procedure
- 5 Complete blood count includes red blood cells, white blood cells, hemoglobin, hematocrit, platelet count



## 10.1 BASELINE EVALUATION

#### 10.1.1 Subject screening

All subjects diagnosed with aortic valve disease requiring aortic valve replacement seen by cardiac surgeons participating in this clinical trial should be pre-screened for eligibility. All subjects who meet initial eligibility requirements will be asked to participate. A Screening Log will be provided to the trial sites to maintain a cumulative log of all screened subjects admitted for aortic valve replacement by the cardiac surgeons participating in this trial. For subjects listed as not eligible for participation in the clinical trial, a reason supporting the disqualification of the subject must be entered on the screening log. The Screening Log shall be completed and faxed to the Trial Sponsor regularly (at least once per month). Any subject deemed ineligible due to active endocarditis, recent myocardial infarction, pregnancy or lactating, or due to participation in another clinical trial may be re-screened later. Re-screened subjects must be re-entered on the Screening Log.

#### 10.1.2 INFORMED CONSENT

Subjects who are eligible for participation in the clinical trial shall be provided with patient consent information, approved by the site's ethics committee (EC). Each subject shall be given ample time to read the Informed Consent in its entirety and ask questions to make an informed decision. The subject must sign and date the trial approved Informed Consent prior to participation, i.e. prior to any trial procedures. Subjects who provide informed consent will be assigned a trial subject identification number. The Investigator, or designee, and any witnesses shall also sign and date the consent form, as applicable. Failure to provide Informed Consent renders the subject ineligible for participation in the clinical trial including undergoing treatment with the trial device. Subjects who do not provide informed consent are recorded on the Screening Log.

#### 10.1.3 BASELINE ASSESSMENT

After a written informed consent has been obtained from the subject the following baseline data will be obtained (see **Table 4**); demographic and medical history, 12-lead electrocardiogram (ECG), transthoracic echocardiograph (TTE) per protocol, blood studies per protocol, an assessment of NYHA Functional Classification, Quality of Life (EQ-5D and SF-12v2), and coagulation profile (via INR or PTT). Test results conducted within 30 days before aortic valve surgery may be used for this trial if all values per protocol are available and there has been no significant change in the subject's condition that would affect the test results.

**Table 4 Baseline Assessment** 

| Clinical/Physical Assessment | | Blood Studies | Echocardiography (TTE) |
|---|---|---|---|
| Date of Assessment | Anti-thromboembolic | Blood Draw Date | Date of Exam |
| Date of Birth | Therapy | White Blood Cell Count | |
| Sex/Gender | (medications) | Red Blood Cell Count | |
| Height | Cardiovascular Risk Factors | Hemoglobin | REFER TO ECHO MANUAL |
| Weight | Cardiovascular Conditions | Hematocrit | |
| Heart Rate | Previous Procedures / | Platelet Count | |
| Blood Pressure | Interventions | Plasma Free | |
| Cardiac Rhythm (12-lead ECG) | Non-Cardiovascular | Hemoglobin | |
| NYHA Classification | Conditions | Serum Creatinine | |
| Quality of Life (EQ-5D & SF-12v2) | Pregnancy Test | Coagulation Profile | |

#### 10.2 SURGICAL PROCEDURE

#### 10.2.1 PROCEDURE PREPARATION

The surgical approach used will be at the discretion of the investigator per his/her routine surgical practice. At the time of aortic valve replacement, a transesophageal echocardiogram to further assess the anatomy is recommended prior to aortic valve (to ensure no withdrawal criteria are met per section 8.4). After performing the aortotomy, the native valve and surrounding anatomy should be examined for compatibility with the device again to ensure no withdrawal criteria are met.

#### 10.2.2 MODEL 11000 IMPLANTING PROCEDURE

A detailed description of device preparation and use is provided in the Instructions for Use (IFU), (See Clinical Investigator's Brochure). Investigators must be familiar with Precautions and Implant Technique described in the IFU prior to use of the index valve.

#### 10.2.3 IMPLANT ASSESSMENT

A Transesophageal echo (TEE) should be performed within 1 hour after the index valve is implanted (from cross clamp removal) to assess placement and index valve function. The echo requirements are in the Echo Manual.

Procedural information, findings, results and device identification information to be recorded is identified in .

Table 5 :Procedural information

| General information | Clinical information | Device performance |
|---|---|---|
| Date of Admission | Etiology | Valve size and serial number |
| Date of Procedure | Diagnosis for replacement | Post-operative TEE (within 1 |
| Implanting Surgeon | Valve implant | hour) |
| Type of Operation | Condition of the native aortic valve Sizing | REFER TO ECHO MANUAL |
| | Concomitant procedures Intraoperative Adverse Events | |

#### 10.3 SUBJECT ENROLLMENT

Subjects will be considered enrolled in the clinical trial after meeting the enrollment criteria, signing the informed consent and the surgeon determines that the index valve can be implanted. The point of enrollment in the clinical trial is established in the Operating Room when the investigator confirms that the subject is an appropriate candidate for the index valve or trial device and attempts to implant the valve. Additional subjects will not be enrolled to replace those subjects implanted with the index valve who choose to withdraw from the clinical trial.

## 10.4 POST-PROCEDURE

#### 10.4.1 POST-PROCEDURE CARE

At the discretion of the investigator, bioprosthetic heart valve recipients should be maintained on anticoagulant therapy (except when contraindicated) during the initial healing stages after implant, approximately 2 to 3 months in accordance with the ACC/AHA 2008 Guidelines for the Management of Patients with Valvular Heart Disease. Anticoagulants should then be discontinued over a period of 10 days, except in those patients for whom ongoing anticoagulant protection is indicated, i.e. in the absence of sinus rhythm and in patients with a dilated left atrium, calcification of the atrial wall, history of previous atrial thrombus, or any other medical condition requiring anticoagulation therapy. However, the appropriate anticoagulation therapy must be determined by the physician on an individual basis.

#### 10.4.2 DISCHARGE

**Table 6** identifies the medical information and clinical evaluation of trial subjects at discharge, which includes an echocardiogram (refer to Section 10.5).

Table 6 Discharge Information

| Table 6 District 8c Internation | | |
|---|---|---|
| Clinical/Physical Assessment | Blood Studies | Echocardiography (TTE) |
| Date of Discharge | Blood Draw Date | Date of Exam |
| Weight | White Blood Cell Count | |
| Heart Rate | Red Blood Cell Count | REFER TO ECHO MANUAL |
| Blood Pressure | Hemoglobin | |
| Cardiac Rhythm (12-lead ECG) | Hematocrit | |
| Anti-thromboembolic Therapy | Platelet Count | |
| (medications) | Plasma Free Hemoglobin | |
| Adverse Events | Coagulation Profile | |

Subjects, who are not discharged within 10 days post procedure must have an echocardiogram (refer to Section 10.5) to further assess placement and performance of the index valve. This echocardiogram is required to complete the evaluation of valve short-term function. Those subjects will not require an additional echocardiogram at discharge.

#### 10.4.3 FOLLOW-UP ASSESSMENTS

Post-procedure clinical evaluation will be performed on all enrolled trial subjects at scheduled visits at the trial site. The follow-up windows are listed in **Table 7**.

Table 7: Follow-up Windows

| Follow-up Assessment* | Assessment Window |
|-----------------------|-------------------|
| 3 months | ± 1 month |
| 1 year | ± 1 month |
| 2 years | ± 3 month |
| 3 years | ± 3 month |
| 4 years | ± 3 month |
| 5 years | ± 3 month |

<sup>\*</sup>Follow-up visits are calculated from the implant date.



During each postoperative follow-up visit, the investigator(s) will determine the subject's availability for future follow-up visits. If any subject needs to be seen, at a time other than a regularly scheduled follow-up visit, due to an index device related event, the required data collection would be the same as the 1 year follow-up evaluation.

Table 8 Follow-Up Information at all Post-Discharge Visits (3 months and annually to 5 years)

| Clinical/Physical Assessment | Blood Studies | Echocardiography (TTE) <sup>3</sup> |
|---|---|---|
| Date of Discharge | Blood Draw Date | Years 1, 3, 5: |
| Physical Assessment | White Blood Cell Count | Date of exam |
| Cardiac Rhythm (12-lead ECG) | Red Blood Cell Count | SEE ECHO MANUAL |
| NYHA Classification | Hemoglobin | Years 2, 4: |
| Quality of Life (EQ-5D & SF12-v2)1 | Hematocrit | Date of exam |
| Anti-thromboembolic Therapy | Platelet Count | |
| (medications) | Plasma Free Hemoglobin | Auscultation <sup>4</sup> |
| Adverse Events | Coagulation Profile <sup>2</sup> | |

<sup>1</sup> Quality of Life (EQ-5D and SF12-v2) will be completed only at the 1-year follow-up visit

#### 10.5 ECHOCARDIOGRAM

Echocardiograms will be independently analyzed by the Echocardiography Core Lab. Each sonographer participating in the clinical trial must be trained on the requirements of the Echo Manual.

#### 10.6 DEVICE REMOVAL / EXPLANT

Index valve 'removal' is the excision of the investigational valve, before implant of the investigational valve is complete, i.e., the heart is not restarted with the investigational valve in place. If the surgeon is unable to satisfactorily position or sew in the index valve, it will be removed and returned to the trial Sponsor who will provide a return valve kit. If the heart is restarted, the valve will be considered implanted and if removal is required from this point forward, it will be considered an explant.

In the event a valve is explanted, a copy of the procedure report must be provided to the trial Sponsor. Information on the cause of explant and its relationship to the valve will be provided by the investigator(s). Explanted valves must be returned to the trial Sponsor for analysis. Return kits for devices will be provided by the trial Sponsor.

## 10.7 MISSED SUBJECT VISITS

The Investigator(s) will make every attempt to follow the subjects and subjects will be encouraged by the Investigator(s) to report any address or telephone number changes to the trial site. They will also be informed of the importance of returning for scheduled follow-up visits even if they are not having any problems.

<sup>&</sup>lt;sup>2</sup>Coagulation profile will be completed only at years 1, 3, and 5

<sup>&</sup>lt;sup>3</sup> Exam to be performed as described in the Echo Manual. Data evaluation performed by a Core Lab.

<sup>&</sup>lt;sup>4</sup> TE will be the standard echo assessment for the aortic valve but will only be completed if murmur is heard on auscultation at year 2 and year 4 interval visits.



If a subject cannot be reached for a follow-up visit, the Investigator will document on the CRF, the efforts undertaken to contact the subject or the subject's primary health care provider. These efforts should include 2 attempts of telephone contact at separate dates and times, and a registered letter before the end of the follow-up window. If a subject cannot be reached for a follow-up visit, or misses a scheduled visit, the visit will be recorded as a missed visit on the date of last attempted contact. Subjects who miss a visit will not be considered withdrawn. At the next visit interval, the Investigator and/or designee will attempt to contact the subject again for follow-up. Should this attempt to contact the subject fail, a family member should be contacted in addition to the subject. Subjects who miss 2 sequential follow-up visits will be considered lost to follow-up at the second missed visit and exempt from further trial follow-up. After the subject is terminated from the trial, the Investigator will attempt to determine if the subject is alive, including searching national mortality registries as permitted by local laws.

#### 10.8 TRIAL SUBJECT EXIT

Trial Subjects exit the trial when no additional follow-up visits, procedures, or data collection are required. A subject is exited from the trial in the following instances:

- Subject fails enrollment criteria after written consent
- Subject is considered enrolled as "intent to treat" however surgeon is unable to complete the implant procedure\*
- Subject has trial device explanted\*
- Subject is lost-to-follow-up
- Subject withdraws from the trial
- Subject death
- Subject completes trial follow-up

#### 10.9 CLINICAL TRIAL TERMINATION

The principal investigator(s) will be notified in writing upon termination of the clinical trial. The Trial Sponsor retains the right to suspend or terminate this clinical trial at any time. Upon trial termination, the Investigator will contact the trial subjects to perform a final follow-up assessment within 2 months of trial termination. If a subject completed a protocol scheduled clinical evaluation within 6 months prior to trial termination, the final follow-up assessment may be completed by telephone. Subjects should continue seeing their physicians as part of routine clinical follow-up after heart valve replacement surgery.

## 11 ADVERSE EVENTS

## 11.1 REPORTING PROCEDURE

Adverse event information will be reported throughout the clinical trial as they occur. Adverse events will be followed until they are adequately resolved or explained. The investigator(s) should report any serious adverse event to the Trial Sponsor's Clinical Research department within 48 hours after the investigator's first knowledge of the event, followed by a written working days. Notification should be done via email ten HVTClinicalResearch@edwards.com or faxed to +1 (949) 250-5010. In addition, trial sites will

<sup>\*</sup> Subjects will be followed for 30 days or until any adverse events experienced by this cohort are resolved and then will be exited from the trial.



report all adverse events to their local EC in accordance with the review committee's requirements.

## 11.2 ADVERSE EVENT DEFINITIONS

## 11.2.1 ADVERSE EVENT

An adverse event (AE) is defined in ISO 14155:2011 (referred to hereafter as ISO 14155) as any untoward medical occurrence in a subject.

#### 11.2.2 ADVERSE DEVICE EFFECT

An adverse device effect (ADE) is defined in ISO 14155 as any untoward or unintended response to a medical device. This definition includes any event resulting from insufficiencies or inadequacies in the instructions for use or the deployment of the device or any event that is a result of user error.

#### 11.2.3 SERIOUS ADVERSE EVENT

A serious adverse event (SAE) is defined in ISO 14155 an adverse event that: led to death, led to a serious deterioration in the health of the subject that resulted in a life-threatening illness or injury, resulted in a permanent impairment of a body structure or a body function, required inpatient hospitalization or prolongation of existing hospitalization, or resulted in medical or surgical intervention to prevent permanent impairment to body structure or a body function, or led to fetal distress, fetal death or a congenital abnormality or birth defect.

#### 11.2.4 SERIOUS ADVERSE DEVICE EFFECT

A serious adverse device effect (SADE) is defined in ISO 14155 as an adverse device effect that resulted in any of the consequences characteristics of a serious adverse event or that might have led to any of these consequences if suitable action had not been taken or intervention had not been made or if circumstances had been less opportune.

#### 11.2.5 UNANTICIPATED SERIOUS ADVERSE DEVICE EFFECT

An unanticipated serious adverse device effect (USADE) is defined as serious adverse device effect, which by its nature, incidence, severity or outcome is not identified in the Clinical Investigator's Brochure.

## 11.3 DEATHS AND EXPLANTS

#### 11.3.1 SUBJECT DEATHS

In the event of subject death, every effort should be made to obtain a copy of the autopsy report and/or death summary. Information on the cause of death and its relationship to the device used in this clinical trial will be determined by the principal investigator. Copies of an autopsy report, if available, and/or a death summary are to be sent to the Trial Sponsor.

If a device is explanted during autopsy, the device should be returned to the Trial Sponsor for analysis. Return kits for devices will be provided upon request by the clinical monitor.



## 11.4 CLINICAL EVENTS COMMITTEE

The Clinical Events Committee (CEC) evaluates adverse events that are endpoint related. The CEC adjudicates events for their relatedness to the investigational device and/or the surgical procedure. The CEC will be composed of physicians familiar with the treatment of valvular heart disease and cardiac surgery who are not participating in the investigational trial.

The trial Sponsor will provide the CEC completed case report forms and any relevant source documentation/subject information as provided by the clinical site investigators. Trial Sponsor will insure that all information is de-identified before presenting to the committee. The CEC documents its findings or rulings on each event. All meeting minutes and supporting documentation are maintained by the CEC administrator with a copy provided to the trial Sponsor.

## 12 TRIAL AND DATA MANAGEMENT

#### 12.1 TRIAL CORE LABS

#### 12.1.1 ECHOCARDIOGRAPHY CORE LAB

The Echo Core Lab is responsible for independently evaluating echocardiograms submitted preoperatively and postoperatively by trial sites, and for reporting of hemodynamic and other valvular function results. Echocardiograms will be sent directly from the investigational sites to the Echo Core Lab. See **Appendix 15.7** for the Echo Core Lab Manual.

#### 12.2 DEVICE SHIPMENTS

An initial set of Edwards's aortic valve, Model 11000 will be shipped to the trial site once the following conditions are met: the trial site has obtained Ministry of Health and Ethics Committee approval, a signed Clinical Trial Agreement is in place, and the Site Initiation Visit, including Principal Investigator training, has been completed. Additional devices will be sent to the trial site as devices are used or as needed.

#### 12.3 INVENTORY AND ACCOUNTABILITY RECORDS

All device shipments will have inventory and shipment records. Devices may be hand carried to participating trial sites by Trial Sponsor personnel. Shipment will be accompanied by trial device documentation of delivery. The principal investigator(s) or designee will take inventory of the product and complete the delivery documentation with receipt date, condition of the device and signature. Both the trial site and the trial Sponsor will retain copies of these documents.

The investigator will maintain a Device Accountability Log of all trial devices received for use during this clinical trial. The log will be kept with the documents for the clinical trial and will be available for review during Trial Sponsor monitoring visits.

#### 12.4 DEVICE STORAGE

The device inventory will be stored in a locked, controlled, cool, dry and clean area as described in the Instructions for Use (IFU). This storage area shall be accessible only to the principal investigator(s), his/her co-investigator or approved designee. Only cardiac surgeons identified in



the Clinical Trial Agreement and/or on the Delegation of Authority form on file at the Trial Sponsor may implant the trial device.

#### 12.5 DEVICE RETURN

The principal investigator(s) will be notified in writing upon termination of the clinical trial. All unused devices in original package and/or those in opened packages as well as those removed from the original package will be returned upon receipt of this notice as described in the IFU. The Investigator's copy of the Device Accountability log must document any unused devices that have been returned. Contact Edwards Lifesciences, the Trial Sponsor, for additional instructions.

#### 12.6 PROTOCOL DEVIATIONS

A protocol deviation is defined as an event where the Investigator or trial personnel did not conduct the trial according to the clinical protocol or the Clinical Trial Agreement.

Deviations shall be reported to the Trial Sponsor regardless of whether medically justifiable or taken to protect the subject in an emergency. Subject specific deviations and non-subject specific deviations, (e.g. unauthorized use of a trial device outside the trial, unauthorized use of a trial device by a physician who is not listed in the Clinical Trial Agreement, etc.) will be reported in writing. Investigators will also adhere to procedures for reporting trial deviations to their EC in accordance with their specific EC's reporting policies and procedures.

For reporting purposes, deviations are classified as major or minor:

- Major deviations:
  - Any deviation from subject inclusion and exclusion criteria;
  - Any deviation from subject informed consent procedures;
  - Unauthorized use of an trial device outside the trial;
  - Unauthorized use of a trial device by a physician who is not listed in the Clinical Trial Agreement.
- Minor deviations:
  - Deviation from a protocol requirement such as incomplete/inadequate testing procedures;
  - Follow-up performed outside specified time windows.

#### 12.6.1 EXCEPTIONS

Some information collected in this trial is not essential to the trial endpoints and will not be considered deviation if absent.

#### 12.7 TRAINING

#### 12.7.1 TRAINING OF TRIAL SITE PERSONNEL

Principal investigator(s) and support staff will be trained by the Trial Sponsor on the use of the Edwards aortic valve, Model 11000 and accessories, the Protocol, the Clinical Investigator's Brochure, electronic Case Report Forms (eCRF) and Electronic Data Capture (EDC) system, device accountability procedures, GCP (Good Clinical Practices) Guidelines and other trial documents as applicable. A "Delegation of Authority Form" will be completed at each trial site designating which individuals are allowed to perform specific clinical trial related tasks. The



delegated tasks will determine what the training requirements are for each member of the trial support staff.

#### 12.7.2 DEVICES

Each cardiac surgeon participating in the clinical trial must be trained on the use of the device and the clinical protocol before screening potential subjects or using the Edwards aortic valve, Model 11000.

#### 12.8 MONITORING

#### 12.8.1 SITE INITIATION

Prior to subject enrollment, an initiation visit will be completed at each trial site to ensure the following:

- Ethics Committee and applicable regulatory body approvals have been obtained and documented,
- The investigators and clinical trial personnel are appropriately trained and clearly understand the trial,
- The investigators and clinical trial personnel accept the obligations incurred in undertaking this clinical trial.
- The Delegation of Authority form has been completed properly

#### 12.8.2 MONITORING METHODS

The Trial Sponsor will assign a monitor to monitor the progress of the clinical trial at each trial site. The monitor will remain in close contact with each trial site throughout the duration of the trial to provide any needed materials, (i.e. trial forms) or answer any questions. The monitor will be responsible for verifying that the subject signed the consent, reviewing date recorded on the eCRF, and visiting each trial site periodically to observe trial progress and compliance with clinical protocol and regulations applicable to this clinical trial.

Monitoring visits will be scheduled throughout the duration of the clinical trial between the monitor and the principal investigator at a mutually convenient and available time. These visits will assure that the facilities are still acceptable, the protocol and investigational plan are being followed, the EC has been notified of approved protocol changes as required, complete records are being maintained, appropriate timely reports have been made to the Trial Sponsor and the EC, device inventory are accounted for and controlled, and the investigator is carrying out all agreed activities. Any personnel changes must be reported to the monitor immediately and a training program scheduled and documented.

Periodic monitoring visits will be made at all enrolling trial sites in accordance with center enrollment rates. Trial sites should be visited a minimum of once each year by the monitor. Upon termination or conclusion of the clinical trial, the monitor will perform a close-out visit.

## 12.9 DOCUMENTATION REQUIREMENTS

Training will be documented on a training record provided by the Trial Sponsor, which the trainee must sign and date. The training of trial support staff must be completed and



documented before the staff member may perform the specific clinical trial related tasks delegated to them by the Principal Investigator.

## 12.9.1 Source documentation requirements

Clinical regulations require that Investigators maintain information in the clinical trial subject's medical records that corroborate data collected on the eCRF. Some examples of critical information to be maintained for review by the regulatory inspectors and Trial Sponsor monitors are:

- Medical history and physical condition of the clinical trial subject before involvement in the clinical trial sufficient to verify protocol entry criteria
- Dated and signed notes in the subject's medical record on the day of entry into the clinical trial.
- Dated and signed notes, laboratory records, and test reports, from each clinical trial subject visit with reference to the eCRF for further information, if appropriate (for specific results of procedures and exams).
- Notations on abnormal lab results, adverse events reported and their resolution.
- Notes regarding concomitant anticoagulant/antithrombotic medications taken during the clinical trial
- · Subject's condition upon completion of or withdrawal from the clinical trial.

To protect subject confidentiality, the subject's name must not appear anywhere on the imaging media sent to Edwards e.g. for reporting serious adverse events (SAE), or prepared for evaluation by the core lab. Each page should be identified with the subject's unique trial ID number. All other subject identifiers (i.e. medical record number, personal number) are to be obscured. Original copies of all data must be kept at the site.

## 12.9.2 DATA COLLECTION METHODS

All required data for this trial are to be collected with standardized Case Report Forms (CRF) for individual subjects; the eCRF outline is included in Appendix 16.5. Electronic CRF (eCRF) will be utilized for this trial. All eCRF must be electronically signed by the Principal Investigator or co-Investigator listed in the Clinical Trial Agreement and Delegation of Authority Log. If for any reason the eCRF are unavailable and/or inaccessible, paper CRF will be provided by the Trial Sponsor to be completed, signed by the Principal Investigator or designee and submitted to the Trial Sponsor.

Primary data collection should be drawn from the subject's hospital chart and operator worksheet (source document) reviews. All eCRF must be kept current to reflect subject status during the course of the trial.

Case Report Form Instructions will be provided to assist the Investigator(s) and appropriate trial staff with the completion of the required eCRF.

Data Management personnel will employ a full-featured relational Oracle database application on a central server. The application provides the capability of data collection remotely through the Internet so the participating site personnel may log on to the system securely and enter the data. Other data management programming and/or data analyses will be done in the database



system through the sponsor's internal network. All subjects' data collected in the system will be extensively verified through data validation programs, database integrity rules, and trial-specific data entry conventions for data accuracy and logical meaningfulness. Periodic analysis of all subjects' collected data will be performed in order to examine the expected distributions of data and to identify outliers for possible data entry errors.

#### 12.9.3 QUALITY CONTROL AND QUALITY ASSURANCE PROCEDURES

All data collected for the purposes of the trial must be documented in the subject's medical notes. Copies of relevant procedural records, examinations and laboratory test results should be kept on file in the Investigator's subject files, e.g. a copy of echo examination sent to the core lab should be kept with the subject records. Medical notes, eCRF and copies of test results must be available at all times for inspection by the trial monitor.

#### 12.9.4 COMMUNICATION PROCEDURES

During the course of the clinical trial, all correspondence (letters, records of telephone calls, emails and faxes) regarding the trial must be maintained in the trial binder provided by the Trial Sponsor. This binder must be made available for monitoring visits or audits.

#### 12.10 PROTOCOL AMENDMENTS

Changes in the protocol may be made only by written amendment agreed upon by the sponsor, the regulatory agency, and if pertinent, the EC. As appropriate, the Trial Sponsor will submit changes in the protocol to the pertinent regulatory agencies and investigators to obtain EC reapproval.

#### 12.11 AUDITS AND INSPECTIONS

In the event that audits are initiated by the sponsor or national/international regulatory authorities, the investigator shall allow access to the original medical records and provide all requested information.

#### 13 ETHICAL AND REGULATORY CONSIDERATIONS

#### 13.1 APPLICABLE REGULATIONS AND GUIDELINES

The regulations listed in Table 9 must be observed to comply with the Trial Sponsor's policy for conduct of clinical studies; they also represent sound research practice. It is the responsibility of the investigator(s) to comply with the requirements set forth in their country specific regulations.



Table 9: Applicable Regulations and Guidelines

| Region | Regulation / Guideline |
|---|---|
| Europe | - 93/42/EEC European Medical Device Directive (MDD) |
| | <ul> <li>ISO 14155:2011 (Clinical Investigation of Medical Devices for Human Subjects)</li> </ul> |
| | - ISO 5840: 2009 (Cardiovascular implants-Cardiac valve prostheses) |
| | - Declaration of Helsinki (2008) |
| Canada | - Canadian Medical Device Regulations (CMDR) |
| | - Canadian Investigational Testing Authorization as defined in the Medical Devices |
| | Regulation, May 1998 |

Furthermore, the investigator should use *Good Clinical Practice (GCP)* and must comply with the laws of the country, whichever will afford greater protection to subjects screened for participation in the clinical trial and subjects who participate in the trial.

#### 13.2 DATA PROTECTION AND SUBJECT CONFIDENTIALITY

The Trial Sponsor is dedicated to maintaining the confidentiality and privacy of subjects who volunteer to participate in the clinical trial. Passwords are issued to appropriate personnel to insure confidentiality and protection of the database by allowing variable levels of access to the computer system. In addition, the principal investigator is responsible for maintaining confidentiality throughout the clinical trial. Hard copies of source documentation are to be maintained in a secure area with limited access. All subject identifiers will be obliterated from all photocopies of source documents that have been removed from the trial site. Subject identifiers include, but are not limited to subject's name, subject's initials, social security number or equivalent, and medical / hospital number. All documents for the clinical trial will identify the subject by a subject identification number assigned by the Trial Sponsor.

#### 13.3 INFORMED CONSENT AND REVIEW COMMITTEES

All subjects must provide written informed consent in accordance with the local trial site's EC rules and regulations. A copy of the consent form from each center must be forwarded to the Trial Sponsor for review and approval prior to submitting it to the EC. Each center must provide the Trial Sponsor with a copy of the trial site's EC approval letter (stating at a minimum, the clinical trial name or identification number, protocol revision being approved and an approval date) and the informed consent prior to the initiation of enrollment at that center. If yearly approvals for the continuation of the trial at each trial site are required, they must also be forwarded to the Trial Sponsor.

#### 13.4 INVESTIGATOR RESPONSIBILITIES

### 13.4.1 GENERAL DUTIES

The investigator shall ensure that all work and services described herein, or incidental to those described herein, shall be conducted in accordance with the highest standards of medical and clinical research practice and the applicable regulations. The investigator shall be responsible for the day to day conduct of the clinical trial and for the safety and well-being of human subjects enrolled. The investigator will provide copies of the current clinical protocol to all staff responsible for conduct of the clinical trial.



The principal investigator is responsible for obtaining EC approval to start the clinical trial at his/her trial site.

If there is a change or addition of co-investigator, an amended Clinical Trial Agreement must be completed promptly.

#### 13.4.2 INVESTIGATOR RECORDS

The principal investigator will maintain accurate, complete, and current records relating to the site and their subjects participation in this clinical trial. Records including eCRF and supporting data, hardcopies of all blood and diagnostic exams, signed Clinical Trial Agreement, protocols and protocol amendments, signed informed consents, device tracking log and use of devices, EC approval letters, EC submissions, correspondence, including required reports and other documents pertaining to the conduct of the clinical trial must be kept on file by the investigator. If the investigator(s) wishes to assign the responsibility for maintaining files to someone else or remove them to another location, he/she should consult with the Trial Sponsor in writing as to this change. Files for the clinical trial must be maintained in a known location for a period in accordance with Edwards Lifesciences record retention requirements.

#### 13.4.3 INVESTIGATOR REPORTS

The principal investigator will prepare and submit the following accurate and complete reports to the Trial Sponsor and EC in a timely manner:

- Unanticipated serious adverse device effects (USADE) occurring during the clinical trial will be reported immediately (without any delay that could not be justified) after the principal investigator first learns of the event.
- Serious adverse device effects (SADE) occurring during the clinical trial will be reported as described in Section 11.1
- Deviation from the clinical protocol. Deviations to protect the subject's life or physical well-being in an emergency will be reported to the Trial Sponsor within 5 working days and the EC within their reporting policy.
- Use of devices without informed consent will be reported to the Trial Sponsor within 5 working days after the use occurs.
- A final written report is submitted to the Trial Sponsor and the EC within three months
  of completion or termination of the trial.
- Upon request by a reviewing EC or the pertinent regulatory agencies, the principal investigator will provide current information about any aspect of the trial.

#### 13.5 TRIAL SPONSOR RESPONSIBILITIES

#### 13.5.1 GENERAL DUTIES

As the sponsor of this clinical trial, Edwards Lifesciences has the overall responsibility for the conduct of the clinical trial, including assurance that the trial meets the regulatory requirements of the pertinent regulatory agencies. In this clinical trial, Edwards Lifesciences will have certain direct responsibilities and will delegate other responsibilities to an Echocardiography Core Laboratory.



## 13.5.2 SELECTION OF INVESTIGATORS

Edwards Lifesciences will select qualified investigators and will ship trial devices to participating trial sites only. Edwards Lifesciences will obtain signed investigator agreements and provide the Investigators with the information and supplies necessary to conduct the clinical trial.

#### 13.5.3 Monitoring the clinical trial

Edwards will ensure compliance with the signed investigator's agreement, the protocol (investigational plan), the requirements of applicable regulations and guidelines (see section 13.1), and any conditions of clinical trial approval by the EC and regulatory bodies per written monitoring procedures.

Edwards will conduct an immediate investigation of any unanticipated serious adverse device effects (USADE). If an event is found to present an unreasonable risk to subjects, participating in this clinical trial Edwards will inform investigators as required.

#### 13.5.4 Sponsor records

Edwards Clinical Research will maintain accurate, complete, and current records relating to this clinical trial. Records include eCRF, signed Investigator Agreement, financial disclosure, protocols and protocol amendments, signed informed consents, device use, EC approval letters, EC submissions, correspondence, including required reports, and other documents. Edwards will maintain documentation during the clinical trial and for a period of 100 years after the clinical trial is terminated or completed, or the records are no longer required to support a regulatory submission. Storage of the records may be designated to a third party.

#### 13.5.5 Sponsor reports

Edwards Clinical Research will prepare and submit the following accurate and complete reports to the EC and the pertinent regulatory agencies in a timely manner:

- Withdrawal of EC approval will be reported to all EC and the pertinent regulatory agencies within 5 working days of receipt of withdrawal of approval.
- Withdraw of the pertinent regulatory agencies approval will be reported to trial sites and EC within 5 working days after receiving the notice of approval withdrawal.
- Current investigator list will be submitted to the pertinent regulatory agencies at 6month intervals.
- Progress reports to the EC at least annually and to the pertinent regulatory agencies as required.
- A final written report is to be completed and submitted to the EC and the pertinent regulatory agencies within six months after completion or termination of the trial.
- Use of the devices without informed consent will be reported to regulatory authorities within 5 working days after notification of device use.
- Upon request by a reviewing EC or the pertinent regulatory agencies, Edwards will
  provide current information about any aspect of the trial.

#### 13.6 PUBLICATION POLICY

The publication of trial results will require prior approval and consent from the trial sponsor. Any analyses generated from the trial database for a manuscript will require review and approval by the trial sponsor prior to publication submission.



## 14 REFERENCES

- Rosenhek R, Binder R, Porenta G et al. Predictors of outcome in severe asymptomatic aortic stenosis. N Engl J Med 2000; 343(9): 611-7.
- Horstkotte D, Loogen F. The natural history of aortic valve stenosis. Eur Heart J Supp E 1998; 57-64.
- Carpentier A. Cardiac valve surgery. The French Correction. J Thorac Cardiovasc Surg 1983; 86: 323-37.
- 4. Carpentier A. Carpentier's Reconstructive Valve Surgery. Maryland Heights: Saunders, 2010.
- Craver JM. Aortic valve debridement by ultrasonic surgical aspirator: A word of caution. Ann Thorac Surg 1990; 49: 746-52.
- 6. Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2008 focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to revise the 1998 guidelines for the management of patients with valvular heart disease). Endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol 2008; 52(13):e1-142.

## 15 APPENDICES

Appendices could be updated independently from the Clinical Investigation Plan



# 15.1 ADVERSE EVENT (CODES AND DEFINITIONS)


Edwards

| | | AECODELIST |
|---|---|---|
| CODE | LABELINAME | DEFINITION |
| AE.1 | BLOOD AND LYMPHATIC (INCLUDING ALL BLEEDIN | G COMPLICATIONS) |
| AE101 | ANEMIA — NON-BLEEDING RELATED | A CONDITION IN WHICH RED BLOOD CELL COUNT AND/OR HEMOGLOBIN ARE LESS THAN NORMAL DUE TO LACK OF PRODUCTION OF RED BLOOD CELLS, AND THAT REQUIRES TREATMENT OR TRANSFUSION. |
| AE102 | ANEMIA – BLEEDING RELATED - MAJOR | A CONDITION IN WHICH RED BLOOD CELL COUNT AND/OR HEMOGLOBIN ARE LESS THAN NORMAL DUE TO BLOOD LOSS, AND THAT REQUIRES TREATMENT OR TRANSFUSION. |
| AE103 | ANEMIA — BLEEDING RELATED - MINOR | A CONDITION IN WHICH RED BLOOD CELL COUNT AND/OR HEMOGLOBIN ARE LESS THAN NORMAL DUE TO BLOOD LOSS, AND THAT REQUIRES TREATMENT OR TRANSFUSION. |
| AE104 | BLEEDING - CARDIOVASCULAR - MAJOR | ANY EPISODE OF MAJOR INTERNAL OR EXTERNAL BLEEDING THAT CAUSES DEATH, HOSPITALIZATION, OR PERMANENT INJURY (E.G., VISION LOSS) OR NECESSITATES TRANSFUSION. MAJOR BLEEDING UNEXPECTEDLY ASSOCIATED WITH MINOR TRAUMA SHOULD BE REPORTED AS A BLEEDING EVENT, BUT BLEEDING ASSOCIATED WITH MAJOR TRAUMA OR A MAJOR OPERATION (INCLUDING THE INDEX PROCEDURE) SHOULD NOT. THE LOCATION OF THE BLEEDING (GASTROINTESTINAL, GENITOURINARY, ETC.) MUST BE REPORTED. FOR EACH REPORTED BLEEDING EVENT, INDICATE IF SUBJECT IS TAKING ANTICOAGULANTS OR ANTI-PLATELET AGENTS. |
| AE105 | BLEEDING - CARDIOVASCULAR - MINOR | |
| AE106 | BLEEDING - GENITOURINARY - MAJOR | |
| AE107 | BLEEDING - GENITOURINARY - MINOR | The state of the s |
| AE108 | BLEEDING - GASTROINTESTINAL UPPER -MAJOR | |
| AE109 | BLEEDING - GASTROINTESTINAL UPPER -MINOR | |
| AE110 | BLEEDING - GASTROINTESTINAL LOWER -MAJOR | |
| AE111 | BLEEDING - GASTROINTESTINAL LOWER -MINOR | |
| AE112 | BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL -MAJOR | " (E.G. ECCHYMOSIS) |
| AE113 | BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL -MINOR | " (E.G. ECCHYMOSIS) |
| AE114 | BLEEDING - NEUROLOGICAL - MAJOR | " (E.G. CEREBRAL VASCULAR ACCIDENT) |
| AE115 | BLEEDING - NEUROLOGICAL - MINOR | " (E.G. CEREBRAL VASCULAR ACCIDENT) |
| AE116 | BLEEDING - PERIPHERAL VASCULAR -MAJOR | " (E.G. NOSEBLEEDS; HEMATOMAS) |
| AE117 | BLEEDING - PERIPHERAL VASCULAR - MINOR | " (E.G. NOSEBLEEDS; HEMATOMAS) |
| AE118 | BLEEDING - PULMONARY/RESPIRATORY - MAJOR | " (E.G. HEMOTHORAX) |
| AE119 | BLEEDING - PULMONARY/RESPIRATORY MINOR | " (E.G. HEMOTHORAX) |
| AE120 | BLOOD SEPSIS | POSITIVE BLOOD CULTURE AND CLINICAL EVIDENCE OF INFECTION (E.G. FEVER, ELEVATED WBC COUNT, HYPOTENSION, END ORGAN DYSFUNCTION) EVENT MUST BE CONFIRMED BY 2 CONSECUTIVE POSITIVE BLOOD CULTURES, EXPLANT OR AUTOPSY. |

CONFIDENTIAL AND PROPRIETATARY DATA: THIS DOCUMENT AND THE INFORMATION CONTAINED HEREIN MAY NOT BE REPRODUCED, USED, OR DISCLOSED WITHOUT WRITTEN PERMISSION FROM EDWARDS LIFESCIENCES LLC  



| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.1 | BLOOD AND LYMPHATIC (INCLUDING ALL BLEEDING | NG COMPLICATIONS) (CONTINUED) |
| AE122 | HEMOLYSIS WITHOUT PARAVALVULAR LEAK | PLASMA -FREE HEMOGLOBIN > 40 MG/DL ON TWO CONSECUTIVE MEASUREMENTS WITHIN 48 HOURS; OR CLINICAL DIAGNOSIS OF HEMOLYSIS EVIDENCED BY LABORATORY TESTING SUCH AS SERUM HEMOGLOBIN, HEMATOCRIT, AND/OR PLASMA-FREE HEMOGLOBIN (NOT IMMUNOLOGICALLY BASED) |
| AE123 | DISSEMINATED INTRAVASCULAR COAGULATION (DIC) | DIFFUSE, NONSURGICAL, MICROVASCULAR HEMORRHAGE AND/OR THROMBOSES. |
| AE124 | THROMBOCYTOPENIA - HEPARIN INDUCED (HIT) | THROMBOCYTOPENIA (<150,000 PER CUBIC MILLIMETER), OR A RELATIVE DECREASE OF 50 PERCENT OR MORE FROM BASELINE, OR NEW THROMBOSIS IN A SUBJECT RECEIVING HEPARIN OR LIMMH; CONFIRMED BY SEROLOGIC TESTING FOR PF4—HEPARIN ANTIBODIES. |
| AE125 | THROMBOCYTOPENIA - NON-HEPARIN INDUCED | THROMBOCYTOPENIA (<150,000 PER CUBIC MILLIMETER), OR A RELATIVE DECREASE OF 50 PERCENT OR MORE FROM BASELINE, ACCOMPANIED BY A LOW INDEX OF SUSPICION FOR HIT (I.E., NOT ASSOCIATED WITH HEPARIN USE, THE PRESENCE OF OTHER CAUSES OF THROMBOCYTOPENIA, SUCH AS DRUGS OTHER THAN HEPARIN, DIC OR OTHER CONSUMPTIVE PROCESSES, POST-TRANSFUSION PURPURA). |
| AE126 | BLOOD/LYMPHATIC - OTHER | OTHER BLOOD OR LYMPHATIC EVENT THAT DOES NOT FIT IN ONE OF THE OTHER "BLOOD" CATEGORIES THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.2 | CARDIOVASCULAR - ARRHYTHMIA | |
| AE158 | ARRHYTHMIA - PERMANENT ATRIAL FIBRILLATION | AN ABNORMAL HEARTBEAT IN WHICH THE HEART RHYTHM IS FAST AND IRREGULARLY IRREGULAR. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. AF IS CONSIDERED PERMANENT WHEN IT HAS PERSISTED BEYOND 1 YEAR AND ATTEMPTS AT CARDIOVERSION HAVE FAILED OR COULD NOT BE ATTEMPTED. |
| AE149 | ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) | AN ABNORMAL HEARTBEAT IN WHICH THE HEART RHYTHM IS FAST AND IRREGULARLY IRREGULAR, EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. AF IS CONSIDERED PARCXYSMAL WHEN EPISODES OF AF TERMINATE SPONTANEOUSLY WITHIN 7 DAYS (MOST EPISODES LAST LESS THAN 24 HOURS) |
| AE157 | ARRHYTHMIA - PERSISTENT ATRIAL FIBRILLATION | AN ABNORMAL HEARTBEAT IN WHICH THE HEART RHYTHM IS FAST AND IRREGULARLY IRREGULAR. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. AF IS CONSIDERED PERSISTENT WHEN EPISODES OF AF LAST MORE THAN 7 DAYS AND MAY REQUIRE EITHER PHARMACOLOGIC OR ELECTRICAL INTERVENTION TO TERMINATE |
| AE141 | ARRHYTHMIA - ATRIAL FLUTTER | WELL ORGANIZED BUT OVERLY RAPID CONTRACTIONS OF HEART ATRIUM (USUALLY AT A RATE OF 250-350 CONTRACTIONS PER MINUTE). EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE142 | ARRHYTHMIA - AV BLOCK - 1ST DEGREE | AV BLOCK I: A CONDUCTION DISORDER OF NERVOUS IMPULSE AT THE LEVEL OF THE ATRIOVENTRICULAR JUNCTION, I.E. BETWEEN ATRIUM AND VENTRICLE. |
| AE143 | ARRHYTHMIA - AV BLOCK - 2ND DEGREE | " AV BLOCK II: THERE ARE TWO TYPES: MOBITZ I PROGRESSIVE PROLONGATION OF PR INTERVAL WITH DROPPED BEATS (THE PR INTERVAL GETS LONGER AND LONGER; FINALLY ONE BEAT DROPS) MOBITZ II PR INTERVAL REMAINS UNCHANGED PRIOR TO THE P-WAVE WHICH SUDDENLY FAILS TO CONDUCT TO THE VENTRICLES; |
| AE144 | ARRHYTHMIA - AV BLOCK - 3RD DEGREE | " AV BLOCK III: , NO P-WAVES CONDUCT TO THE VENTRICLE AND AV DISSOCIATION IS COMPLETE. ANY LEVEL OF AV BLOCK EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |

Edwards

| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE145 | ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT | BUNDLE BRANCH BLOCK IS AN INTRAVENTRICULAR CONDUCTION DEFECT (IVCD) THAT DISRUPTS THE NORMAL FLOW OF ELECTRICAL IMPULSES THAT RESULT IN A NORMAL HEART BEAT. QRS DURATION OF GREATER THAN 110 MILLISECONDS IS A DIAGNOSTIC INDICATION OF BBB. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE.2 | CARDIOVASCULAR - ARRHYTHMIA (CONTINUED) | |
| AE146 | ARRHYTHMIA - BUNDLE BRANCH BLOCK - RIGHT | = |
| AE147 | ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (SVT) | SUSTAINED TACHYARRHYTHMIA IN WHICH THE QRS APPEARS NORMAL AND HAS DURATION OF < 120 MSEC. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE148 | ARRHYTHMIA - PAROXYSMAL ATRIAL TACHYCARDIA (PAT) | A RAPID HEART RHYTHM ORIGINATING ABOVE THE VENTRICULAR TISSUE DUE TO AV NODAL REENTRANT TACHYCARDIA. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE150 | ARRHYTHMIA - VENTRICULAR FIBRILLATION | A RAPID IRREGULAR VENTRICULAR RHYTHM DUE TO MULTIPLE REENTRANT ACTIVITIES ASSOCIATED WITH ESSENTIALLY ZERO CARDIAC OUTPUT. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE151 | ARRHYTHMIA - TACHYCARDIA - VENTRICULAR | AN ABNORMALLY FAST HEART RATE (TYPICALLY DEFINED AS > 100 BPM IN ADULTS) WHICH MAY REQUIRE IMPLANT OF A PACEMAKER TO MAINTAIN A NORMAL HEART RATE. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. VENTRICULAR TACHYCARDIA: DEFINED AS A REGULAR HEART RHYTHM ORIGINATING FROM THE VENTRICLE WITH A FREQUENCY OF 160 TO 200 BEATS PER MINUTE. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE152 | ARRHYTHMIA - TACHYCARDIA - NON-VENTRICULAR | ASSUMED" |
| AE153 | ARRHYTHMIA - BRADYCARDIA | AN ABNORMALLY SLOW HEART RATE (TYPICALLY DEFINED AS <60 BPM IN ADULTS) EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE154 | ARRHYTHMIA - TACHY-BRADYCARDIA | A VARIANT OF SICK SINUS SYNDROME IN WHICH SLOW ARRHYTHMIAS AND FAST ARRHYTHMIAS ALTERNATE. EVENT SHOULD BE DOCUMENTED AND CONFIRMED BY ECG TEST RESULTS. |
| AE155 | ARRHYTHMIA - PACEMAKER/ICD MALFUNCTION | PACEMAKER/ICD DOES NOT FUNCTION AS INTENDED. |
| AE156 | ARRHYTHMIA - OTHER | ARRHYTHMIA THAT IS NOT COVERED BY ANY OF THE DEFINITIONS ABOVE. PLEASE SPECIFY |
| AE.3 | CARDIOVASCULAR - REGURGITATION | |
| | IF THE VALVE INVOLVED IS THE STUDY VALVE, THEN THIS DEFINITION SHOULD DYSFUNCTION (AS APPROPRIATE) REGURGITATION, AORTIC: ALSO KNOWN AS ACT VENTRICULAR FORWARD STROKE VOLUME RETURNS TO THE CHAMBER DURING DI UNDER NON-STRUCTURAL VALVE DYSFUNCTION. REGURGITATION, CENTRAL: OC BACK INTO THE HEART. REGURGITATION, INDETERMINATE: OCCURS WHEN BLOX REGURGITATION, MITRAL: ALSO KNOWN AS MITRAL INCOMPETENCE AND MITRAL IN LEFT VENTRICLE CONTRACTS. DIAGNOSED BY AUSCULTATION (MURMUR) OR ECHIBLE WOOD FLOW FROM THE RIGHT VENTRICLE TO THE RIGHT ATRIUM DURING SYSTOLE. | IF THE VALVE INVOLVED IS THE STUDY VALVE, THEN THIS DEFINITION SHOULD BE USED, BUT THE EVENT SHOULD BE REPORTED AS STRUCTURAL OR NON-STRUCTURAL VALVE DYSFUNCTION (AS APPROPRIATE) REGURGITATION, AORTIC: ALSO KNOWN AS AORTIC INSUFFICIENCY AND INCOMPETENCE OF THE AORTIC VALVE, IN WHICH SHOULD BE CAPTURED VENTED TO THE CHAMBER DURING DIASTOLE. THIS CATEGORY DOES NOT INCLUDE PARAVALVULAR LEAK, WHICH SHOULD BE CAPTURED BUNDER NON-STRUCTURAL VALVE DYSFUNCTION. REGURGITATION, CENTRAL: OCCURS WHEN THE VALVE LEAFLETS DO NOT COMPLETELY CLOSE AND ALLOW SOME BLOOD TO LEAK BACK INTO THE HEART AND CANNOT BE CATEGORIZED BY LOCATION AND OR SEVERITY. REGURGITATION, MITRAL: ALSO KNOWN AS MITRAL INCOMPETENCE AND MITRAL INSUFFICIENCY IN WHICH THE BLOOD FLOWS BACKWARDS THROUGH THE MITRAL VALVE EACH TIME THE LEFT VENTRICLE CONTRACTS. DIAGNOSED BY AUSCULTATION (MURMUR) OR ECHOCARDIOGRAPHY. REGURGITATION, TRICUSPID: INSUFFICIENCY OF THE TRICUSPID VALVE CAUSING BLOOD FLOW FROM THE RIGHT VENTRICLE TO THE RIGHT ATRIUM DURING SYSTOLE. |
| AE160 | REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+1 | TRIVIAL/TRACE |
| AE161 | REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+2 | MILD |

CONFIDENTIAL AND PROPRIETATARY DATA: THIS DOCUMENT AND THE INFORMATION CONTAINED HEREIN MAY NOT BE REPRODUCED, USED, OR DISCLOSED WITHOUT WRITTEN PERMISSION FROM EDWARDS LIFESCIENCES LLC  





AE CODE LIST TRIVIAL/TRACE TRIVIAL/TRACE TRIVIAL/TRACE TRIVIAL/TRACE TRIVIAL/TRACE TRIVIAL/TRACE DEFINITION MODERATE MODERATE MODERATE MODERATE MODERATE MODERATE MODERATE SEVERE SEVERE SEVERE SEVERE SEVERE SEVERE SEVERE MLD MILD Q W MICO MILD MILD REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+3 REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+4 REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+2 REGURGITATION - PULMONARY-CENTRAL/TRANSVALVULAR-+1 CARDIOVASCULAR - REGURGITATION (CONTINUED) REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+1 REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+2 REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+3 REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR-+4 REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+3 REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+4 REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+2 REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+3 REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+4 REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR-+1 REGURGITATION - PULMONARY-INDETERMINATE-+3 REGURGITATION - PULMONARY-INDETERMINATE-+2 REGURGITATION - PULMONARY-INDETERMINATE-+4 REGURGITATION - PULMONARY-INDETERMINATE-+1 REGURGITATION - AORTIC-INDETERMINATE-+2 REGURGITATION - AORTIC-INDETERMINATE-+3 REGURGITATION - MITRAL-INDETERMINATE-+2 REGURGITATION - MITRAL-INDETERMINATE-+3 REGURGITATION - AORTIC-INDETERMINATE-+4 REGURGITATION - MITRAL-INDETERMINATE-+1 REGURGITATION - MITRAL-INDETERMINATE-+4 REGURGITATION - AORTIC-INDETERMINATE-+1 LABEL/NAME CODE AE170 AE181 AE183 AE190 AE193 AE199 AE202 AE203 **AE204** AE205 AE162 AE163 AE168 AE171 AE172 AE173 AE174 AE182 AE192 AE198 AE169 AE175 AE180 AE200 AE201 AE.3 AE191



Clinical Investigational Plan Protocol Number: 2010-03

| | | AE CODE LIST |
|---|---|---|
| CODE | LABEUNAME | DEFINITION |
| AE210 | REGURGITATION - TRICUSPID-INDETERMINATE-+1 | TRIVIAL/TRACE |
| AE211 | REGURGITATION - TRICUSPID-INDETERMINATE-+2 | MILD |
| AE212 | REGURGITATION - TRICUSPID-INDETERMINATE-+3 | MODERATE |
| AE213 | REGURGITATION - TRICUSPID-INDETERMINATE-+4 | SEVERE |
| AE.5 | CARDIOVASCULAR - STENOSIS | *IF THE VALVE INVOLVED IS THE STUDY VALVE, THEN THIS DEFINITION SHOULD BE USED, BUT THE EVENT SHOULD BE REPORTED AS STRUCTURAL OR NON-STRUCTURAL VALVE DYSFUNCTION (AS APPROPRIATE) |
| AE220* | STENOSIS - AORTIC - MILD | AORTIC: FLOW OBSTRUCTION OF THE AORTIC VALVE DUE TO RESTRICTED LEAFLET OPENING. THE SEVERITY IS CATEGORIZED AS: MILD - JET VELOCITY (M/S) <3.0; MEAN GRADIENT (MMHG) <25; VALVE AREA (CMZ) >1.5. OR SEVERE - JET VELOCITY (M/S) 3.0-4.0; MEAN GRADIENT (MMHG) 25-40; VALVE AREA (CMZ) 1.0-1.5. OR SEVERE - JET VELOCITY (M/S) >-4.0; MEAN GRADIENT (MMHG) >-40; VALVE AREA (CMZ) 1.0-1.5. OR SEVERE - JET VELOCITY (M/S) >-4.0; MEAN GRADIENT (MMHG) >-40; VALVE AREA (CMZ) -1.0; VALVE AREA (INDEX<0.6. MITRAL: MITRAL: MITRAL STENOSIS (MS) REFERS TO NARROWING OF THE MITRAL VALVE ORFICE, RESULTING IN IMPEDANCE OF FILLING OF THE LETT VENTRICLE IN DIASTOLE. THE SEVERITY OF MS IS CATEGORIZED AS: MILD - MEAN GRADIENT (MM HG) > 45, PULMONARY ARTERY SYSTOLIC PRESSURE (MM HG) > 40, VALVE AREA (CMZ) >-1.5. MODERATE - MEAN GRADIENT (MM HG) > 10, PULMONARY ARTERY SYSTOLIC PRESSURE (MM HG) >-50, VALVE AREA (CMZ) <-1.0. TRICUSPID: A NARROWING OF THE TRICUSPID VALVE OPENING THAT INCREASES RESISTANCE TO BLOOD FLOW FROM THE RIGHT ATRIUM TO THE RIGHT VENTRICLE. SEVERE TRICUSPID STENOSIS IS DEFINED AS A VALVE AREA LESS THAN 1.0 CMZ. |
| AE221* | STENOSIS - AORTIC - MODERATE | |
| AE222* | STENOSIS - AORTIC - SEVERE | |
| AE223 | STENOSIS - MITRAL- MILD | |
| AE224 | STENOSIS - MITRAL - MODERATE | |
| AE225 | STENOSIS - MITRAL - SEVERE | |
| AE226 | STENOSIS - PULMONARY- MILD | |
| AE227 | STENOSIS - PULMONARY - MODERATE | |
| AE228 | STENOSIS - PULMONARY - SEVERE | |
| AE229 | STENOSIS - TRICUSPID- MILD | |
| AE230 | STENOSIS - TRICUSPID- MODERATE | |
| AE231 | STENOSIS - TRICUSPID - SEVERE | |



| | | AECODELIST |
|---|---|---|
| CODE | LABEUNAME | DEFINITION |
| AE.6 | CARDIOVASCULAR - THROMBOEMBOLIC<br>EVENT/VALVE THROMBOSIS | ANY EMBOLIC EVENT THAT OCCURS IN THE ABSENCE OF INFECTION AFTER THE IMMEDIATE PERIOPERATIVE PERIOD AND MAY BE MANIFESTED BY A NEUROLOGIC EVENT OR A NON-CEREBRAL EMBOLIC EVENT. EMBOLI CONSISTING OF NON-THROMBOTIC MATERIAL (E.G., ATHEROSCLEROSIS, MYXOMA) ARE NOT COUNTED. |
| AE250 | THROMBOEMBOLIC EVENT - STROKE | INCLUDES ANY CENTRAL, NEW NEUROLOGIC DEFICIT, WHETHER TEMPORARY OR PERMANIBIT AND WHETHER FOCAL OR GLOBAL, THAT OCCURS AFTER THE SUBJECT EMERGES FROM ANESTHESIA. POSTOPERATIVE NEUROLOGIC SYMPTOMS THAT OCCURS AFTER THE SUBJECT EMERGES FROM ANESTHESIA. POSTOPERATIVE NEUROLOGIC EVENT AND THAT ARE CONFIRMED RADIOGRAPHICALLY TO BE CONSISTENT WITH THE FORMER EVENT ARE NOT COUNTED. CENTRAL NEUROLOGIC EVENTS THAT ARE CLEARLY RELATED TO AORTIC, INTERNAL CAROTID ARTERY, OR VERTEBRAL ARTERY DISEASE ARE ALSO NOT COUNTED. PSYCHOMOTOR DEFICITS FOUND BY SPECIALIZED TESTING ARE NOT CONSIDERED NEUROLOGIC EVENTS. STROKE: A PROLONGED (>72 HOURS) OR PERMANENT NEUROLOGIC DEFICIT THAT IS USUALLY ASSOCIATED WITH ABNORMAL RESULTS OF MRI OR CT SCANS. SUBJECTS WITH MINIMAL, ATYPICAL, OR PROTEAN SYMPTOMS THAT LEAD TO RADIOGRAPHIC IMAGING DIMONSTRATING AN ACUTE ISCHEMIC EVENT ARE CONSIDERED TO HAVE SUSTAINED A STROKE. TIA: CHARACTERIZED BY FULLY REVERSIBLE SYMPTOMS OF SHORT DURATION. IF RADIOGRAPHIC IMAGING DEMONSTRATES AN ACUTE CENTRAL NEUROLOGIC LESION, HOWEVER, SUCH SUBJECTS ARE RECLASSIFIED AS HAVING SUSTAINED A STROKE. |
| AE255 | THROMBOEMBOLIC EVENT — TRANSIENT ISCHEMIC ATTACK (TIA) | INCLUDES ANY CENTRAL, NEW NEUROLOGIC DEFICIT, WHETHER TEMPORARY OR PERMANIENT AND WHETHER FOCAL OR GLOBAL, THAT OCCURS AFTER THE SUBJECT EMERGES FROM ANESTHESIA. POSTOPERATIVE NEUROLOGIC SYMPTOMS THAT OCCURS AFTER THE SUBJECT EMERGES FROM ANESTHESIA. POSTOPERATIVE NEUROLOGIC SYMPTOMS THAT MINIED THAT ARE CONSIDERED TO THAT ARE CLEARLY TO BE CONSISTENT WITH THE FORMER EVENT ARE NOT COUNTED. CENTRAL NEUROLOGIC EVENTS THAT ARE CLEARLY RELATED TO AORTIC, INTERNAL CAROTID ARTERY OR VERTEBRAL ARTERY DISEASE ARE ALSO NOT COUNTED. PSYCHOMOTOR DEFICITS FOUND BY SPECIALIZED TESTING ARE NOT CONSIDERED NEUROLOGIC EVENTS. STROKE: A PROLONGED (>72 HOURS) OR PERMANENT NEUROLOGIC DEFICIT THAT IS USUALLY ASSOCIATED WITH ABNORMAL RESULTS OF MRI OR CT SCANS. SUBJECTS WITH MINIMAL, ATYPICAL, OR PROTEAN SYMPTOMS THAT LEAD TO RADIOGRAPHIC IMAGING DEMONSTRATING AN ACUTE ISCHEMIC EVENT ARE CONSIDERED TO HAVE SUSTAINED A STROKE. TIA: CHARACTERIZED BY FULLY REVERSIBLE SYMPTOMS OF SHORT DURATION. IF RADIOGRAPHIC IMAGING DEMONSTRATES AN ACUTE CENTRAL NEUROLOGIC LESION, HOWEVER, SUCH SUBJECTS ARE RECLASSIFIED AS HAVING SUSTAINED A STROKE. |
| AE256 | THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL NO PARESIS | A PERIPHERAL EMBOLIC EVENT IS AN OPERATIVE, AUTOPSY, OR CLINICALLY DOCUMENTED EMBOLUS THAT PRODUCES SYMPTOMS FROM COMPLETE OR PARTIAL OBSTRUCTION OF A PERIPHERAL (NON-CEREBRAL) ARTERY. LOCATION SHOULD BE REPORTED. REPORT UNDER PULMONARY EMBOLISM IF EVENT OCCURS IN THE LUNG. |
| AE257 | THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL | " HEMIPARESIS |
| AE258 | THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL THROMBOEMBOLIC EVENT - OTHER - CENTRAL | "FULL PARESIS "NO PARESIS |
| | INORDERMENT CALL CALLES | 253161.02 |

CONFIDENTIAL AND PROPRIETATARY DATA: THIS DOCUMENT AND THE INFORMATION CONTAINED HEREIN MAY NOT BE REPRODUCED, USED, OR DISCLOSED WITHOUT WRITTEN PERMISSION FROM EDWARDS LIFESCIENCES LLC 

Edwards

| | 000000 | |
|---|---|---|
| | | AECODELIST |
| CODE | LABEL/NAME | DEFINITION |
| AE260 | THROMBOEMBOLIC EVENT - OTHER - CENTRAL | " HEMIPARESIS |
| AE.6 | CARDIOVASCULAR - THROMBOEMBOLIC EVENT/VALVE THROMBOSIS (CONTINUED) | LVE THROMBOSIS (continued) |
| AE261 | THROMBOEMBOLIC EVENT - OTHER - CENTRAL | " FULL PARESIS |
| AE262 | VALVE THROMBOSIS - AORTIC | ANY THROMBUS NOT CAUSED BY INFECTION ATTACHED TO OR NEAR AN OPERATED VALVE THAT OCCLUDES PART OF THE BLOOD FLOW PATH, INTERFERES WITH VALVE FUNCTION, OR IS SUFFICIENTLY LARGE TO WARRANT TREATMENT. VALVE THROMBUS FOUND AT AUTOPSY IN A SUBJECT WHOSE CAUSE OF DEATH WAS NOT VALVE RELATED OR FOUND AT OPERATION FOR AN UNRELATED INDICATION SHOULD ALSO BE COUNTED. |
| AE263 | VALVE THROMBOSIS - MITRAL | II . |
| AE264 | VALVE THROMBOSIS - PULMONARY | = |
| AE265 | VALVE THROMBOSIS - TRICUSPID | II. |
| AE.7 | CARDIOVASCULAR - MISC | |
| AE270 | ANGINA, STABLE | CHEST PAIN, TIGHT OR HEAVY FEELING IN THE CHEST, OR DISCOMFORT WHICH SPREADS FROM THE CHEST TO THE ARM, BACK, NECK, JAW, OR STOMACH, NUMBNESS OR TINGLING IN THE SHOULDERS, ARMS OR WRISTS, SHORTNESS OF BREATH, AND NAUSEA RELIEVED BY REST OR NITROGLYCERINE AND/OR CONFIRMED BY ECG. STABLE ANGINA IS ANGINA THAT IS CONTROLLED BY ORAL AND/OR TRANSCUTANEOUS MEDICATION. |
| AE271 | ANGINA, UNSTABLE | UNSTABLE ANGINA IS ANGINA, WHICH NECESSITATES THE INITIATION, CONTINUATION OR INCREASE OF ANGINA CONTROL THERAPIES THAT MAY INCLUDE: NITROGLYCERIN DRIP, HEPARIN DRIP, OR IABP PLACEMENT. THE TYPE OF ANGINA MAY INCLUDE, BUT IS NOT LIMITED TO: REST ANGINA, NEW ONSET EXERTIONAL ANGINA OF AT LEAST NEW YORK HEART ASSOCIATION (NYHA) CLASS III IN SEVERITY, RECENT ACCELERATION IN PATTERN AND INCREASE OF ONE NYHA CLASS TO AT LEAST NYHA CLASS III, VARIANT ANGINA, NON-Q WAVE MYOCARDIAL INFARCTION, OR POST-INFARCTION ANGINA. |
| AE272 | ANNULAR DISSECTION | DISSECTION OF THE VALVULAR ANNULUS EXTENDING INTO THE AORTA. ANNULAR DISSECTION OCCURRING WITHIN 30 DAYS OF THE INDEX PROCEDURE WILL BE CONSIDERED VALVE RELATED. SHOULD BE CONFIRMED BY IMAGING, OR DIRECT VISUAL INSPECTION. |
| AE273 | AORTIC DISSECTION | DISRUPTION OF THE MEDIA LAYER OF THE AORTA WITH BLEEDING WITHIN AND ALONG THE WALL OF THE AORTA. AORTIC DISSECTION MAY OCCUR IN THE ASCENDING THORACIC AORTA (TYPE A DISSECTION) OR IN THE DESCENDING THORACIC AORTA (TYPE B DISSECTION). DISSECTION SHOULD BE CONFIRMED BY IMAGING OR DIRECT VISUAL INSPECTION. |
| AE274 | ARTERIAL DISSECTION | DISRUPTION OF THE MEDIA LAYER OF AN ARTERY OTHER THAN THE AORTA WITH BLEEDING WITHIN AND ALONG THE WALL OF THE VESSEL. SHOULD BE CONFIRMED BY IMAGING OR DIRECT VISUAL INSPECTION. |
| AE275 | CARDIAC ARREST | CARDIAC ARREST DOCUMENTED BY ONE OF THE FOLLOWING: VENTRICULAR FIBRILLATION, RAPID VENTRICULAR TACHYCARDIA WITH HEMODYNAMIC INSTABILITY, ASYSTOLE. |
| AE276 | CARDIAC DECOMPENSATION | AN INABILITY OF THE HEART TO MAINTAIN ADEQUATE CIRCULATION; IT IS MARKED BY DYSPNEA, VENOUS ENGORGEMENT, CYANOSIS AND EDEMA. |



Clinical Investigational Plan Protocol Number: 2010-03

| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE277 | CARDIOGENIC SHOCK | A CLINICAL STATE OF HYPOPERFUSION SUSTAINED FOR GREATER THAN 30 MINUTES, WITH EITHER SYSTOLIC BLOOD PRESSURE < 80 MM HG, AND /OR CARDIAC INDEX < 1.8 DESPITE MAXIMAL TREATMENT (FLUIDS) OR REQUIRING INTRAVENOUS INOTROPES AND/OR PRESSOR AGENT OR AN INTRA-AORTIC BALLOON PUMP (IABP). |
| AE.7 | CARDIOVASCULAR - MISC (CONTINUED) | |
| AE278 | CHORDAE TENDINEAE DAMAGE | |
| AE279 | CORONARY ARTERY OSTIAL OBSTRUCTION | OBSTRUCTION OF THE CORONARY OSTIA. SHOULD BE CONFIRMED BY IMAGING AND THE SOURCE OF THE OBSTRUCTION (AORTIC VALVE, THROMBUS, ETC. SHOULD BE REPORTED. |
| AE280 | ENDOCARDITIS | ANY INFECTION INVOLVING THE STUDY VALVE. THE DIAGNOSIS OF OPERATED VALVULAR ENDOCARDITIS IS BASED ON ONE OF THE FOLLOWING CRITERIA: (1) REOPERATION WITH EVIDENCE OF ABSCESS, PARAVALVULAR LEAK, PUS, OR VEGETATION CONFIRMED AS SECONDARY TO INFECTION WITH EVIDENCE OR MICROBIOLOGIC STUDIES; (2) AUTOPSY FINDINGS OF ABSCESS, PUS, OR VEGETATION INVOLVING A REPAIRED OR REPLACED VALVE; OR (3) IN THE ABSENCE OF REOPERATION OR AUTOPSY, MEETING OF THE DUKE CRITERIA FOR ENDOCARDITIS [4]. MORBIDITIES ASSOCIATED WITH ACTIVE INFECTION, SUCH AS VALVE THROMBOSIS, THROMBOTIC EMBOLUS, BLEEDING EVENT, OR PARAVALVULAR LEAK, ARE INCLUDED UNDER THIS CATEGORY, BUT NOT COUNTED IN OTHER CATEGORIES OF MORBIDITY. |
| AE281 | HEART FAILURE — ACUTE | ACUTE HEART FAILURE DESCRIBES EXACERBATED OR DECOMPENSATED HEART FAILURE, REFERRING TO EPISODES IN WHICH A SUBJECT IS CHARACTERIZED AS HAVING A CHANGE IN HEART FAILURE SIGNS AND SYMPTOMS RESULTING IN A NEED FOR URGENT THERAPY OR HOSPITALIZATION. |
| AE282 | HEART FAILURE CHRONIC (CHF) | AN EVENT IN WHICH THE HEART FALS TO MEET THE CIRCULATORY REQUIREMENTS OF THE BODY UNDER DIFFERING PHYSIOLOGICAL CIRCUMSTANCES, AND/OR A STATE IN WHICH CARDIAC OUTPUT IS REDUCED RELATIVE TO THE DEMANDS OF THE BODY, ASSUMING THE EVIDENCE OF ADEQUATE VENOUS RETURN. EVENT IS CONFIRMED CLINICALLY OR BY DIAGNOSTIC TESTING. |
| AE283 | HYPERTENSION — SYSTEMIC | DEFINED AS BLOOD PRESSURE > 140/90 MM HG FOR SUBJECT WITHOUT DIABETES OR KIDNEY DISEASE; > 130/80 MMHG FOR SUBJECTS ON 2 OCCASIONS WITH DIABETES OR RENAL DISEASE. UNLESS DUE TO PRESENCE OF MEDICATION, E.G. BETA BLOCKERS FOR 10 YEARS |
| AE284 | HYPERTENSION - PULMONARY | MEAN PULMONARY ARTERY PRESSURE THAT IS GREATER THAN 25 MMHG AT REST AND/OR GREATER THAN 30 MMHG DURING EXERCISE CONFIRMED BY SWAN GANZ CATHETER OR DIAGNOSTIC PLACEMENT IN THE PULMONARY ARTERY BED AND CONDITION REQUIRES MEDICAL INTERVENTION TO RESOLVE OR TREAT THE CONDITION. |
| AE285 | HYPOTENSION | ABNORMALLY LOW BLOOD PRESSURE. FOR AN ADULT, HYPOTENSION IS DEFINED AS BLOOD PRESSURE LESS THAN 90/50 MMHG. |



| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.7 | CARDIOVASCULAR - MISC (CONTINUED) | |
| AE286 | MYOCARDIAL INFARCTION | AN ACUTE MYOCARDIAL INFARCTION IS EVIDENCED BY ANY OF THE FOLLOWING: 1. A RISE AND FALL OF CARDIAC BIOMARKERS (PREFERABLY TROPONIN) WITH AT LEAST ONE OF THE VALUES IN THE ABNORMAL RANGE (CK ≥ 5X ULN) TOGETHER WITH AT LEAST ONE OF THE FOLLOWING MANIFESTATIONS OF MYOCARDIAL ISCHEMIA: A) ISCHEMIC SYMPTOMS; B) ECG CHANGES INDICATIVE OF NEW ISCHEMIA (NEW ST-T CHANGES, NEW LEFT BUNDLE BRANCH BLOCK, OR LOSS OF R WAVE VOLTAGE); C) DEVELOPMENT OF PATHOLOGICAL Q WAVES IN 2 OR MORE CONTIGUOUS LEADS IN THE ECG (OR EQUIVALENT FINDINGS FOR TRUE POSTERIOR MI); D. IMAGING EVIDENCE OF NEW LOSS OF VIABLE MYOCARDIUM OR NEW REGIONAL WALL MOTION ABNORMALITY. 2. DEVELOPMENT OF NEW PATHOLOGICAL Q WAVES IN 2 OR MORE CONTIGUOUS LEADS IN THE ECG, WITH OR REGIONAL WALL MOTION ABNORMALITY. 3. IMAGING EVIDENCE OF A REGION WITH NEW LOSS OF VIABLE MYOCARDIUM AT REST IN THE ABSENCE OF A NON-ISCHEMIC CAUSE. THIS CAN BE MANIFEST AS: A. ECHOCARDIOGRAPHIC, CT, MR, VENTRICULOGRAPHIC OR NUCLEAR IMAGING EVIDENCE OF LEFT VENTRICULAR THINNING OR SCARRING AND FAILURE TO CONTRACT APPROPRIATELY (I.E., HYPOKINESIS, OR DYSKINESIS); OR, B. FIXED (NON-REVERSIBLE) PERFUSION DEFECTS ON NUCLEAR RADIOISOTOPE IMAGING (E.G., MIB), THALLIUM). |
| AE287 | MYOCARDITIS | AN INFECTION OF THE HEART MUSCLE |
| AE296 | PERFORATION - ATRIAL | AN ABNORMAL HOLE OR OPENING IN THE ATRIAL WALL CAUSED BY A DEVICE CAUSING PUNCTURE THROUGH THE WALL OR BY PRESSURE AGAINST A WEAKENED PORTION OF THE WALL. |
| AE297 | PERFORATION - VENTRICULAR | AN ABNORMAL HOLE OR OPENING IN THE VENTRICULAR WALL CAUSED BY A DEVICE CAUSING PUNCTURE THROUGH THE WALL. |
| AE289 | PERFORATION - OTHER | The state of the s |
| AE290 | PERICARDIAL EFFUSION - MAJOR | EXCESS FLUID ACCUMULATION IN THE PERICARDIAL SPACE THAT INTERFERES WITH NORMAL HEART FUNCTION AND REQUIRES MEDICAL INTERVENTION TO RESOLVE. IT SHOULD BE CONFIRMED BY ECHOCARDIOGRAPHY OR CT. |
| AE291 | PERICARDIAL EFFUSION - MINOR | |
| AE292 | PERICARDIAL TAMPONADE - MAJOR | ABNORMAL FLUID ACCUMULATION WITHIN THE PERICARDIAL SPACE THAT CAUSES HEMODYNAMIC COMPROMISE. THIS SHOULD BE DOCUMENTED BY EITHER: 1. ECHO SHOWING PERICARDIAL FLUID AND SIGNS OF TAMPONADE SUCH AS RIGHT HEART COMPROMISE. 2. SYSTEMIC HYPOTENSION DUE TO PERICARDIAL FLUID COMPROMISING CARDIAC FUNCTION. |
| AE294 | PERICARDITIS | AN INFLAMMATION OF THE PERICARDIUM (THE FIBROUS SAC SURROUNDING THE HEART). |
| AE295 | CARDIOVASCULAR - OTHER | |



Clinical Investigational Plan Protocol Number: 2010-03

| | | AECODELIST |
|---|---|---|
| CODE | LABEUNAME | DEFINITION |
| AE.8 | GASTROINTESTINAL/HEPATIC | |
| AE350 | GASTROINTESTINAL - ESOPHAGEAL RUPTURE/TEAR | ANY EVIDENCE OF PUNCTURE/DISSECTION/PERFORATION, VARICES OR OTHER DAMAGE TO THE ESOPHAGUS REQUIRING INTERVENTION. |
| AE351 | GASTROINTESTINAL - INFECTION | SEVERE INFLAMMATION OF THE GASTROINTESTINAL TRACT INVOLVING BOTH THE STOMACH AND SMALL INTESTINE RESULTING IN ACUTE DIARRHEA AND VOMITING. SHOULD BE CONFIRMED BY CULTURE |
| AE352 | GASTROINTESTINAL - OTHER | OTHER GASTROINTESTINAL EVENT THAT DOES NOT FIT IN ONE OF THE OTHER GI/HEPATIC CATEGORIES. |
| AE353 | LIVER FAILURE - ACUTE | A SYNDROME DEFINED BY THE OCCURRENCE OF ENCEPHALOPATHY, COAGULOPATHY AND JAUNDICE IN AN INDIVIDUAL WITH A PREVIOUSLY NORMAL LIVER. |
| AE354 | LIVER FAILURE - CHRONIC | CHRONIC LIVER DISEASE CAUSES CAN BE ANY CONDITION THAT RESULTS IN THE GRADUAL DEGRADATION AND RENEWAL OF THE TISSUE CELLS WITH A BODY'S LIVER. THIS PROCESS USUALLY RESULTS IN FIBROSIS OR CIRRHOSIS. DIAGNOSIS MAY BE CONFIRMED BY ABNORMAL BLOOD ENZYMES AND/OR BIOPSY |
| AE355 | HEPATIC COMPLICATION - OTHER | OTHER LIVER EVENTS THAT DO NOT MEET THE DEFINITION OF LIVER FAILURE (E.G. LIVER DYSFUNCTION) REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE356 | PANCREATIC COMPLICATION (PANCREAS) | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE PANCREAS REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE357 | SPLENIC COMPLICATION (SPLEEN) | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE SPLEEN REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE358 | BILIARY (GALLBLADDER) | AN EVENT PERTAINING TO BILE OR TO THE GALLBLADDER AND BILE DUCTS, WHICH TRANSPORT BILE REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE359 | ENDOCRINE COMPLICATIONS | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE ENDOCRINE SYSTEM REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE360 | METABOLIC COMPLICATIONS | AN EVENT PERTAINING TO, CONNECTED WITH, OR AFFECTING THE METABOLIC SYSTEM REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.9 | GENITOURINARY/RENAL | |
| AE370 | URINARY TRACT INFECTION (UTI) | INFECTION THAT AFFECTS ANY PART OF THE URINARY TRACT THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE371 | VAGINAL INFECTION | INFECTIONS AFFECTING THE VAGINAL AREA THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE372 | GENITOURINARY - OTHER | OTHER GENITOURINARY EVENT NOT PREVIOUSLY DESCRIBED REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE373 | RENAL DYSFUNCTION | AN ACUTE EVENT OR WORSENING OF RENAL FUNCTION POST-OPERATIVELY (INCREASE OF SERUM CREATININE TO < 2.0, AND < 2x MOST RECENT PREOPERATIVE CREATININE LEVEL) AND DOES NOT REQUIRE DIALYSIS. |

CONFIDENTIAL AND PROPRIETATARY DATA: THIS DOCUMENT AND THE INFORMATION CONTAINED HEREIN MAY NOT BE REPRODUCED, USED, OR DISCLOSED WITHOUT WRITTEN PERMISSION FROM EDWARDS LIFESCIENCES LLC  



AE CODE LIST

Edwards

DEFINITION CODE LABEL/NAME



Clinical Investigational Plan Protocol Number: 2010-03

| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.9 | GENITOURINARY/RENAL (CONTINUED) | |
| AE374 | RENAL FAILURE — ACUTE | AN ACUTE EVENT OR WORSENING OF RENAL FUNCTION RESULTING IN ONE OR MORE OF THE FOLLOWING: 1) INCREASE OF SERUM CREATININE TO >2.0, AND 2X MOST RECENT PREOPERATIVE CREATININE LEVEL. 2) A NEW REQUIREMENT FOR DIALYSIS POSTOPERATIVELY. |
| AE375 | RENAL FAILURE — CHRONIC | A PROGRESSIVE LOSS IN RENAL FUNCTION OVER A PERIOD OF MONTHS OR YEARS RESULTING IN A DIAGNOSIS OF STAGE 5 - CHRONIC KIDNEY DISEASE. |
| AE376 | RENAL - OTHER | OTHER EVENT THAT IS NOT RENAL FAILURE OR RENAL DYSFUNCTION THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.10 | PULMONARY/RESPIRATORY | |
| AE380 | ATELECTASIS | COMPLETE OR PARTIAL COLLAPSE OF A PREVIOUSLY INFLATED LUNG; INABILITY OF LUNG TO FULLY EXPAND. |
| AE381 | HYPOXEMIA | DECREASED PARTIAL PRESSURE OF OXYGEN IN BLOOD SOMETIMES SPECIFICALLY AS LESS THAN 60 MMHG (8.0 KPA) OR CAUSING HEMOGLOBIN OXYGEN SATURATION OF LESS THAN 90%. |
| AE382 | PLEURAL EFFUSION - RIGHT | EXCESS ACCUMULATION OF FLUIDS, SOMETIMES BLOOD IN THE PLEURAL SPACE, WHICH IS COMMON AFTER CARDIAC SURGERY. REPORTABLE WHEN IT BECOMES SYMPTOMATIC AND REQUIRES FLUID TO BE INTERVENTIONALLY REMOVED. |
| AE383 | PLEURAL EFFUSION - LEFT | |
| AE384 | PLEURAL EFFUSION - BILATERAL | |
| AE385 | PNEUMOTHORAX | ACCUMULATION OF AIR OR GAS IN THE PLEURAL CAVITY, OCCURRING BECAUSE OF DISEASE OR INJURY AND REQUIRING SURGICAL INTERVENTION, HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE386 | PULMONARY EDEMA | AN ABNORMAL ACCUMULATION OF FLUID IN THE LUNGS REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE387 | PULMONARY HYPERTENSION | MEAN PULMONARY ARTERY PRESSURE THAT IS GREATER THAN 25 MMHG AT REST AND/OR GREATER THAN 30 MMHG DURING EXERCISE CONFIRMED BY SWAN GANZ CATHETER OR DIAGNOSTIC PLACEMENT IN THE PULMONARY ARTERY BED AND CONDITION REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE388 | PULMONARY REGURGITATION | THE BACKWARD FLOW OF BLOOD FROM THE PULMONARY ARTERY, THROUGH THE PULMONARY VALVE, AND INTO THE RIGHT VENTRICLE OF THE HEART DURING DIASTOLE. |
| AE389 | PULMONARY EMBOLISM - RIGHT | CLINICAL EVIDENCE OF NEW EMBOLISM WITH CONFIRMATION BY LUNG SCAN OR PULMONARY ANGIOGRAPHY. |
| AE390 | PULMONARY EMBOLISM - LEFT | |
| AE391 | PULMONARY EMBOLISM - BILATERAL | |
| AE392 | PULMONARY/RESPIRATORY - OTHER | OTHER RESPIRATORY EVENT THAT IS NOT RESPIRATORY FAILURE. |
| AE393 | RESPIRATORY DYSFUNCTION/INSUFFICIENCY | DETERIORATION OF SUBJECT'S RESPIRATORY EFFORTS LESS THAN 24 HRS AFTER COMPLETION OF THE INDEX PROCEDURE. |



AE CODE LIST

DEFINITION

Edwards

CODE LABEL/NAME



Clinical Investigational Plan Protocol Number: 2010-03

| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE.10 | PULMONARY/RESPIRATORY | |
| AE394 | RESPIRATORY FAILURE -ASTHMA | NEED FOR MECHANICAL VENTILATION REQUIRED GREATER THAN 24 HRS AFTER OF COMPLETION OF THE INDEX PROCEDURE (TIME 0 = WHEN THE SUBJECT LEAVES THE OR), OR NEED FOR RE-INTUBATION AND VENTILATOR SUPPORT OCCURRING ANY TIME WITHIN 30 DAY OF THE INDEX PROCEDURE WILL BE CONSIDERED RELATED TO THE INDEX PROCEDURE. |
| AE395 | RESPIRATORY FAILURE -EMPHYSEMA | |
| AE396 | RESPIRATORY FAILURE -COPD | - |
| AE397 | RESPIRATORY FAILURE -PNEUMONIA | |
| AE398 | RESPIRATORY FAILURE -PNEUMOTHORAX | |
| AE399 | RESPIRATORY FAILURE -HEMOTHORAX | |
| AE400 | RESPIRATORY FAILURE - ARDS | " ACUTE RESPIRATORY DISTRESS SYNDROME |
| AE401 | RESPIRATORY FAILURE -OTHER | · |
| AE402 | RESPIRATORY INFECTION - UPPER (URI) | THE ILLNESSES CAUSED BY AN ACUTE INFECTION WHICH INVOLVES THE UPPER RESPIRATORY TRACT: NOSE, SINUSES, PHARYNX OR LARYNX. THIS COMMONLY INCLUDES: TONSILLITIS, PHARYNGITIS, LARYNGITIS, SINUSITIS, OTITIS MEDIA, AND THE COMMON COLD. |
| AE403 | RESPIRATORY INFECTION - PNEUMONIA | LUNG INFECTION DOCUMENTED BY BLOOD STUDIES OR CHEST X-RAY, REQUIRING TREATMENT WITH ANTIBIOTICS, INHALATION THERAPY, INTUBATION OR SUCTIONING. |
| AE.11 | PERIPHERAL VASCULAR | |
| AE420 | VASCULAR - ACCESS SITE COMPLICATION | COMPLICATIONS OF BLEEDING OR INFECTION AT THE SITE OF CARDIOPULMONARY ACCESS AND OR PERCUTANEOUS CORONARY INTERVENTION OR DIAGNOSTICS THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE421 | VASCULAR - DEEP VEIN THROMBOSIS (DVT) | FORMATION OF BLOOD CLOT (THROMBUS) IN THE LOWER EXTREMITIES (LEGS) CHARACTERIZED BY SWELLING, REDNESS, CLAUDICATION/PAIN IN AFFECTED LIMB. EVENT SHOULD BE CONFIRMED BY DOPPLER OR DUPLEX US STUDY, AND REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION TO RESOLVE. |
| AE423 | VASCULAR - OTHER | OTHER VASCULAR COMPLICATIONS GENERALLY RELATED TO A DISEASE PROCESS AND NOT TRAUMA THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.12 | PSYCHIATRIC | |
| AE431 | PSYCHIATRIC DISORDER | A PSYCHOLOGICAL OR BEHAVIORAL PATTERN GENERALLY ASSOCIATED WITH SUBJECTIVE DISTRESS OR DISABILITY THAT OCCURS IN AN INDIVIDUAL, AND WHICH IS NOT A PART OF NORMAL DEVELOPMENT OR CULTURE. SUCH A DISORDER MAY CONSIST OF A COMBINATION OF AFFECTIVE, BEHAVIORAL, COGNITIVE AND PERCEPTUAL COMPONENTS. |
| AE432 | suicide | A PERSON WHO INTENTIONALLY TAKES HIS OR HER OWN LIFE. |
| AE433 | TRANSIENT PSYCHOTIC SYNDROME | A MENTAL STATE OFTEN DESCRIBED AS INVOLVING A "LOSS OF CONTACT WITH REALITY" THAT LASTS ONLY FOR A |

CONFIDENTIAL AND PROPRIETATARY DATA: THIS DOCUMENT AND THE INFORMATION CONTAINED HEREIN MAY NOT BE REPRODUCED, USED, OR DISCLOSED WITHOUT WRITTEN PERMISSION FROM EDWARDS LIFESCIENCES LLC 



| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| | | SHORT TIME. |
| AE.12 | PSYCHIATRIC (CONTINUED) | |
| AE434 | PSYCHIATRIC – OTHER | OTHER NEUROLOGIC EVENT NOT PREVIOUSLY DESCRIBED THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.13 | MUSCULAR SKELETAL/ DERMATOLOGIC | |
| AE450 | STERNAL WOUND/THORACIC INFECTION | DEEP STERNAL INFECTION INVOLVING MUSCLE, BONE, AND/OR MEDIASTINUM. MUST INCLUDE ONE OF THE FOLLOWING: 1) WOUND OPENED WITH EXCISION OF TISSUE (I&D); 2) POSITIVE CULTURE; 3) TREATMENT WITH ANTIBIOTICS. (LAST SENTENCE REMOVED, WHICH IMPLIES THAT BACTERIAL PNEUMONIA AFFECTING PARTS OF THE LUNG ADJACENT TO THE STERNUM SHOULD BE COUNTED AS A STERNAL WOUND INFECTION.) |
| AE451 | BONE FRACTURE/BREAK | A BREAK IN BONE OR CARTILAGE. ALTHOUGH USUALLY THE RESULT OF TRAUMA, A FRACTURE CAN BE CAUSED BY AN ACQUIRED DISEASE OF BONE SUCH AS OSTEOPOROSIS OR BY ABNORMAL FORMATION OF BONE IN A DISEASE. |
| AE452 | WOUND INFECTION - OTHER | OTHER WOUND INFECTION THAT IS NOT RELATED TO THE SURGICAL ACCESS SITE. |
| AE454 | INFECTION /INFLAMMATION - OTHER | SOURCE OF INFECTION THAT IS CHARACTERIZED BY ELEVATED BLOOD LEVELS AND OR FEVER REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION (FEVER OF UNKNOWN ORIGIN FUO; CLINICALLY SIGNIFICANT ELEVATED WBC) |
| AE456 | MUSCULAR SKELETAL / DERMATOLOGIC - OTHER | OTHER SKIN/MUSCULAR/SKELETAL EVENT NOT PREVIOUSLY DESCRIBED THAT REQUIRES HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.14 | NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM | 8 |
| AE470 | ANAPHYLACTIC REACTION | AN ALLERGIC REACTION TO AN ANTIGEN THAT CAUSES CIRCULATORY COLLAPSE AND SUFFOCATION DUE TO BRONCHIAL AND TRACHEAL SWELLING. |
| AE471 | ALLERGIC REACTION - MEDICATION RELATED | A MILD TO MODERATE TO LIFE THREATENING REACTION TO A SUBSTANCE AND/OR MEDICATION. REPORT REACTIONS THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE472 | ALLERGIC REACTION - OTHER | A MILD TO MODERATE TO LIFE-THREATENING REACTION TO AN ENVIRONMENTAL OR ANIMAL SUBSTANCE. REPORT REACTIONS THAT REQUIRE HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE473 | CANCER - PROGRESSION OF UNDERLYING DISEASE | AN EXACERBATION OR WORSENING OF A CANCER DIAGNOSED/KNOWN PRIOR TO THE INDEX PROCEDURE. |
| AE474 | CANCER - NEWLY DIAGNOSED | A NEWLY DIAGNOSED CANCER FOLLOWING INDEX PROCEDURE. |
| AE475 | HEARING DISORDER | ANY DISORDER RELATED TO HEARING IMPAIRMENT REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE476 | MULTI-SYSTEM ORGAN FAILURE | OCCURS WHEN MORE THAN ONE ORGAN OF THE BODY STOPS FUNCTIONING NORMALLY AND HOMEOSTASIS CANNOT BE MAINTAINED WITHOUT INTERVENTION. |
| AE477 | SPEECH DISORDER | ANY DISORDER RELATED TO A SPEECH IMPEDIMENT REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE479 | VISION DISORDER | ANY DISORDER RELATED TO VISION IMPAIRMENT REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE480 | FEVER - UNKNOWN ORIGIN | (1) A TEMPERATURE GREATER THAN 38.3°C (101°F) ON SEVERAL OCCASIONS, (2) MORE THAN 3 WEEKS' DURATION OF ILLNESS, AND (3) FAILURE TO REACH A DIAGNOSIS DESPITE 1 WEEK OF INSUBJECT INVESTIGATION. |

 AND PROPRIETATARY DATA: THIS DOCUMENT AND THE INFORMATION CONTAINED HEREIN MAY NOT BE REPRODUCED, USED, OR DISCLOSED WITHOUT WRITTEN PERMISSION FROM EDWARDS LIFESCIENCES LLC REVISION C: 8 MAY 2012



Clinical Investigational Plan Protocol Number: 2010-03

| | | AECODELIST |
|---|---|---|
| CODE | LABEUNAME | DEFINITION |
| AE481 | NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION | ANY COMPLICATION THAT CANNOT OTHERWISE BE CATEGORIZED REQUIRING HOSPITALIZATION OR MEDICAL INTERVENTION. |
| AE.15 | DEVICE DYSFUNCTION | |
| AE500 | SVD - STUDY VALVE WEAR | INCLUDES DYSFUNCTION OR DETERIORATION INVOLVING THE OPERATED VALVE (EXCLUSIVE OF INFECTION OR THROMBOSIS). THE TERM STRUCTURAL VALVE DETERIORATION REFERS TO CHANGES INTRINSIC TO THE VALVE SUCH AS: WEAR, FRACTURE, CALCIFICATION, LEAFLET TEAR, MANUFACTURED SUTURE LINE DISRUPTION |
| AE501 | SVD - STUDY VALVE FRACTURE | ı |
| AE502 | SVD - STUDY VALVE POPPET ESCAPE | ıı e |
| AE503 | SVD - STUDY VALVE CALCIFICATION | - |
| AE504 | SVD - STUDY VALVE LEAFLET TEAR | II . |
| AE505 | SVD - STUDY VALVE STENT CREEP | n e e e e e e e e e e e e e e e e e e e |
| AE506 | SVD - STUDY VALVE SUTURE LINE DISRUPTION | n e e e e e e e e e e e e e e e e e e e |
| AE507 | SVD - STRUCTURAL VALVE DETERIORATION, OTHER | ıı e |
| AE525 | SVD - ANNULAR FRAME DAMAGE | ii a |
| AE526 | SVD - ANNULAR FRAME SEPARATION | II . |
| AE527 | SVD - STENT FRAME FRACTURE | ii e e e e e e e e e e e e e e e e e e |
| AE528 | SVD - STENT FRAME DEFORMATION | II . |
| AE529 | SVD - STENT FRAME SEPARATION | a contract of the contract of |
| AE512 | NSD - ENTRAPMENT BY PANNUS, TISSUE, OR SUTURE | ANY ABNORMALITY NOT INTRINSIC TO THE VALVE (DO NOT DIRECTLY INVOLVE VALVE COMPONENTS) ITSELF THAT RESULTS IN STENOSIS OR REGURGITATION OF THE OPERATED VALVE OR HEMOLYSIS (EXCLUDES THROMBOSIS AND INFECTION). EXAMPLES INCLUDE: ENTRAPMENT BY PANNUS, TISSUE, OR SUTURE, PARAVALVULAR LEAK, INAPPROPRIATE SIZING, INAPPROPRIATE POSITIONING, REGURGITATION AS A RESULT OF TECHNICAL ERROR, STJ DILATION OF THE VALVE ANNULUS, OBSTRUCTION OF THE CORONARY OSTIA BY THE STUDY VALVE. |
| AE164 | NSD - PARAVALVULAR LEAK - +1 | LEAKAGE BETWEEN THE SEWING RING AND THE ANNULUS. |
| AE165 | NSD - PARAVALVULAR LEAK - +2 | II . |
| AE166 | NSD - PARAVALVULAR LEAK - +3 | ı, |
| AE167 | NSD - PARAVALVULAR LEAK - +4 | n e e e e e e e e e e e e e e e e e e e |
| AE176 | NSD - STUDY VALVE STENOSIS - MILD | "OSN |



Clinical Investigational Plan Protocol Number: 2010-03

| | | AECODELIST |
|---|---|---|
| CODE | LABEL/NAME | DEFINITION |
| AE177 | NSD - STUDY VALVE STENOSIS - MODERATE | "GSN |
| AE178 | NSD - STUDY VALVE STENOSIS - SEVERE | "QSN |
| AE121 | NSD - PARAVALVULAR LEAK WITH HEMOLYSIS | "OSN |
| AE514 | NSD - INAPPROPRIATE SIZING | "QSN |
| AE515 | NSD - INAPPROPRIATE POSITIONING | "GSN |
| AE516 | NSD - RESIDUAL LEAK OR OBSTRUCTION | "QSN |
| AE517 | NSD - INTRAVASCULAR HEMOLYTIC ANEMIA | NSD " CLINICALLY IMPORTANT |
| AE518 | NSD - DEVELOPMENT OF REGURGITATION | NSD " AS A RESULT OF TECHNICAL ERRORS |
| AE519 | NSD - DILATATION OF THE SINOTUBULAR JUNCTION | "GSN |
| AE520 | NSD - DILATION OF THE VALVE ANNULUS | "QSN |
| AE521 | NSD - CORONARY OSTIAL OBSTRUCTION | "QSN |
| AE522 | NSD - STUDY VALVE INSTABILITY | "QSN |
| AE523 | NSD - STUDY VALVE MIGRATION | "GSN |
| AE524 | NSD - LVOT DAMAGE | "GSN |

Clinical Trial Number: 2010-03



# 15.2 SAMPLE INFORMED CONSENT FORM

## Patient Information

#### CLINICAL STUDY # 2010-03:

## "Clinical Study of the Edwards Pericardial Aortic Bioprosthesis, Model 11000"

You are invited to take part in a clinical research study. This information sheet tells you why the research is being done and what it would involve for you if you chose to take part. Please read the following information carefully and feel free to discuss this with your family or your Doctor. If you are unclear about anything or would like more information, please contact, <Name> on <Tel. number>. Take time to decide whether or not you wish to take part. Your participation in this research study is voluntary. If you decide to participate we will ask you to sign this consent document in order to state your agreement.

This study has been given a favorable opinion by the <Ethics Committee> and by the <Competent Authority>. It will be conducted according to the regulations governing clinical research.

#### INTRODUCTION

The heart is a muscle, that works like a pump, moving blood into the lungs and the entire body. In the heart there are 4 valves, whose role is to allow blood to flow in the correct direction. When a valve doesn't work properly, the heart muscle has to work harder to pump the normal amount of blood around the body. This may cause symptoms such as tiredness, difficulty in breathing, fainting or in some cases a condition called angina pectoris. The symptoms are different depending on the valve that is damaged and the amount of the damage. If the symptoms are serious the valve can be surgically removed and replaced with a new valve. There are different types of replacement valves that are used based on a patients condition and symptoms. One type is the biological valve, sometimes refered to as a tissue valve or bioprosthesis. Bioprostheses made with pericardial tissue have been used for many years.

## WHAT IS THE PURPOSE OF THIS STUDY?

The purpose of this observational trial is to gather further clinical data to confirm the safety and performance of the Edwards Pericardial Aortic Bioprosthesis, Model 11000 (also referred to as the Model 11000).

## WHY CAN YOU PARTICIPATE IN THIS RESEARCH STUDY?

You are being invited to participate in this clinical research study because it has been determined that your aortic heart valve needs replacement and your doctor believes that you may benefit from receiving a biological valve.

A variety of biological heart prostheses are available from different manufacturers. In this study we intend to test the Model 11000 aortic biological prosthesis. The Model 11000 prosthesis is a new CE marked product. This new aortic valve was developed to treat patients having aortic valve diseases called stenosis or insufficiency, like you.

1 of 9

Patient Informed Consent Form DRAFT: 8 MAY 2012

#### STUDY DESIGN

This study will be conducted in up to 6 participating hospitals.

You may be one of approximately 200 participants invited to participate.

Your participation will last for 5 years. All participants will have to return to the hospital where the surgery was done and be checked by the study doctor or his colleagues on a regular basis. Following discharge you will be asked to return to the hospital at 3 months, 1 year, and annually until 5 years after the valve was implanted in your heart.

# DESCRIPTION OF THE EDWARDS PERICARDIAL AORTIC BIOPROSTHESIS MODEL 11000

The Edwards Pericardial Aortic Bioprosthesis Model 11000A is a CE marked device. The Model 11000A is identical to the Model 11000.

The Model 11000 valve is a CE marked Carpentier-Edwards PERIMOUNT Magna Ease 3300TFX valve, with modifications in tissue processing and valve sterilization.

The Magna Ease valve consists of three tissue leaflets made of bovine (cow) pericardium (heart tissue). These leaflets have been treated with a new Edwards tissue process, built on the CE marked Edwards ThermaFix process to stabilize and preserve tissue. This process also allows the Model 11000 to be stored in non-liquid packaging and to not require rinsing prior to implant.

#### HOW WAS THE VALVE UNDER INVESTIGATION TESTED?

The valve was tested in conformity with European Regulations. The results of these tests have shown that the valve is suitable for implant in humans.

The technique used for implanting the valve is similar to the one your doctor uses with other biological heart valves. Each of the study doctors involved in this clinical study has been properly trained on how to implant the Model 11000.

#### WHAT WILL HAPPEN TO ME IF I TAKE PART?

If you agree to participate in this study, you receive the same treatment as any other patient having a similar operation, although you will also have some more tests (described below). The extra tests will enable us to to collect more information about the valve and the surgery.

The decision about participating in this study is entirely yours.

Before your surgery, your doctor will discuss the study and answer any questions you may have. If you consent to participate you will be asked to sign and date an informed consent form. A copy of this form will be given to you.

The study doctor will then ask you questions and will run tests and procedures to see if you can participate in the study. These tests and procedures include:

- A screening assessment to see if you are eligible to participate in the study
- Your medical history will be reviewed
- You will be given a physical examination (a clinical evaluation of your condition), and any findings will be written down in the study chart

- The severity of your health will be graded using a standard scale called NYHA based on your ability to do physical activities.
- Your quality of life will be measured by two short health questionnaires
- You will have an echocardiogram (a machine that creates sound waves that can see the
  inside of your heart. The pictures are taken with a small probe that is put on the outside of
  your chest)
- You will have an electrocardiogram (a machine that records the electrical activity of your heart. The recording is done by putting self adhesive discs on your chest)
- Your blood will be collected for laboratory testing. The blood test will require a needle being
  inserted into a vein in your arm (or other area where a vein can be accessed). Approximately
  three teaspoons (15ml) of blood will be drawn at this visit for routine tests. Any remaining
  blood sample will be discarded according to hospital regulations.
- If you are a woman of child-bearing age (and are not sterile) a small amount of blood or urine
  will be obtained to check for pregnancy.

If the results of the tests and examinations do not meet the study requirements and your doctor assesses that you are not qualified to participate in the study, you will be excluded from the study and the study doctor will discuss with you an alternative treatment for your disease. No further commitments related to this study will be requested of you.

If, as a result of the above mentioned tests and examinations, your doctor assesses that you are eligible to participate in the study, you will be scheduled for your surgery.

This surgical procedure is performed under general anaesthesia as is normal for heart valve replacement. The cardiac surgeon will open the chest to enable access to the heart and will place your heart on a "heart-lung" machine while they operate on the valve. During your surgery and before the Model 11000 is implanted a small tube called a transesophageal ultrasound will be entered through your mouth and advanced down to the area of the heart. The doctor will use this ultrasound to take pictures of your heart and ensure it functions well once implanted. These are parts of every surgery to replace a heart valve.

If during surgery your study doctor finds a reason not to implant the Model 11000, you will receive another equivalent aortic Bioprosthesis approved in the market. You will be excluded from the study and you will not have any further commitments related to this study.

If your study doctor assesses that there are no further contraindications, your will receive the Model 11000 valve and will be considered enrolled in the study.

After your surgery and before you go home, you will have some more tests and examinations as described below:

- A physical examination will be performed
- Your blood will be collected for laboratory testing in order to determine the best pharmacological treatment for you
- An echocardiogram (a sound wave taking pictures of your heart) will be obtained to see that the newly implanted Model 11000 valve sits well in its position and that it works well
- You will have an electrocardiogram (recording of the electrical activity of your heart)

Patient Informed Consent Form DRAFT: 8 MAY 2012

- You will be asked if you have experienced any unusual symptoms or side effects since the procedure – any finding will be recorded in order to control your health
- An appointment will be scheduled for you to return to the study center approximately 3 months after your procedure date.

During your 3 months and subsequent annual follow-up visits, you will be asked to provide information about your health status and you will undergo the following procedures:

- A physical examination
- An electrocardiogram (electrical recording of the heart)
- An echocardiogram (sound wave taking pictures of your heart)
- Your health condition will be graded based on your ability to perform physical activities (NYHA class)
- Your quality of life will be measured by two short health questionnaires (only at 1-year follow-up visit)
- Your blood will be collected for laboratory testing in order to determine the best pharmacological treatment for you
- You will be asked if you have experienced any unusual symptoms or side effects since your last assessment
- An appointment will be scheduled for you to return to the study center approximately at 1 year from your procedure date.

#### PARTICIPANT RESPONSIBILITIES

If you decide to participate in this research study, you will have to follow the instructions given by your study doctor and his colleagues and come back to the hospital for all the follow up visits until the fifth follow up year. Completing all study visits is important to make sure that the study results are complete and accurate. If you wish to stop participating in the study or if you find you have not followed instructions listed above, it is important that you notify the study doctor or study staff.

Your participation in this research study is entirely voluntary and it is your right to refuse to participate or withdraw at any time without penalty or loss of benefits to which you are otherwise entitled. You are free to withdraw from the study at any time without giving any reason, even if you have confirmed in writing that you want to take part. Your decision to withdraw will not have any adverse effect whatsoever on your further treatment in our hospital.

Giving false, incomplete, or misleading information about your medical history, including past and present use of medications, could have a very serious effect on your health. It is very important that you give a true and complete medical history.

## WHAT ARE THE POSSIBLE BENEFITS OF TAKING PART?

There are no guaranteed benefits from participation in this clinical investigation.

The potential benefit resulting from this clinical study beyond those afforded by a routine valve replacement may be a slightly shortened procedure time.

DRAFT: 8 MAY 2012

Information gained from the conduct of this study may be of benefit to other people with the same medical condition in the future. The long-term results of using the study valve are not known at the present time. Alternative treatments may include palliative medical therapy, aortic balloon valvuloplasty and surgical replacement of the aortic valve with another prosthesis.

## WHAT ARE THE POSSIBLE RISKS OF TAKING PART?

You must understand that the treatment of choice for your condition is a heart valve replacement and that alternative valves are available.

As with all prosthetic heart valves, there is a possibility that serious complications, sometimes leading to death, could develop that were not anticipated. In addition, complications due to individual patient reaction to an implanted device, or to physical or chemical changes in the components, particularly those of biological origin, may occur at varying intervals (hours or days) necessitating reoperation and replacement of the prosthetic device. These risks will be explained to you by your study doctor. Should any side effects occur, they will be fully assessed and you will be monitored closely.

You may experience events and/or outcomes that may include, but are not necessarily limited to, the following:

- Allergic reaction or immunological response
- Angina (chest pain)
- · Aortic wall and or annulus damage
- Cardiac arrhythmias / Conduction interference (change in the heartbeat rhythm)
- Chordae damage or trauma (damage to the mitral valve structure)
- Coronary ostia blockage (occlusion)
- Endocarditis (infection of the valve)
- Heart failure
- · Hemolysis (Breaking open of red blood cells with release of hemoglobin)
- Hemolytic anemia
- Hemorrhage (bleeding related to the use of anticoagulant therapy)
- Myocardial infarction
- Prosthesis leaflet entrapment (Impingement)
- Prosthesis nonstructural dysfunction
- · Prosthesis pannus (excessive tissues growth around the valve)
- Prosthesis Paravalvular leak (blood leaking around the valve when it is closed)
- · Prosthesis regurgitation (blood leaking through the valve when it is closed)
- Prosthesis stenosis / Effective Orifice Area reduction (narrowing of the valve)
- Prosthesis structural deterioration (physical or chemical deterioration of valve components)
- Prosthesis thrombosis (blood clot attachment to the valve)
- Stroke or transient ischemic attack (TIA)
- Tissue deterioration including infection, calcification, thickening, perforation, de-generation, suture abrasion, instrument trauma, and leaflet detachment from the valve
- Thromboembolism
- Thrombotic obstruction

It is possible that these complications could lead to:

- Reoperation
- Explantation
- · Permanent disability

#### WHAT HAPPENS IF I DECIDE AGAINST PARTICIPATING IN THE CLINICAL STUDY?

If you decide not to participate in the study you can discuss with your doctor which options of heart valve replacement best suit your requirements. This does not in any way affect your further medical care.

#### WHAT IF SOMETHING GOES WRONG?

Your doctor and the company that makes the valve (Edwards Lifesciences LLC (Irvine, CA)) will take all appropriate efforts to prevent you having any injury or illness which may occur as a result of your participation in this study. If you suffer any injury or illness as a direct result of participating in this study, you will receive medical care and treatment at this hospital. Signing this consent does not affect any legal rights you have.

As per the laws in your country, insurance has been taken out (Insurance company details).

Make sure you notify the insurance company without delay if you notice any deterioration in your state of health which may be related to the clinical study. Any such report may also be made by the study Investigator, your doctor.

## WILL MY TAKING PART IN THIS STUDY BE KEPT CONFIDENTIAL?

This section explains how your medical and health records might be used and disclosed if you agree to participate in this study.

All physicians involved in the study follow a strict clinical protocol. You have the right to determine who has access to your health records. Records collected in this study may include your medical history, the results of physical examinations, laboratory tests and other diagnostic or treatment procedures, as described above in this consent form, as well as basic demographic information.

By signing this form:

- You allow the study staff and/or the study doctor to use your medical records for the study and to disclose your health information to the sponsor, Edwards Lifesciences, LLC., or to the sponsor's representatives, in order to review the results of the study and to monitor the safety of participants.
- You allow the study doctor and/or sponsor to publish the results of the study or discuss the
  results at conferences. If this is done, no information will be included that would reveal your
  identity.

The information sent by the study doctor and/or study staff to the Sponsor will be anonymised, that means it will not include your name, address, or any other means of identification. Instead, the study doctor will use an assigned coded number to the records that are provided to the sponsor. However, your entire medical record may be reviewed at the study doctor's office and/or hospital by the Sponsor and/or Sponsor representatives, by regulatory/government agencies and the independent ethics committee (EC - is a group that has been formally designated to review and monitor research involving human subjects). The purpose of these reviews is to assure the quality of the study and patient safety.

The study doctor and/or study staff will make every effort to protect the privacy of your information. However, absolute confidentiality cannot be guaranteed because of the need to disclose information as described above.

You can cancel this authorization at any time by giving a written notice to the study doctor. If you cancel this authorization, then you will no longer be able to participate in the study, and the information that has been collected prior to canceling the authorization may still be used and disclosed to the above-mentioned parties. You will receive a signed copy of this consent for your records.

All data collected within the scope of the study may be forwarded to other persons or institutions not authorized for direct data inspection in an anonymized form only. We will inform your local doctor (general practitioner), only if you allow.

## PARTICIPATION AND WITHDRAWAL

You have the right to choose not to participate in this study or to stop participating at any time, without any consequences. This means that there will be no penalty or loss of medical benefits to which you are entitled.

If you choose to stop being a part of this study, you must first notify the study doctor immediately so that a plan can be provided for your continued medical care. At the time you stop taking part in the study, you will be asked to return for a final safety evaluation that will include gathering information about your current medical condition and conducting any required procedures. For your own safety, you should go through the study exit procedures any time you leave the study and make arrangements for your follow up care.

It is possible that your participation in this study may be stopped at any time. This might happen if you do not follow the instructions given by the study doctor or if the study doctor believes it to be in your best interest. The study may also be stopped for administrative, medical, or other reasons as determined by the study doctor or Edwards Lifesciences, LLC., or the regulatory authorities of the counties where this clinical study is conducted. Any significant new findings developed during the course of this research that might affect your willingness to participate will be provided to you by your doctor.

While participating in this study, you should not take part in any other study. This is to protect you from possible unforeseen injuries that may arise.

#### WHO IS ORGANISING AND FUNDING THE RESEARCH?

This study/research is organized by Edwards Lifesciences, LLC. the medical device company manufacturing the Model 11000 valve and the Sponsor of this study.

- The Sponsor reimburses the institution for tests and procedures needed for this study.
- 2. The study staff will not be paid to include you in this study but the hospital will be reimbursed for the costs incurred in conducting this research.

#### COSTS AND COMPENSATION

There will be neither charge, nor compensation, for your participation in this study. The investigational device, study-related procedures, and study visits will be provided at no charge.

DRAFT: 8 MAY 2012

You will be reimbursed for the travel expenses you face in order to come back to the hospital for the follow-up visits requested by this study

You will still be responsible for the cost of your usual ongoing medical care, including procedures and/or non-study drugs that are not required by this study. If you have any questions, please ask the study doctor, a member of the study staff.

## CONTACT DETAILS FOR FURTHER INFORMATION

| If you require any further information before or during the study, or if you have any questions at | fter |
|---|---|
| you have read this Patient Information, please contact the investigator responsible for you: | |

| | <br> | <br> | <br> |
|------------|------|------|------|
| Telephone: | <br> | | <br> |

## **FURTHER INFORMATION**

You consent to participate in a scientific study and in the statistical analysis of the results of that study. It is understood that your personal data continue to be subject to data protection and shall not be disclosed to any third parties. Participation in this study is voluntary, and you can discontinue participation at any time without giving reasons, and without penalty. The Principal Investigator or the sponsor may also decide on your premature discontinuation of this study.

DRAFT: 8 MAY 2012

# CONSENT FORM

| Title of the project: | Clinical study of an Edv | wards model 11000 a | ortic valve | | |
|---|---|---|---|---|---|
| Name of the Principal I | nvestigator: | | | | |
| Center number: | | | | | |
| Study number: | | | | | |
| Patient Indentification | Number: | | | Please init | ial box |
| | | | | | _ |
| (version | have read and understa<br>_) for the above study. I<br>k questions and have ha | have had the opport | unity to consid | | |
| | nat my participation is vo<br>ut giving any reason, wi | | | | |
| during the stud<br>from regulator | nat relevant sections of r<br>ly, may be looked at by<br>y authorities where it is<br>on for these individuals t | individuals from Edwarelevant to my taking | ards Lifescience<br>part in this re | es, | |
| 4. I agree to my G | P being informed of my | participation in the s | tudy. | Yes 🗌 | No 🗌 |
| | | | | | _ |
| 5. I agree to take | part in the above study. | | | | |
| Name of Patient | | Signature | D | ate | • |
| Name of legal represen | atative | Signature | D | ate | • |
| | this study with the abo<br>on, had an opportunity | | | | |
| Name of person taking | consent | Signature | | ate | - |

Patient Informed Consent Form DRAFT: 8 MAY 2012



# 15.3 CASE REPORT FORMS

| The same of the sa | | | |
|---|---|---|---|
| Edv | vards Life | esciences | Study Doc# |
| Subject | ID _ | | Site Visit Date Status |
| Visit Nar | me | | Subevent# CRF Name Blank CRF |
| | | | PREOPERATIVE INCLUSION / EXCLUSION CRITERIA Rev B |
| Plea | se indi | cate wh | ether or not the subject meets the following inclusion criterion |
| 1. | ON₀ | O Yes | Subject is 18 years or older |
| 2. | ON∘ | ○ Yes | Subject is diagnosed with aortic valve disease requiring a planned replacement as indicated in the preoperative evaluation |
| 3. | ON∘ | O Yes | Subject is scheduled to undergo planned aortic replacement with or without concomitant coronary bypass surgery |
| 4. | ON₀ | ○ Yes | Subject provided written informed consent prior to trial procedures |
| | | | Please indicate when the subject signed the informed consent form: Date: (DD/MMM/YYYY) Time: (HH:MM) |
| 5. | ON₀ | ○ Yes | Subject is geographically stable and agrees to attend follow-up assessments at the hospital of surgical services for up to 5 years |
| Plea | se indi | cate who | ether or not the subject meets any of the following exclusion criterion |
| 1. | ON₀ | O Yes | Subject requires emergency surgery |
| 2. | ON∘ | ○ Yes | Subject has prior mitral, tricuspid or pulmonic valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain in situ |
| 3. | O N∘ | ○ Yes | Subject requires multiple valve replacement/repair |
| 4. | ON₀ | ○ Yes | Subject requires a surgical procedure outside of the cardiac area (e.g. vascular bypass) |
| 5. | O No | O Yes | Subject has aneurysm of the aortic root and/or ascending aorta requiring surgical intervention |
| 6. | O No | ○ Yes | Subject has active endocarditis/myocarditis or endocarditis/myocarditis within 3 months to the scheduled aortic valve replacement (AVR) surgery |
| 7. | ON∘ | O Yes | Subject has renal insufficiency as determined by creatinine (S-Cr) level >= 2.5 mg/dL or end-stage renal disease requiring chronic dialysis at screening visit |
| 8. | O No | ○ Yes | Subject has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months (180 days) prior to AVR surgery |
| 9. | ON∘ | ○ Yes | Subject has acute myocardial infarction (MI) within 30 days prior to AVR surgery |
| 10. | ON∘ | ○ Yes | Subject has presence of non-cardiac disease limiting life expectancy to less than 12 months |
| 11. | ON₀ | ○ Yes | Subject is diagnosed with hypertrophic obstructive cardiomyopathy (HOCM) |

| Edwards Lifesciences | Study Doc# | | |
|---|---|---|---|
| Subject ID | Site Visit Date Status | | $\neg$ |
| Visit Name | Subevent# CRF Name | Blank CRF | |
| | | | _ |
| 12. ONo OYes | Subject is diagnosed with hyperparathyroidism | | |
| 13. ONo OYes | Subject exhibits left ventricular ejection fraction =< 30% as validated by procedure within 30 days prior to AVR surgery | by diagnostic | С |
| 14. ONo OYes | Subject has echocardiographic evidence of an intra-cardiac mass, three or vegetation | ombus, | |
| 15. No Yes | Subject has hemodynamic or respiratory instability requiring inotropic mechanical circulatory support, or mechanical ventilation within 60 da AVR surgery | | |
| 16. No Yes | Subject has documented leukopenia (WBC < 3.5x 10^3/uL), acute and (Hgb < 10.0 gm/dL or 6 mmol/L), thrombocytopenia (platelet count < 5 or history of bleeding diathesis or coagulopathy | | |
| 17. ONo OYes | Subject is diagnosed with myxomatous disease/connective tissue disease. (e.g. Marfan's Syndrome) | orders | |
| 18. O No O Yes | Subject has prior organ transplant | | |
| 19. ONo OYes | Current or recent participation (within 6 weeks prior to surgery) in an indrug or device trial | investigation | al |
| 20. O No O Yes | Subject was previously implanted with trial device | | |
| 21. ONo OYes | Subject is pregnant (female subject of childbearing potential only), lac<br>or planning to become pregnant during the duration of participation in | _ | |
| 22. O No O Yes | Subject is currently incarcerated or unable to give voluntary informed | consent | |
| 23. No Yes | Subject has documented history of substance (drug or alcohol) abuse last 5 years prior to implant | within the | |
| Based on the answers to the preoperative inclusion and exclusion criteria, is this subject eligible for intraoperative evaluation? O No O Yes | | | |
| Has a surgery of | date for this subject been scheduled? ONO OYes | | |
| Please indi | dicate the estimated surgery date: (DD/MMM/YYYY | <b>(</b> ) | |

| Edwards Lifesciences | Study | | Doc# | |
|---|---|---|---|---|
| Subject ID | Site Visit Date | | Status | |
| Visit Name | Subevent# CRF Name | | | Blank CRF |
| | TRA-OPERATIVE EXCLUSION ( | | | Rev B |
| boes the subject have the | Tollowing anatomic variances willo | ii contrain | alcate imple | int of the valve |
| Position of the corons that would result in obsi | ary ostia relative to the study valve truction of blood flow | O No | O Yes | |
| <ol><li>The device is not ava<br/>subject</li></ol> | ailable in the correct size for the | O No | O Yes | |
| | mically unstable during the<br>procedure to be aborted prior to<br>vice | O No | O Yes | |
| | that a trial valve cannot be implanted<br>duation and prior to a trial valve<br>other reason | O No | O Yes | |
| Please specify: | | | | |
| Was the subject enrolle | d in the study? | O No | O Yes | ) |

| E Edward | s Lifesciences | Study | | | | Doc# | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | | Site | $\overline{}$ | Visit Date | | Status | | | $\overline{\neg}$ |
| Visit Name | | Subevent# | | CRF Name | | J | Blank | CRF | |
| DEMOGRAPHICS Rev B | | | | | | | | | |
| Age: | | | | | | | | | |
| What fo | rmat will be used t | o indicate the sub | oject's | age? | | | | | |
| 0 | Birth date (DD/MM | M/YYYY) | | | | | | | |
| | Birth date: | | | | | | | | |
| 0 | Year (YYYY) and a | age | | | | | | | |
| | Year: | | | | | | | | |
| | Age: | | | | | | | | |
| Gender | | | | | | | | | |
| | Male<br>Female | | | | | | | | |
| O | | | | | | | | | |
| | Was a pregnancy | y test performed? | | | | | | | |
| | What was | the result? | | | | | | | |
| | ON- | | | | | | | | |
| O № | | | | | | | | | |
| | Why was | the pregnancy tes | st not | performed? | | | | | |
| | | N I | | | | | | | _ |
| | - | Please specify: | | | | | | | |
| | | | | | | | | | _ |
| Is the s | ubject willing to i | dentify their rac | e/ethr | nicity? | )No (Yes | | | | |
| Ple | ase indicate the su | ıbject's race: | | | | | | | |
| | | | | | | | | | _ |
| | Please spe | cify: | | | | | | | |
| | | | | | | | | | l |
| Ple | ase indicate the su | hiect's ethnicity: | | | | | | | - |
| 1 10 | and majorite the st | ,coto cumoty. | | | | | | | |
| | Please spe | cify: | | | | | | | ٦ |
| | • | | | | | | | | |
| | | | | | | | | | 1 |

| E Edwards Lifesciences Study | | | Doc# |
|---|---|---|---|
| Subject ID Site | \ | /isit Date | Status |
| Visit Name Subevent# | | CRF Name | Blank CRF |
| Subject height: | ) in | | |
| What is the subject's Canadian Cardiovascular Society (CCS) Angina Class? | | | |
| What is the subject's current Left Ventricular Ejection Fraction (LVEF)? | | | |
| What is the subject's baseline serum creatinine value (mg/dL)? | | | |
| Is this value within the normal range? | O No | ○ Yes | |
| Was this result clinically significant? | O No | ○ Yes | |

| E Edwards | Lifesciences | Stud | ty | | | Doc# | |
|---|---|---|---|---|---|---|---|
| Subject ID | | Site | | Visit Date | | Status | |
| Visit Name | | Sub | event# | CRF Name | | | Blank CRF |
| | | ME | DICAL HISTO | ORY (Part | 1) | | Rev B |
| | VASCULAR M | | | | | | |
| _ | | | | | the following diseas | ses / cond | litions? |
| O No | | | ery Disease (C | | | | |
| | _ | _ | | - | have >= 50% narr | | |
| | O No | O Yes | | _ | (LAD) coronary art | ery | |
| | O No | O Yes | Circumflex of | | er y | | |
| | O №<br>O № | O Yes<br>O Yes | Right corona<br>Left main cor | - | v | | |
| O No | OYes Ca | • | | oriary arter | y | | |
| 00 | | _ | severity of the | disease: [ | | | |
| O No | _ | | ery/Vascular [ | - | | | |
| One | | | | | | | |
| | _ | _ | | ne subject r | as experienced: | | |
| | O No | O Yes | Claudication | is of any ne | ripheral artery | | |
| | O No | ○ Yes | | | eripheral artery | | |
| _ | O No | O Yes | Aortic aneury | /sm | | | |
| O No | O Yes Pu | monary Hy | pertension | | | | |
| | What is the | ne severity | of the conditio | n? | | | |
| O No | ○Yes Sys | stemic Hyp | ertension | | | | |
| 0 140 | | dicate if the | | | | | |
| | O No | O Yes | - | ented histo | ry of hypertension | diagnose | d and treated |
| | Ono | 0 163 | with medicat | | | ulagilose | and treated |
| | ○ No | ○ Yes | Has prior documentation of blood pressure >140 mmHg systolic or 90 mmHg diastolic for patient without diabetes or chronic kidney disease; or prior documentation of blood pressure > 130 mmHg systolic or 80 mmHg diastolic on at least 2 occasions for patients with diabetes or chronic kidney disease | | | | |
| | O No | OYes | Is currently o | n pharmac | ologic therapy to co | ntrol hype | ertension |
| O No | ○Yes Ca | rdiomyopat | thy | | | | |
| _ | Please in | dicate the t | ype of cardion | nyopathy | | | |

| E Edwards l | Lifesciences | Stud | У | | | Doc# | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | | Site | | Visit Date | | Status | | |
| Visit Name | | Sube | event# | CRF Name | | | Blank CRF | |
| O No | O Ves | Congestive He | art Failure // | CHE/ | | | | |
| | • | | , | ZHF) | | | | |
| O No | O Yes | Aortic Stenosi | S | | | | | |
| O No | O Yes | Aortic Insuffici | ency | | | | | |
| | Pleas | e indicate the la | ast known se | verity: | | | | |
| O No | O Yes | Mitral Stenosis | 5 | | | | | |
| O No | O Yes | Mitral Insuffici | ency | | | | | |
| | Pleas | e indicate the la | ast known se | verity: | | | | |
| O No | O Yes | Tricuspid Ster | osis | | | | | |
| O No | O Yes | Tricuspid Insu | fficiency | | | | | |
| | Pleas | e indicate the la | ast known se | verity: | | | | |
| O No | O Yes | Myocardial Inf | arction (MI) | | | | | |
| | What | types of myoca | ardial infraction | n (MI) has the | e subject experienc | ed? | | |
| | 01 | No OYes | ST elevatio | n MI (STEMI) | ) | | | |
| | 01 | No OYes | Non ST-ele | vation MI (NS | STEMI) | | | |
| | 01 | No OYes | Other type | of MI | | | | |
| | | Pleas | e specify: | | | | | $\neg$ |
| | 01 | No OYes | Unknown ty | pe of MI | | | | |
| | Is the | date (DD/MMN | I/YYYY) wher | n the last kno | wn MI occurred kno | own? ( | )No ⊜Yes | 3 |
| | | ate of last know | | | ٦ | | | |
| | Is | the approximat | e number of r | months since | —<br>the occurrence of t | he last M | 1l known? | |
| | | ONo OY | es | | | | | |
| | | N | umber of mor | iths: | | | | |
| | | Di | d the event o | ccur >5 years | ago? ONo C | ) Yes | | |

| E Edwards Lifesciences | | Stud | Study | | | | | Doc# | | |
|---|---|---|---|---|---|---|---|---|--|--|
| Subject ID | | Site | | Visit Date | | | Status | | | |
| Visit Name | | Sub | event# | CRF Name | | | _ | Blank CRF | | |
| ○ No ○ Yes Cardiac rhythm abnormalities/conduction disturbances Has the subject ever had the following cardiac rhythms? | | | | | | | | | | |
| | O No | O Yes | Sinus tach | ycardia | | | | | | |
| | O No | O Yes | Sinus brad | lycardia | | | | | | |
| | O No | O No O Yes Atrial fibrillation / Supraventricular tachycardia | | | | | | | | |
| | Please indicate the episodic pattern: | | | | | | | | | |
| Is this a permanent condition? O No O Yes | | | | | | | | | | |
| | O No | O Yes | Atrial flutte | r | | | | | | |
| | O No | O Yes | Tachycardi | a-bradycardia | syndro | me | | | | |
| | O No | <b>○</b> Yes | Ventricular | tachycardia | | | | | | |
| Please indicate the episodic pattern for VT | | | | | | | | | | |
| | O No | O Yes | Other card | iac rhythm abr | ormalit | ty | | | | |
| | | Please | e specify: | | | | | | | |
| Has the subject ever shown sign of the following conduction disturbances? | | | | | | | | | | |
| | O No | <b>○</b> Yes | AV block | | | | | | | |
| | | Indica | te the last re | corded degree | e of AV | Block: | | 1 | | |
| | O No | O Yes | Bundle bra | nch block | | | | | | |
| | | Indica | ate branch: | | | | | | | |
| | O No | O Yes | Other cond | luction disturba | ance | | | | | |
| | | Pleas | e specify: | | | | | | | |
| Edwards Li | fesciences | Stud | у | | | Doc# | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | | Site | | Visit Date | | Status | | |
| Visit Name | | Sube | event# | CRF Name | | | Blank CRF | |
| 0 | • | | | | | | | |
| ○ No | | erebrovascu<br>cate if the si | | perienced the | following types of | cerebrova | scular even | ts: |
| | O No | OYes T | ransient ische | emic attack ( | TIA; recovered with | nin 24 hour | rs) | |
| | | Is the da | ate when the I | ast known T | A occurred known | ? ONo | <b>○</b> Yes | |
| | | Date | of last known | TIA: | | ] | | |
| | | | approximate | | onths since the oc | currence o | f the last | |
| | | | | Num | ber of months: | | | |
| | | | Die | d the event o | ccurr > 5 years ago | o? () No | ○ Yes | |
| | O No | _ | | | Stroke (CVA; did no | _ | _ | urs) |
| | | | | | VA occurred know | n? ∪No<br>1 | O Yes | |
| | | | of last known | | | ] | | |
| | | | approximate<br>(nown? O No | | eeks since the occ | urrence of | the last | |
| | | | | Num | ber of weeks: | | | |
| | | | Die | d the event o | ccur > 5 years ago | ? () No | ○ Yes | |
| | Does the si | | severe impair<br>O Yes | ment of mob | ility as a result of a | neurologio | cal | |

| E Edwards | Lifesciences | Study | | Doc# | | |
|---|---|---|---|---|---|---|
| Subject ID | | Site | Visit Date | | Status | |
| Visit Name | | Subevent# | CRF Name | | | Blank CRF |
| O No | • | Endocarditis<br>n was the subject last being | treated for en | docarditis? | | |
| O No | | Myocarditis<br>n was the subject last being | treated for my | ocarditis? | | |
| O No | O Yes | Hyperlipidemia or Hyperch | olesterolemia | | | |
| O N₀ | O Yes | Rheumatic fever | | | | |
| O No | O Yes | Pulmonary valve stenosis | | | | |
| O No | ○ Yes | Pulmonary valve insufficier | ncy | | | |
| | Pleas | se indicate the last known se | everity: | | | |
| Does the | subject h | nave a history of: | | | | |
| O N₀ | O Yes | Smoking | | | | |
| | Is the | e subject a current smoker? When did the subject quit? | | ) Yes | | |
| O No | ○ Yes | Alcohol/Drug Abuse | | | | |

| Edwards Lifesciences Study GLX_EXT_2010_03 Doc# |
|---|
| Subject ID Site Visit Date Status |
| Visit Name BASELINE Subevent# CRF Name MEDICAL_HISTORY_P2 Blank CRF |
| MEDICAL HISTORY (Part 2) Version A |
| PRIOR CARDIOVASCULAR SURGICAL INTERVENTIONS |
| How many previous cardiovascular surgeries has the subject had? |
| How many cardiac/heart surgeries has the subject previously had? |
| Has the subject required amputation of a limb due to arterial disease? ONO OYes |
| Has the subject been implanted with a permanent pacemaker or an implantable cardioverter defibrillator (ICD)? O No O Yes |
| Please specify the type of implant the subject has: |
| Is the date of the implant known? ONo OYes |
| Date of implant: |
| Is the approximate number of months since the implant known? O No O Yes |
| Approximately how many months ago was the subject implanted? |
| Did the event occur > 5 years ago? O No O Yes |
| Were surgical interventions performed on any of the following cardiovascular components? |
| O No O Yes Carotid Arteries |
| What type of intervention was done on the carotids? |
| Please specify: |
| O No O Yes Abdominal Aorta |
| O No O Yes Thoracic Aorta |
| ONo OYes Limb Arteries |

\_

| areas . | | _ | |
|---|---|---|---|
| Edwards Life | esciences | Study | GLX_EXT_2010_03 Doc# |
| Subject ID | | Site | Visit Date Status |
| Visit Name BAS | ELINE | Subever | ent# CRF Name MEDICAL_HISTORY_P2 Blank CRF |
| - | | | |
| O No | O Yes Cor | onary Arte | teries |
| | What type | of interver | entions have been performed? |
| | O No | ○ Yes | CABG |
| | | How | w many grafts were done? |
| | O No | ○ Yes | Percutaneous transluminal coronary angioplasty (PTCA) /<br>Percutaneous coronary intervention (PCI) |
| | | Was | s a stent employed for any of the past PTCA / PCI procedures? |
| | | ( | ○ No ○ Yes ○ Unknown |
| | O No | ○ Yes | Other intervention on the coronary arteries |
| | | Pleas | ase specify: |
| O No | OYes Aorti | ic Valve | |
| | Were the f | following ir | interventions performed? |
| | O No | O Yes | Valvuloplasty |
| | O No | <b>○</b> Yes | Valve Replacement |
| | O No | <b>○</b> Yes | Other repair |
| | | Pleas | ase specify: |

\_

| Edwards Lif | esciences | Study | GLX_EXT_2 | 010_03 | | Doc# | | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | | Site | | Visit Date | | Status | | |
| Visit Name BAS | SELINE | Subeve | nt# | CRF Name | MEDICAL_HISTOR | Y_P2 | Blank CRF | Ī |
| ON∘ | Yes Mitro Were the f | O Yes O Yes O Yes O Yes O Yes O Yes | Annulopla Valvulopla Valve rep Other rep | asty<br>lacement | , | | | 7 |
| | | | | <u></u> | | | | ┙ |
| O No | ○Yes Pulr | nonary val | ve | | | | | |
| | Were the | following in | nterventions | performed? | • | | | |
| | O No | <b>○</b> Yes | Valvulopl | asty | | | | |
| | O No | O Yes | Valve rep | lacement | | | | |
| | O No | ○ Yes | Other rep | air | | | | |
| | | Plea | se specify: | | | | | |
| O No | OYes Tric | uspid valve | е | | | | | |
| | Were the f | ollowing ir | nterventions | performed? | • | | | |
| | O N₀ | O Yes | Annulopla | asty | | | | |
| | ON₀ | ○ Yes | Valvulopl | asty | | | | |
| | O No | O Yes | Valve rep | | | | | |
| | O No | O Yes | Other rep | air | | | | |
| | | Pleas | se specify: | | | | | |
| O No | ○ Yes Oth | er Cardiov | ascular Cor | mponent | | | | |
| | Please specify | the location | on of the int | ervention ar | nd the type of surgi | cal proce | dure performe | ed |
| | 1 | | | | | | | |

| BTTOTAL | | | | | | _ | |
|---|---|---|---|---|---|---|---|
| Edwards Life | sciences | Study GL | X_EXT_2 | 010_03 | | Doc# | |
| Subject ID | | Site | | Visit Date | | Status | |
| Visit Name BAS | ELINE | Subevent | # | CRF Name | MEDICAL_HISTOR | Y_P2 | Blank CRF |
| - | | | | | | | |
| | IOVASCULAR RI | | | | | _ | |
| _ | _ | | | ject ever had | d the following dise | ases? | |
| O No | ○ Yes Blood | Diatheses | | | | | |
| | Please spec | cify the typ | e: | | | | |
| | Plea | se specify | <i>'</i> : | | | | |
| O No | O Yes Calcium | m Metabo | lic Disord | lers | | | |
| O No | O Yes Cance | r | | | | | |
| | Please spec | eify: | | | | | |
| | Has the sub | ject receiv | ed or will | the subject | receive chemother | apy within | |
| | 30 days prio | or to the st | udy proce | edure? | No OYes | | |
| O No | O Yes Chroni | c obstruct | ive pulmo | onary diseas | se (COPD) / Chroni | ic lung dise | ase |
| | Please indic | ate the FE | V1/FVC | value | | | |
| | What type of | f treatmen | t did the | subject rece | eive for this condition | n? | |
| | O No | ○ Yes | Chronic | inhaled or | oral bronchodilator | therapy | |
| | O No | O Yes | Chronic | steroid ther | rapy | | |
| | O No | O Yes | | or ventilation | | | |
| | O No | O Yes | | reatment | | | |
| | 0 | | specify: | | | | |
| | | | _p_0j. | | | | |

\_

| E Edwards Life | sciences Study GLX_EXT_2010_03 Doc# |
|---|---|
| Subject ID | Site Visit Date Status |
| Visit Name BASI | ELINE Subevent# CRF Name MEDICAL_HISTORY_P2 Blank CRF |
| - | |
| O No | ○ Yes Diabetes |
| | Please indicate the type of diabetes: |
| | Is the subject currently receiving the following treatments? |
| | O No O Yes Diet |
| | ○ No ○ Yes Oral |
| | O No O Yes Insulin |
| O No | O Yes Obesity (BMI >=30) |
| O No | O Yes Liver Disease |
| O No | O Yes Musculoskeletal Dysfunction |
| Do | pes the subject have severe impairment of mobility due to this condition? ONo OYes |
| ONe | O Voc. Bond Failure/Incufficionary |
| O No | O Yes Renal Failure/Insufficiency |
| | Is the date when the subject was diagnosed known? O No O Yes |
| | Date diagnosed |
| | Is the approximate number of months since the subject was diagnosed known? |
| | O No O Yes |
| | Approximately how many months ago was the subject diagnosed? |
| | Was the subject diagnosed > 5 years ago? ONO Yes |
| | Is the subject currently on dialysis? O No O Yes |
| O No | O Yes Other disease which requires immunosuppressive therapy inhaled or systemic steroid therapy or chemotherapy within 30 days of the study procedure |

-

| Edwards Lifesciences | Study | | Doc# | |
|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | |
| Visit Name | Subevent# | CRF Name | | Blank CRF |
| ASSESSMENT Rev B | | | | |
| What was the primary method of contact with the subject? | | | | |
| PLEASE PROVIDE THI | E FOLLOWING PHYSI | CAL ASSESSMENT I | PARAMETERS: | |
| Weight: Heart Rate: | Okg C | ) lb | | |
| Blood pressure: | BPM / Diastolic | mmHg | | |
| NYHA Classification | , | | | |
| NTIA Classification | | | | |
| Was an auscultation p | erformed? | | | |
| ○ No | | | | |
| ○ Yes | | | | |
| Date of auscul | tation exam: | (DD/MMM/YY | YY) | |
| Was an aortic | murmur heard? | | | |
| | f No, a transthoracic ec<br>Applicable for 2 and 4 y | | s not needed for this visi | t |
| ○ Yes I | Yes, please complete | transthoracic echocar | diogram (TTE) | |
| Was information abou | t the subject's curren | t medications collect | ed? | |
| _ | ase fill out a Medicatior | form (MED) | | |
| Was a transthoracic e | chocardiogram (TTE) | performed? | | |
| O No | | | | |
| Yes If Yes, plea | ase fill out a Echocardi | ogram form (ECHO (S | " | |
| Was an electrocardiog | ram (ECG) performed | l? | | |
| O No | ase fill out a Electrocard | diagram form (ECC) | | |
| O Tes II Yes, pied | ase IIII out a Electrocar | ulogram lorm (ECG) | | |
| Was a blood test perfo | rmed? | | | |
| ○ No<br>○ Yes If Yes, plea | ase fill out a Blood Data | a form (LABS) | | |
| Was Quality of Life ass | sessed? (Required at | Baseline and 1 Year o | nly) | |
| O No | | | | |
| O Yes If Yes, plea | ase fill out a Quality of | Life (QOL) form | | |

| E Edward | s Lifescien | ices | Study | | | | Doc# | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | | | Site | | Visit Date | | Status | | $\exists$ |
| Visit Name | | | Subev | /ent# | CRF Name | | • | Blank CRF | |
| 0 0 | No<br>Not applic | cable at B | aseline | | | sly reported? | for each | event. | |
| | Are the | event(s | that occi | urred within | the followin | ng AE classification | ons? | | |
| | O No | O Yes | Blood and | d Lymphatic | (Including Al | L Bleeding compli | cations) | | |
| | O No | ○ Yes | Cardiovas | scular - Arrh | ythmia | | | | |
| | O No | ○ Yes | Cardiovas | scular - Reg | urgitation | | | | |
| | O No | ○ Yes | Cardiovas | scular - Sten | nosis | | | | |
| | O No | ○ Yes | Cardiovas | scular - Emb | oolic Event/Va | alve Thrombosis | | | |
| | O No | ○ Yes | Cardiovas | scular - Misc | ; | | | | |
| | O No | ○ Yes | Device D | ysfunction | | | | | |
| | O No | ○ Yes | Gastrointe | estinal/Hepa | atic | | | | |
| | O No | ○ Yes | Genitouri | nary/Renal | | | | | |
| | O <sub>No</sub> | ○ Yes | Pulmonar | y/Respirator | ry | | | | |
| | O No | ○ Yes | Periphera | al Vascular | | | | | |
| | O No | O Yes | Psychiatri | ic | | | | | |
| | O No | ○ Yes | Muscular | Skeletal/De | rmatologic | | | | |
| | O No | ○ Yes | Nonspeci | fic or Unkno | wn Body Sys | tem | | | |
| Comme | nts | | | | | | | | 7 |

| E Edwards Li | fesciences | Study | | | | Doc# | |
|---|---|---|---|---|---|---|---|
| Subject ID | | Site | | Visit Date | | Status | |
| Visit Name | | Subeve | ent# | CRF Name | | | Blank CRF |
| SURGERY DATA Rev B | | | | | | | |
| Date of hos | spital adn | nission: | | (DD/MM | M/YYYY) | | |
| Date of sur | rgery: | | | (DD/MM | M/YYYY) | | |
| Implanting | surgeon | : | | | | | l |
| PREOPER | ATIVE CO | NDITION | | | | | |
| For Purpos<br>within 21 d | | k Score Asses:<br>○ No ○ Yes | sment, did a | a Myocardia | al Infarction (MI) o | occur | |
| Please | indicate t | the time interval | when the las | st MI occurre | ed: | | |
| Within 2 w | eeks prio | r to the surgica | l procedure | : | | | |
| Was th | e subject | in congestive he | eart failure? | O № ( | ) Yes | | |
| Did the | subject e | xperience an ar | rhythmia? | ONo C | ) Yes | | |
| W | as the obs | served arrhythm | ia considere | d Atrial fibril | lation or Atrial flutte | er? O No | Yes |
| | | | | | | | _ |
| | | | • | | ifter hospital adm | ission? ( | ONo OYes |
| What is | s the likely | cause of these | symptoms? | | | | |
| L | | | | | | | |
| | | | | | rs preceding surg<br>contraindicated? | | lo OYes |
| On the day | of surge | ry but prior to g | going under | anesthesia | a, did the subject | experience | or require: |
| O No | <b>○</b> Yes | Ventricular fibr | illation | | | | |
| O No | <b>○</b> Yes | Ventricular tac | hycardia | | | | |
| O No | O Yes | Cardiogenic sh | nock | | | | |
| O No | <b>○</b> Yes | Aborted sudde | n death | | | | |
| O No | <b>○</b> Yes | Acute renal fai | lure (anuria | or oliguria < | (10 ml/hr) | | |
| O No | <b>○</b> Yes | Cardiopulmona | ary resuscita | tion <1hr pri | ior to surgery | | |
| O No | <b>○</b> Yes | Ventilation bef | ore arrival in | anesthetic | room | | |
| O No | <b>○</b> Yes | Inotropic supp | ort or IABP | | | | |
| O No | ○ Yes | Another cardia | c interventio | n <= 6 hour | s prior to schedule | d surgery | |

| TT. | | | | | |
|---|---|---|---|---|---|
| Edwards Lifesciences | Study | | | Doc# | |
| Subject ID | Site | Visit Date | | Status | $\neg$ |
| Visit Name | Subevent# | CRF Name | | Blank CR | F 🗌 |
| What is the urgency of th | e surgery being per | formed? | | | |
| OELECTIVE (Admiss to the op | | oject's cardiad | function is stable | in the days/weeks pri | or |
| OURGENT (Not adm<br>they can | itted for the operation<br>be discharged) | n, but requires | surgery on the cu | rrent admission befor | e |
| OSALVAGE (Require | s cardiopulmonary re | suscitation p | rior to induction of | anesthesia) | |
| OEMERGENCY (Ope<br>to ope | | ginning of the | next working day a | after the decision mad | de |
| INTRA-OPERATIVE ETIO | OGY AND DIAGNO | SIS | | | |
| Were any of the following disease? | intraoperative diag | noses made | concerning the e | tiology of the valve | |
| ONo OYes Dege | enerative | | | | |
| ONo OYes Dystr | ophic calcification | | | | |
| ONo OYes Rheu | ımatic | | | | |
| ONo OYes Rem | ote endocarditis | | | | |
| ONo OYes Othe | r etiology | | | | |
| Please spe | ecify: | | | | $\neg$ |
| • | | | | | |
| Please confirm the diagno | osis for the current | renlacement | <b>.</b> - | | |
| ○ Stenosis | osis for the current | replacemen | • | | |
| O Stenosis with insuffi | ciency | | | | |
| O Pure insufficiency | olerioy | | | | |
| O Prosthetic valve dys | function | | | | |
| Other diagnosis | id redori | | | | |
| Please specify: | | | | | $\neg$ |
| , lease speeling. | | | | | |
| What surgical approach v | vas used? | | | | |
| Full sternotomy | | | | | |
| Mini upper sternotor | ny | | | | |
| O Right thoracotomy | | | | | |
| Other MIS approach | ı | | | | |
| Please specify: | | | | | $\neg$ |
| • • | | | | | |

| TOTAL I | | _ | | | | | _ | | |
|---|---|---|---|---|---|---|---|---|---|
| Edwards I | Lifesciences | Study | | | | ' | Doc# | | |
| Subject ID | | Site | | Visit Date | | , | Status | | |
| Visit Name | | Subevent# | | CRF Name | | | | Blank CRF | |
| Is there e<br>arteries? | evidence of the | following con | ditions o | f the aortic | valve, annu | ılus, ao | rtic wa | all, or coronar | y |
| ON | o O Yes Calc | ification | | | | | | | |
| | Was calci | fication observe | ed in the | following loc | ations? | | | | |
| | O No | Yes Anr | nulus | | | | | | |
| | O No | Yes Lea | ıflets | | | | | | |
| | O No | Yes Aor | tic wall | | | | | | |
| | O No | Yes Cor | onary art | eries | | | | | |
| ON | o OYes Leaf | let fusion | | | | | | | |
| ON | o OYes Leaf | let perforation | | | | | | | |
| ON | O Yes Myx | omatous | | | | | | | |
| ON | O Yes Vege | etation | | | | | | | |
| ON | o OYes Othe | er disease cond | lition | | | | | | |
| | Please sp | ecify: | | | | | | | |
| | AL APPROACH | | | | | | | | |
| | following conc | - | _ | | | | | | |
| ON | o O Yes Cor | | _ | TIING (CABG) | ) | | | | |
| | now many | y grafts were d | one? _ | | | | | | |
| ON | o O Yes Perm | nanent pacema | aker impla | ant | | | | | |
| | Was Card | iac Resynchro | nization 1 | Technique (C | RT) used? | O No | 0 | Yes | |
| ON | o O Yes Aut | omatic Implant | ed Cardio | overter Defib | rillator (AICE | D) impla | nt | | |
| | Was Card | iac Resynchror | nization T | echnique (C | RT) used? | O No | 0 | Yes | |

| Edwards Lit | fesciences § | Study | | | | Doc# | |
|---|---|---|---|---|---|---|---|
| Subject ID | | Site | Visit D | ate | | Status | |
| Visit Name | | Subevent# | CRF | lame | | | Blank CRF |
| O No | ○ Yes Atrial ablati<br>What type of ab<br>○ Primarily<br>○ Primarily | lation proce | | ne? | | | |
| O No | O Yes Aortic aneu | ırysm/dissed | tion repair | | | | |
| O No | Yes Occlusion / Please indicate | | | dage | | | |
| O No | O Yes Atrial septa<br>What was the t | | | | | | |
| O No | O Yes Septal mye | ctomy | | | | | |
| O No | Yes Other proce<br>Please specify: | edure | | | | | |
| Why w<br>Was th | unplanned procedure ne<br>ras this procedure ne<br>e unplanned procedure | ecessary?<br>ure a Ventrio | cular Assist [ | Device (\ | /AD) insertion? | O No | ) Yes |
| ○ No<br>○ Yes<br>W | | nserted? | | | | | |

| E Edwards I | Lifesciences | Study | | | | Doc# | |
|---|---|---|---|---|---|---|---|
| Subject ID | | Site | | Visit Date | | Status | |
| Visit Name | | Subeve | nt# | CRF Name | | | Blank CRF |
| O M | o valve implar ** <i>If Model 11</i> On what a | (If selected, power (If selected attempt was the (If '1' is selected) | d, please d<br>ject death<br>d, please d<br>e study val | omplete *** Complete the complete the ve implanted fill out one (1 | ) Device Performa | *** section<br>rudy Exit fo<br>ons: **<br>nce form) | orm) |
| | | | | | Device Performa | ic <del>e</del> iornis, | 1 |
| | Pleas | | e following<br>logram star<br>chocardiog<br>everity of o | questions: rted: ram was done central regurg | (HH:MM) e? iitation for the stud | y valve?<br>alve? | ) Yes |
| | After which | ch study valve a<br>(If '1' is select<br>Why was a se | attempt wa<br>ed, please | s a commerc | ete the following<br>ial valve implanted<br>() Device Performa<br>the study valve no | nce form | (PERF). |
| | Please pr<br>Manu | | wing inform | | ) Device Performa<br>he commercial val | | (PERF). |

| E Edward | s Lifescien | ices | Study | | | | Doc# | |
|---|---|---|---|---|---|---|---|---|
| Subject ID | | | Site | | Visit Date | | Status | |
| /isit Name | | | Subev | ent# | CRF Name | | • | Blan |
| 01 | No<br>Yes If Y | es, please | e ensure ar | | event form has | s been completed fo | | event. |
| | ON₀ | <b>○</b> Yes | Blood and | d Lymphati | c (Including Al | LL Bleeding compli | cations) | |
| | ONo | ○ Yes | Cardiovas | scular - Arri | hythmia | | | |
| | ΟNo | <b>○</b> Yes | Cardiovas | scular - Re | gurgitation | | | |
| | ONo | ○ Yes | Cardiovas | scular - Ste | nosis | | | |
| | ON₀ | ○ Yes | Cardiovas | scular - Em | bolic Event/Va | alve Thrombosis | | |
| | ON₀ | ○ Yes | Cardiovas | scular - Mis | sc | | | |
| | ΟNo | O Yes | Device Dy | ysfunction | | | | |
| | ON₀ | ○ Yes | Gastrointe | estinal/Hep | atic | | | |
| | ONo | ○ Yes | Genitourir | nary/Renal | | | | |
| | ON₀ | ○ Yes | Pulmonar | ry/Respirato | ory | | | |
| | ONo | ○ Yes | Periphera | al Vascular | | | | |
| | ON∘ | ○ Yes | Psychiatri | ic | | | | |
| | ON₀ | O Yes | Muscular | Skeletal/D | ermatologic | | | |

ONo OYes Nonspecific or Unknown Body System

| E Edwards Lifesciences | Study | | | Doc# | | |
|---|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | | Status | | |
| Visit Name | Subevent# | CRF Name | | | Blank | CRF |
| Was there a bleeding-related | d reoperation | within the first | 24 hours after sur | gery? | ON₀ | ○ Yes |
| Please provide the times at | which the foll | owing procedur | al steps were per | formed: | | |
| Start skin incision: | | (HH:MM) | | | | |
| Start ECC (Pump): | | (HH:MM) | | | | |
| Start cross clamp: | | (HH:MM) | | | | |
| Start sizing: | | (HH:MM) | | | | |
| Remove cross clamp: | | (HH:MM) | | | | |
| End ECC (Pump): | | (HH:MM) | | | | |
| End Skin closure: | | (HH:MM) | | | | |
| Comments | | | | | | |

| Edwards Lifesciences | Study | | Doc# | |
|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | |
| Visit Name | Subevent# | CRF Name | _ | Blank CRF |
| DEVICE PERFORMANCE Rev B | | | | |
| What study valve implant attempt was being performed? | | | | |
| Please provide the follow Valve size: Serial Number: | ving information abo | out the study valve: | : | |
| What type of sizer was u | sed? | | | |
| Please specify: | | | | |
| What was the barrel size | of the valve sizer? | mm | | |
| What suture technique w | as used to secure t | he valve? | | |
| Please specify: | | | | |
| How was the valve positi | oned? | | | |
| Did the study valve perfo | orm as intended? | | | |
| Please indicate | the types of valve f | ailures observed: | | |
| Failure type: | | | | |
| Please spe | ecify: | | | |
| Failure type: | | | | |
| Please spe | ecify: | | | |
| Failure type: | | | | |
| L<br>Please spe | ecify: | | | |
| Failure type: | | | | |
| Please spe | ecify: | | | |

| 100 m | | | | | |
|---|---|---|---|---|---|
| Edwards Lifesciences | Study | | | Doc# | |
| Subject ID | Site | Visit Date | | Status | |
| Visit Name | Subevent# | CRF Name | | | Blank CRF |
| DEVICE TECHNICAL SUCCE | ESS: | | | | |
| Did the subject leave the | operating room wit | h the study v | alve in place for | this attempt? | • |
| O No | | | | | |
| Why did the imp | lant attempt fail? | | | | |
| | specify: | | | | |
| Was the heart re | estarted after this in | mplant attem | pt? ONo ( | Yes | |
| O Yes | | | | | |
| VALVE IMPLANT TIMES: | | | | | |
| Start the study procedure | (first stitch): | | | | |
| | (HH:MN | 1:SS) | | | |
| Complete the study proce | dure (last stitch tie | d down on th | e valve): | | |
| | (HH:MN | 1:SS) | | | |
| Comments | | | | | |

| E Edwards Lifesciences | Study GLX_EXT_2 | 2010 03 | Doc# | |
|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | |
| Visit Name DISCHARGE | Subevent# | CRF Name DISCHAR | GE | Blank CRF |
| | DISCH | ARGE | | Version A |
| Date of discharge | (DD/MMM | I/YYYY) | | |
| Where was the subject disc | charged to? | | | |
| Please provide the following valve procedure | g information abo | ut the subject's hosp | italization after the | study |
| Duration of time in the In | tensive Care Unit (I | CU) | | |
| Days | and Hours | | | |
| Duration of time in the In | termediate Care / H | ligh Dependency Unit | | |
| Days | and Hours | | | |
| Duration of time in the G | eneral Ward | | | |
| Days | and Hours | | | |
| When was the transthoracic | echocardiogram (TT | E) performed? | | |

| Edwards Lifesciences Study | Doc# |
|---|---|
| Subject ID Site Visit Date | Status |
| /isit Name Subevent# CRF Name | Blank CRF |
| ADVERSE EVENT | Rev B |
| Event Onset Date (DD/MMM/YYYY) Site Awareness Date (DD/MMM/YYYY) Timing of Event Onset | |
| Please select the AE Classification: O Blood and Lymphatic (Including ALL Bleeding complications) | |
| C Blood and Lymphado (moldang ALL Blooding complications) | |
| Cardiovascular - Arrhythmia | |
| O Cardiovascular - Regurgitation | |
| O Cardiovascular - Stenosis | |
| Cardiovascular - Embolic Event/Valve Thrombosis | |
| O Cardiovascular - Misc | |
| O Device Dysfunction | |
| O Gastrointestinal/Hepatic | |
| O Genitourinary/Renal | |
| O Pulmonary/Respiratory | |
| O Peripheral Vascular | |
| O Psychiatric | |
| Muscular Skeletal/ Dermatologic | |
| Nonspecific or Unknown Body System | |

| E Edwards Lit | escience | s | Study Doc# |
|---|---|---|---|
| Subject ID | | | Site Visit Date Status |
| Visit Name | | | Subevent# CRF Name Blank CRF |
| Event Sum | manulC | omme | ante |
| Event Sum | mar y/C | , Cilling | anta - |
| Method of | Detecti | on | |
| O No | 0 | Yes | Lab finding |
| O No | 0 | Yes | Echocardiogram |
| O No | 0 | Yes | Angiogram |
| | | | Date of Angiogram: (DD/MMM/YYYY) |
| O No | 0 | Yes | MRI |
| | _ | | Date of MRI: (DD/MMM/YYYY) |
| O No | _ | Yes | Electrocardiogram (ECG) |
| O No | _ | Yes | Autopsy |
| O No | 0 | Yes | Observation |
| • | _ | | Date AE first observed: (DD/MMM/YYYY) |
| O No | 0 | Yes | Clinical Exam |
| O 11 | _ | | Date of Clinical Exam: (DD/MMM/YYYY) |
| O No | , 0 | Yes | Re-operation CD (CD (MANAGE) CD (MANAGE) C |
| <b>~</b> | _ | | Date of Re-operation: (DD/MMM/YYYY) |
| O No | . 0 | Yes | Other method |
| | | | Please, specify: |

| E Edward | s Lifescie | ences | | Stud | у | | | | Doc# | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | | | | Site | | Visit | Date | | Status | | |
| Visit Name | | | | Sube | event# | CRF | Name | | | Blank C | RF |
| Causali | t la tl | .i | t | lated to | anu of the f | iallawi | 2 | | | | |
| Causaii | ty: is tr<br>No | _ | | _ | any of the feterminate | | - | l Procedure | | | |
| 0 | No | _ | Yes<br>Yes | _ | eterminate | | • | | | | |
| 0 | No | _ | Yes | _ | eterminate | | Study \<br>User Er | | | | |
| 0 | No | _ | Yes | _ | eterminate | | | | | | |
| 0 | No | _ | | _ | eterminate | | | ncy in Instructio | IIIS | | |
| O | NO | • | | _ | | | Onderly | ring Condition | | | _ |
| | | vvna | ı wası | ne unde | rlying condition | OH! | | | | | |
| Did | antithre | ombo | tic me | dication | contribute to | this ev | ent? | O No O | Yes | | |
| | Was th | nis m | edication | on preso | ribed due to | study | valve in | nplant? O N | lo () | Yes . | |
| | Please | indi | cate wi | hat type | s) of medicat | tion co | ntribute | d to this event: | | | |
| | C | ) No | 0 | Yes | Anticoagula | nt med | dication | | | | |
| | C | ) No | 0 | Yes | Aspirin | | | | | | |
| | C | ) No | 0 | Yes | Other antiple | atelet i | medicat | tion | | | |
| | C | ) No | 0 | Yes | Other antith | rombo | tic med | ication | | | |
| | | | | | Please | , speci | fy: | | | | $\neg$ |
| | | | | | | | L | | | | |
| Did | non-ar | ntithro | mbotio | medica | tion contribut | te to th | is even | t? O No | O Yes | | |
| | Please | e, spe | cify: | | | | | | | | $\neg$ |
| | | | Į | | | | | | | | |
| ls ti | his a se | rious | advers | se event | (SAE)? O | No | O Y | 'es | | | |
| | Please | indi | cate all | condition | ons of a SAE | that a | oply: | | | | |
| | C | ) No | 0 | Yes | Resulted in | death | | | | | |
| | C | ) No | 0 | Yes | Resulted in | life-thr | eatenin | g illness/injury | | | |
| | C | ) No | 0 | Yes | Resulted in | perma | nent im | pairment | | | |
| | C | ) No | 0 | Yes | Resulted in | hospit | alization | n or prolongatio | n or curren | ıt hospitaliza | ition |
| | С | ) No | 0 | Yes | Resulted in body structu | | | ention to preve | ent perman | ent impairme | ent to |
| | С | ) No | 0 | Yes | Resulted in defect | fetal d | istress | or death, conge | enital abnor | mality or bir | th |
| | С | ) No | 0 | Yes | Resulted in to body stru | | | ervention to pre | vent perma | nent impairr | ment |

| Edwards | Life | science | S | | Study Doc# |
|---|---|---|---|---|---|
| Subject ID | | | | | Site Visit Date Status |
| /isit Name | | | | | Subevent# CRF Name Blank CRF |
| Is this a | ı un | antici | inate | d devi | rice related adverse effect (UDAE)? O No O Yes |
| | | | | | to treat this adverse event? O No O Yes |
| | | | | | the following interventions were needed: |
| | 0 | No | 0 | Yes | Prolonged hospitalization |
| | 0 | No | 0 | Yes | Re-hospitalization required |
| | | | | | Hospital admission date: (DD/MMM/YYYY) |
| | | | | | Was the subject discharged from the hospital? O No O Ye |
| | | | | | Discharge date: (DD/MMM/YYYY) |
| | 0 | No | 0 | Yes | Cardioversion |
| | 0 | No | 0 | Yes | Transfusion |
| | 0 | No | 0 | Yes | Medication given |
| | | | | | What type of medication was given? |
| | 0 | No | 0 | Yes | Permanent Pacemaker implanted (not planned prior to AVR) |
| | | | | | Date of pacemaker implant: (DD/MMM/YYYY) |
| | 0 | No | 0 | Yes | Surgical intervention - reoperation on the study valve |
| | | | | | Date of surgical intervention: (DD/MMM/YYYY) |
| | | | | | Was this adverse event the primary cause of O No O Ye reoperation on the study valve? |
| | | | | | Did the reoperation result in O No O Yo removal/replacement of the study valve? |
| | 0 | No | 0 | Yes | Surgical intervention - not reoperation on the study valve |
| | | | | | Date of surgical intervention: (DD/MMM/YYYY) |
| | 0 | No | 0 | Yes | Other intervention |
| | | | | | Please, specify: |
| Indicate | the | outco | ome o | of the | event: |
| | | | | | Date resolved: (DD/MMM/YYYY) |

| Edwards Lifesciences | Study | | | Doc# | | |
|---|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | | Status | | $\neg$ |
| /isit Name | Subevent# | CRF Name | | | Blank CRF | |
| | BLOO | DATA (LAB | 3S) | | Rev | В |
| Date Blood Drawn: | (DI | D/MMM/YYYY) | ) | | | |
| White Blood Cells (WBC) Is this value within norm Was the result clinic | | | O Not Applicat | ble | | |
| Red Blood Cells (RBC) Is this value within norm Was the result clinic | | | Not Applicat | ble | | |
| Hemoglobin: Is this value within norm Was the result clinic | | | O Not Applicat | ble | | |
| Hematocrit: Is this value within norm Was the result clinic | | No O Yes | O Not Applical | ble | | |
| Platelet Count: Is this value within norm Was the result clinic | _ | _ | O Not Applicat | ble | | |
| Plasma Free Hemoglobin: Is this value within norm Was the result clinic | | _ | O Not Applical O Yes | ble | | |
| Coagulation Profile INR: PTT: PT (seconds): | | | | | | |

| Edwards Lifescie Subject ID Visit Name BASELII | | Sit | | | Visit Date Status Blank CRF Blank CRF |
|---|---|---|---|---|---|
| MEDICATIONS Version A Date Information Collected: (DD/MMM/YYYY) Please indicate what type of medications the subject is currently taking: | | | | | |
| O No O Ye | ease indic | ate if th | e sul | bject is | oolytics) taking anticoagulants: O No O Yes f anticoagulant(s): |
| | 0 0 0 | No<br>No<br>No<br>No | 0 0 | Yes<br>Yes<br>Yes<br>Yes | Warfarin - Coumadin (or derivatives) Heparin Low Molecular Weight Heparin Other anticoagulant |
| | | | | | e specify: |
| Ple | | | | | taking antiplatelets: O No O Yes |
| | 0 | No | 0 | Yes | Dipyridamole - Persantine |
| | 0 | No | 0 | Yes | Aspirin - Ecotrin or Entrophen |
| | 0 | No | 0 | Yes | Ticlopidine |
| | 0 | No | 0 | Yes | Clopidogrel-Plavix |
| | 0 | No | 0 | Yes | Other antiplatelet |
| | | | | Please | e specify: |

| and the same of th | | | | |
|---|---|---|---|---|
| Edwards Lifes | ciences | Study GLX_EXT_ | 2010_03 | Doc# |
| Subject ID | | Site | Visit Date | Status |
| Visit Name BASE | ELINE | Subevent# | CRF Name MEDICATIO | NS Blank CRF |
| O No C | Yes ACI | E or ARB Inhibitors | | |
| O No C | Yes Ant | iarrhythmics | | |
| | Please ind | icate if the subject is | taking the following antian | hythmics: |
| | ON | lo 🔘 Yes Beta | Blockers (Propanolol, Es | nolol) |
| | O N | lo O Yes Othe | er (Sodium/Potassium cha | nnel blockers, i.e. Amiodarone) |
| O No C | Yes Cal | cium Blocker | | |
| O No C | ) Yes Diu | retic | | |
| O No C | Yes Lipi | d Lowering | | |
| O No C | ) Yes Nitr | ates | | |
| O No C | Yes Ste | roids | | |

| E Edwards | Lifesciences Study GLX_EXT_2010_03 Doc# |
|---|---|
| Subject ID | Site Visit Date Status |
| Visit Name | BASELINE Subevent# CRF Name ECG Blank CRF |
| | ELECTROCARDIOGRAM (ECG) EXAM Version A |
| Date of ele | ectrocardiogram (ECG) exam: (DD/MMM/YYYY) |
| Is the sub | ject implanted with a permanent pacemaker? ONO OYes Please specify the type: |
| Dose the | subject have an implantable cardioverter defibrillator (ICD/AICD)? ONO OYes |
| Please inc | dicate if the following cardiac rhythms were observed during the ECG: |
| O No | O Yes Sinus rhythm with no abnormalities |
| O No | ○ Yes Sinus tachycardia |
| O No | O Yes Sinus bradycardia |
| O No | Yes Atrial fibrillation / Supraventricular tachycardia |
| | Please indicate the episodic pattern: |
| O No | ○ Yes Atrial flutter |
| O No | Yes Tachycardia-bradycardia syndrome |
| O No | ○ Yes Ventricular tachycardia |
| | Please indicate the episodic pattern: |
| O No | Yes Other cardiac arrhythmia Please specify: |
| Please inc | dicate if evidence of the following conduction disturbances was found during exam: |
| O No | ○Yes AV block |
| | Please indicate degree: |
| O No | ○Yes Bundle branch block / Intraventricular block |
| | Please indicate branch: |
| | Left ONo OYes |
| | Right ONo OYes |
| O No | O Yes Other conduction disturbance |
| | Please specify: |

| E Edward | s Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|---|
| Subject ID | | Site | Visit Date | | Status | |
| Visit Name | | Subevent# | CRF Name | | | Blank CRF |
| | | QUALI | TY OF LIFE | • | | Revision A |
| QUALIT | Y OF LIFE (QOL) AS | SESSMENT | | | | |
| Was an | EQ-5D questionnaire | completed? ONo | Yes | | | |
| EQ | -5D Questionnaire | | | | | |
| Dat | e of assessment | (DI | D/MMM/YYY | Y) | | |
| Ind | icate which statemer | nt the subject mar | ked on the | survey: | | |
| Mol | bility | | | | | |
| Self | f-care | | | | | |
| Usi | ual Activities (e.g. wor | k. studv. housewor | k family or le | eisure activities) | | |
| | iai / totavities (o.g. won | n, olday, modeonor | n, ranny or n | Jiouro donvinos, | | |
| Pai | n/Discomfort | | | | | |
| _ | | | | | | |
| Anx | ciety/Depression | | | | | |
| Ove | erall State (Indicate ho | ow the subject rate | d their overa | ll health today) | | |
| Comme | ents: | | | | | |

| Edwards Lifesciences | Study | | | Doc# | | |
|---|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | | Status | | $\neg$ |
| Visit Name | Subevent# | CRF Name | | | Blank CRF | |
| Was an SF-12-v2 questionn | naire completed?( | ONo OYes | | | | |
| SF-12 v2 Questionnai | re | | | | | |
| Date of assessment | ( | DD/MMM/YYY | Y) | | | |
| Indicate which statem | ent the subject n | narked on the | survey: | | | |
| 1. In general, would you | u say your health is | s: | | | ] | |
| <ol><li>The following question now limit you in these a</li></ol> | | | do during a typical | l day. Does | your health | |
| <ul> <li>a. Moderate activit<br/>or playing golf.</li> </ul> | ties, such as movir | ng a table, push | ning a vacuum clea | iner, bowlin | g, | |
| b. Climbing severa | al flights of stairs | | | | | |
| 3. During the past 4 we with your work or other | | | | | roblems | |
| a. Accomplished le | ess than you would | like | | | | |
| b. Were limited in | the kind of work or | other activities | | | | |
| <ol> <li>During the past 4 we<br/>your work or other regu<br/>depressed or anxious)?</li> </ol> | ılar daily activities a | | | | | ı |
| a. Accomplished le | ess than you would | l like | | | | |
| b. Did work or activ | vities less carefully | than usual? | | | | ] |
| 5. During the past 4 we outside the home and h | | d pain interfere | with your normal w | vork (includi | ing both wor | k |
| <ol><li>These questions are<br/>weeks. For each questi<br/>feeling. How much of the</li></ol> | ion, please give on | e answer that | comes closest to the | | | |
| a. Have you felt ca | alm and peaceful? | | | | | |
| b. Did you have a | lot of energy? | | | | | |
| c. Have you felt do | wnhearted and de | pressed? | | | | |
| 7. During the past 4 we interfered with your soc | eks, how much of<br>cial activities (like v | the time has yo<br>isiting friends, | our physical health<br>relatives, etc.)? | or emotiona | al problems | |
| Comments | | | | | | |

| E Edwards Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|
| | . ' | | | <u>'</u> | |
| Subject ID | Site | Visit Date | | Status | |
| Visit Name | Subevent# | CRF Name | | | Blank CRF |
| | SITE ECHO<br>******* NO | O TRACKIN | | | Rev B |
| Date of ECHO Exam: | | | | | |
| Name of the Echocardiograph | ner: | | ] | | |
| ECHO Equipment used: | | | | | |
| F | Please specify: | | | | |
| Please provide the following p | hysical assessmen | t parameters | 3: | | |
| Weight: Kg | O Ip | | | | |
| Heart Rate (BPM): | | | | | |
| Blood Pressure (mmHg): | Systolic | / [ | Diastolic | ٦ | |
| Cardiac Rhythm: | | | | _ | |
| Date echocardiographs were | delivered to the Co | re Lab: | | | |
| Delivery Method: | | | | | |
| Please spec | sify: | | | | |
| Shipment Ti | acking Number: | | | | |

| Edwards I | Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|---|
| Subject ID | | Site | Visit Date | | Status | |
| Visit Name | | Subevent# | CRF Name | | | Blank CRF |
| | | <u> </u> | • | | | <u>-</u> |
| Did the ed | chocardiographer as | sess the aortic val | ve? O No | O Yes | | |
| Pleas | se indicate the result | ts of the LVOT asse | essment | | | |
| F | Peak Velocity | | | | | |
| F | Peak Gradient | | | | | |
| ľ | Mean Gradient | | | | | |
| \ | VTI | | | | | |
| Pleas | se indicate the result | ts of the aortic valve | e assessment | | | |
| | Peak Velocity | | | | | |
| | Peak Gradient | | | | | |
| | Mean Gradient | | | | | |
| | /ті 🗀 | | | | | |
| | What was the annulu | · · · <u></u> | | | | |
| V | What was the AV are | ea (cm^2)? | | | | |
| Pleas | se indicate the AR S | everity: | | | | |
| Pleas | se indicate the MR S | Severity: | | | | |
| What | was the LVEF? | | | | | |
| What | was the range of th | e LVEF? Max | Value: | | | |
| | | Min \ | /alue: | | | |
| What | method was used to | o determine the LV | EF? | | | |
| Pleas | se indicate the sever | rity of paravalvular | leak (PVL): | | | ] |
| Pleas | se indicate the trans | valvular leak severi | ty: | | | |
| What | was the assessmer | nt of RV function? | | | | |

| Edwards Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|
| Subject ID | Site | | Visit Date | Status | |
| Visit Name | Subev | ent# | CRF Name | | Blank CRF |
| | ЕСНО | CORE LA | AB RESULTS (Baseline) | | Rev B |
| Date of ECHO Exam | | | | | |
| Date ECHO Received by Co | re Lab [ | | | | |
| Date of Readability Assessm | ent | | | | |
| Please indicate whether or n | ot the im | ages were | readable: | | |
| Was a request sent to the | e site to | resend the | images? ONo OYes | | |
| Date of resend | request | : | | | |
| Was the readability issue | e resolve | ed? O No | ○ Yes | | |
| Date readability | / issue r | esolved: | | | |
| Was the ECHO Assessed by | the Cor | e Lab? O | No OYes | | |
| Physical Assessment | | | | | |
| Height Unit | | | | | |
| Weight Unit | | $\neg$ | | | |
| Body Surface Area (BSA | N) [ | 〒 | | | |
| Heart Rate (BPM) | ¬ | | | | |
| Blood pressure (mmHg) | Sy | stolic | / Diastolic | | |
| Does the Echo indicate the system disturbances? | subjec | t has the fo | ollowing cardiac rhythm / con | ducting | |
| Normal Sinus Rhythm | O No | O Yes | OIndeterminate | | |
| Atrial Fibrillation | O No | O Yes | OIndeterminate | | |
| Atrial Flutter | O No | O Yes | OIndeterminate | | |
| Ventricular Tachycardia | O No | ○ Yes | OIndeterminate | | |
| Ventricular Fibrillation | O No | O Yes | OIndeterminate | | |
| AV Block | ON₀ | O Yes | O Indeterminate | | |
| | | Please | e indicate the degree: | | |
| Bundle Branch Block | O No | O Yes | OIndeterminate | | |
| | | Pleas | e indicate branch: | | |

| E Edwards Lifesciences | Study | | Doc# | |
|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | |
| Visit Name | Subevent# | CRF Name | | Blank CRF |
| Aortic Valve Assessment Please indicate the lev | rel of Aortic Stenosis: | : | | |
| LV Structure / Regional F | unction | | | |
| | y of the following ab | normalities were ob | served: | |
| LV aneurysm O | | | | |
| Please spe | cify the location: | | | |
| | L | | | |
| Wall motion abnor | mality O No O | Yes | | |
| Please spe | cify: | | | |
| Cavity dilation ( | No OYes | | | |
| Apical and/or left | atrial thrombi ONo | Yes | | |
| Other abnormality | ONo OYes | | | |
| Please spe | cify: | | | |
| Global LV Structure / Fu | nction | | | |
| What method of calcu | lation was used for L | V function assessn | nent? | |
| LVEDV (ml): | | | | |
| LVESV (ml): | | | | |
| LVEF (%): | | | | |
| LV Dimensions | | | | |
| Septal thickness (end- | -diastolic) (cm): | | | |
| Posterior wall thickness | ss (end-diastolic) (cm | 1): | | |
| LV end-diastolic dime | nsion (cm): | | | |
| LV end-systolic dimen | sion (cm): | | | |
| LV Mass (g): | | | | |
| BSA corrected LV ma | ss (g/m^2): | | | |

| Edwards Lifessianes | Obs. I | | | | | ь | |
|---|---|---|---|---|---|---|---|
| E Edwards Lifesciences | Study | | | | | Doc# | |
| Subject ID | Site | | Visit Date | | | Status | |
| Visit Name | Subevent# | | CRF Name | | | | Blank CRF |
| • | | | | | | | |
| Aortic Dimensions | | | | | | | |
| LVOT Diameter (cm): | | | | | | | |
| Aortic annulus (cm): | | | | | | | |
| Aortic root diameter (cm): | | | | | | | |
| STJ diameter (cm): | | | | | | | |
| Aortic Valve Assessment: M | easuremen | ts | | | | | |
| VpeakAO (m/sec): | | | | | | | |
| TVI (AO) (cm): | | | | | | | |
| Peak systolic gradient of A | AV (by conti | nuous v | wave) (mmH | g): | | | |
| Mean systolic gradient of | AV (by conti | inuous | wave) (mml | lg): | | | |
| TVI (LVOT) (cm): | | | | | | | |
| Maximum V(LVOT) (m/se | c): | | ] | | | | |
| Mean V(LVOT) (m/sec): | | | ] | | | | |
| Stroke Volume (LVOT De | rived) (ml): | | | | | | |
| Transvalvular flow (ml/s): | | | | | | | |
| Cardiac Output (LVOT de | rived) (L/mir | 1): | | ] | | | |
| Cardiac Index (L/min/m^2 | ): | | ] | | | | |
| Aortic EOA (continuity equ | uation) (cm^ | 2): | | ] | | | |
| Aortic EOA Index (cm^2/n | n^2): | | | | | | |
| Performance Index: | | | | | | | |
| Aortic Valve Assessment: Re | egurgitatio | n | | | | | |
| Please identify all the met | hods of calc | ulation | used: | | | | |
| Color Doppler O No | Yes | | | | | | |
| Regurgitant Fraction | O No | 0 | Yes | | | | |
| Proximal Convergent | Flow O No | 0 | Yes | | | | |
| Continuous wave dop | pler (Pressi | ure half | f-time) ON | No | O Yes | | |
| Aortic Flow Reversal | ONG | 0 | Yes | | | | |

| Edwards Lifescier | ices S | tudy | | Doc# | |
|---|---|---|---|---|---|
| Subject ID | s | ite | Visit Date | Status | ; |
| /isit Name | s | ubevent# | CRF Name | | Blank CRF |
| Ple<br>Ple | PSAX C | e Number of Jets cify: e location of the e image views of No Yes No Yes No Yes No Yes No Yes | jets: | | |
| Please indic | ate the total reg | jurgitation sever | ity | | ] |
| Please indic | re Regurgitation<br>ate the level of the late the level of l | Tricuspid Valve<br>Mitral Valve Reç | | | |
| Pericardial Effu | | | | | |
| | cate the level of<br>Please specify: | Pericardial Effu | sion: | | |
| RV Function | | | | | |
| Please indic | ate overall asse | essment of the R | Right Ventricle: | | $\neg$ |

| Edwards Lifesciences | Study | | Doc# | | |
|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | | |
| Visit Name | Subevent# | CRF Name | | Blank CRF | |
| | | | | | _ |
| ECHO Quality | | | | | |
| Please indicate the over | rall Quality of the EC | HOs: | | | |
| Comments | | | | | |
| | | | | | 7 |
| | | | | | ╛ |
| ı | | | | | |
| E Edwards Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|
| Subject ID | Site | $\overline{}$ | Visit Date | Status | |
| Visit Name | Subevent | # | CRF Name | , L | Blank CRF |
| 5 / /50V0 5 | EC | но соғ | RE LAB RESULTS | | Rev B |
| Date of ECHO Exam | | | | | |
| Date ECHO Received by Cor | | | | | |
| Date of Readability Assessment Please indicate whether or no | _ | es were r | readable: | | |
| Was a request sent to the | e site to re | send the | images? ONo OYes | | |
| Date of resend | request: | | | | |
| Was the readability issue | resolved? | ONo | ○ Yes | | |
| Date readability | issue reso | olved: | | | |
| Was the ECHO Assessed by | the Core L | ab? ()1 | No OYes | | |
| Physical Assessment | | | | | |
| Height Unit Weight Unit | | ] | | | |
| Body Surface Area (BSA | ) <del> </del> | _ | | | |
| Heart Rate (BPM) | <u></u> | | | | |
| | | — | / Diagtalia | | |
| Blood pressure (mmHg) | Systol | lic | / Diastolic | | |
| Does the Echo indicate the system disturbances? | subject h | as the fo | llowing cardiac rhythm / con | ducting | |
| Normal Sinus Rhythm | O No | O Yes | OIndeterminate | | |
| Atrial Fibrillation | O No | O Yes | OIndeterminate | | |
| Atrial Flutter | O No | O Yes | OIndeterminate | | |
| Ventricular Tachycardia | O No | O Yes | OIndeterminate | | |
| Ventricular Fibrillation | O No | O Yes | OIndeterminate | | |
| AV Block | O No | O Yes | OIndeterminate | | |
| | | Please | e indicate the degree: | | |
| Bundle Branch Block | O No | O Yes | OIndeterminate | | |
| | | Pleas | e indicate the branch: | | |

| E Edwards Lifesciences | Study | | | Doc# | | |
|---|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | | Status | | $\exists$ |
| Visit Name | Subevent# | CRF Name | | | Blank CRF | |
| Aortic Valve Assessment | : Stenosis | | | | | |
| Please indicate the lev | _ | | | $\neg$ | | |
| LV Structure / Regional F | _ | | | | | |
| _ | y of the following abnor | malities wer | e observed: | | | |
| LV aneurysm O | | | | | | |
| | cify the location: | | | | | ٦ |
| Wall motion abnor | mality ONo OYe | s | | | | |
| Please spe | | | | | | ٦ |
| · | | | | | | |
| | | | | | | J |
| Cavity dilation ( | No O Yes | | | | | |
| Apical and/or left | atrial thrombi O No | <b>○</b> Yes | | | | |
| Other abnormality | ONo OYes | | | | | |
| Please spe | cify: | | | | | 7 |
| | | | | | | ┙ |
| Global LV Structure / Fur | nction | | | | | |
| What method of calcu | lation was used for LV f | unction asse | essment? | | | |
| LVEDV (ml): | | | | | | |
| LVESV (ml): | | | | | | |
| LVEF (%): | | | | | | |
| LV Dimensions | | | | | | |
| Septal thickness (end- | -diastolic) (cm): | | | | | |
| Posterior wall thickness | ss (end-diastolic) (cm): | | | | | |
| LV end-diastolic dime | nsion (cm): | | | | | |
| LV end-systolic dimen | sion (cm): | | | | | |
| LV Mass (g): | | | | | | |
| BSA corrected LV ma | ss (g/m^2): | $\neg$ | | | | |

| Edwards Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|
| | . ' | | | | |
| Subject ID | Site | Visit Date | | Status | |
| Visit Name | Subevent# | CRF Name | | | Blank CRF |
| Aortic Dimensions | | | | | |
| LVOT Diameter (cm): | | | | | |
| Aortic annulus (cm): | | | | | |
| Aortic root diameter (cm): | | | | | |
| STJ diameter (cm): | | | | | |
| Aortic Valve Assessment: M | easurements | | | | |
| VpeakAO (m/sec): | | | | | |
| TVI (AO) (cm): | | | | | |
| Peak systolic gradient of | AV (by continuous v | vave) (mmHg) | : | | |
| Mean systolic gradient of | AV (by continuous v | wave) (mmHg | ): | $\exists$ | |
| TVI (LVOT) (cm): | | | | | |
| Maximum V(LVOT) (m/se | c): | | | | |
| Mean V(LVOT) (m/sec): | | | | | |
| Stroke Volume (LVOT De | rived) (ml): | | | | |
| Transvalvular flow (ml/s): | | | | | |
| Cardiac Output (LVOT de | rived) (L/min): | | | | |
| Cardiac Index (L/min/m^2 | ): | | | | |
| Aortic EOA (continuity eq | uation) (cm^2): | | | | |
| Aortic EOA Index (cm^2/n | n^2): | | | | |
| Performance Index : | | | | | |
| Aortic Valve Assessment: R | egurgitation | | | | |
| Please identify all the met | - | used: | | | |
| Color Doppler O No | o O Yes | | | | |
| Regurgitant Fraction | _ | | | | |
| Proximal Convergent | Flow O No O | Yes | | | |
| Continuous wave do | opler (Pressure half- | time) O No | O Yes | | |
| Aortic Flow Reversal | ONo OYes | | | | |

| E Edwards | Lifesciences | Study | | Doc# | |
|---|---|---|---|---|---|
| Subject ID | | Site | Visit Date | Status | |
| Visit Name | | Subevent# | CRF Name | | Blank CRF |
| Pleas | se indicate the Parav<br>Please indicate t<br>Please sp | he Number of Jets | | ] | |
| | Please indicate t | he location of the j | ets: | | |
| | Please indicate t | he image views of | the jets: | | |
| | PLAX ( | No OYes | | | |
| | PSAX ( | No OYes | | | |
| | A5C C | No OYes | | | |
| | A3C C | No OYes | | | |
| | se indicate the Trans<br>se indicate the total r | | | | |
| Aortic Va | alve Morphology | | | | |
| Pleas | se indicate the leaflet | mobility: | | | |
| Pleas | se indicate the leaflet | thickening: | | | |
| Pleas | se indicate the degree | e of calcification: | | | |
| Pleas | se indicate whether th | ne following morph | ologies were observe | ed: | |
| | Cusp Perforation | ONo OYes ( | Indeterminate | | |
| | Pannus Formation | ○ No ○ Yes( | Indeterminate | | |
| | Thrombus | ONo OYes ( | Indeterminate | | |
| | Vegetation | ONo OYes ( | Indeterminate | | |
| | Ring Abscess | ONo OYes ( | Indeterminate | | |
| | Pseudoaneurysm | ONo OYes ( | Indeterminate | | |

| E Edwards Lifesciences | Study | | Doc# | | |
|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | | $\overline{\ \ }$ |
| /isit Name | Subevent# | CRF Name | | Blank CRF | |
| | | | | | _ |
| Non-Aortic Valve Regurgita | ation | | | | |
| Please indicate the level | | Regurgitation: | | | |
| Please indicate the level | of Mitral Valve Reg | gurgitation: | | | |
| Pericardial Effusion | | | | | |
| Please indicate the level | of Pericardial Effus | sion: | | | |
| Please speci | fy: | | | | |
| RV Function | | | | | |
| Please indicate overall a | ssessment of the R | Right Ventricle: | | | |
| ECHO Quality | | | | | |
| Please indicate the over | all Quality of the EC | CHOs: | | | |
| Comments | | | | | |
| | | | | | 7 |
| | | | | | ╛ |

| Edwards Lifesciences Study Doc# Subject ID Site Visit Date Status Visit Name Subevent# CRF Name Blank CRF |
|---|
| PROTOCOL DEVIATION (Baseline) Rev B |
| Date of Deviation (DD/MMM/YYYY) |
| Please select type of deviation |
| Please describe the type of deviation What was the reason for the deviation? |
| Please specify: |
| Please indicate the corrective action taken to prevent further deviations |
| Please specify: |

| E Edwards Lifesciences | Study | | | Doc# | |
|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | | Status | |
| Visit Name | Subevent# | CRF Name | | | Blank CRF |
| | PROTO | COL DEVIATION | (Discharge) | | Version A |
| Date of Deviation | (DD/I | MMM/YYYY) | | | |
| Please select type of deviat | ion | | | | |
| Please describe the typ | e of deviation | | | | |
| What was the reason for the | e deviation? | | | | |
| Please | specify | | | | |
| Please indicate the corrective | e action take | n to prevent furthe | er deviations | | |
| Please | specify | | | | |

| Subject ID | Study Doc# Site Visit Date Status CRF Name | Blank CRF |
|---|---|---|
| | PROTOCOL DEVIATION (Procedure) | Version A |
| Date of Deviation | (DD/MMM/YYYY) | |
| Please select type of deviatio | 1 | |
| Please describe the type | of deviation | |
| What was the reason for the | leviation? | |
| Please sp | ecify | |
| Please indicate the corrective | action taken to prevent further deviations | |
| Please spe | cify | |

| Edwards Lifesciences Study Doc# |
|---|
| Subject ID Site Visit Date Status |
| Visit Name Subevent# CRF Name Blank CRF |
| PROTOCOL DEVIATION (3 Month) Version A |
| Date of Deviation (DD/MMM/YYYY) |
| Please select type of deviation |
| Was subject's family or friends contacted? No Please indicate the date when the last attempt to contact the subject was made [DD/MMM/YYYY) Can you confirm through any other sources if the subject is alive? No Yes Yes |
| Date of Contact (DD/MMM/YYYY) Was the subject alive based on the contact? ONO OYes |
| Please describe the type of deviation |
| What was the reason for the deviation? |
| Please specify |
| Please indicate the corrective action taken to prevent further deviations |
| Please specify |

| Edwards Lifesciences Study Doc# |
|---|
| Subject ID Site Visit Date Status |
| Visit Name Subevent# CRF Name Blank CRF |
| PROTOCOL DEVIATION (1 Year) Rev B |
| Date of Deviation (DD/MMM/YYYY) |
| Please select type of deviation |
| Was subject's family or friends contacted? O No Please indicate the date when the last attempt to contact the subject was made |
| (DD/MMM/YYYY) |
| Can you confirm through any other sources if the subject is alive? O No Yes |
| Date of Contact (DD/MMM/YYYY) |
| Was the subject alive based on the contact? O No O Yes |
| Please describe the type of deviation |
| What was the reason for the deviation? |
| Please specify: |
| Please indicate the corrective action taken to prevent further deviations |
| Please specify: |

| Edwards Lifesciences Study Doc# |
|---|
| Subject ID Site Visit Date Status |
| /isit Name Subevent# CRF Name Blank CRF |
| PROTOCOL DEVIATION (2 Year) Version A |
| Date of Deviation (DD/MMM/YYYY) |
| Please select type of deviation |
| Was subject's family or friends contacted? No Please indicate the date when the last attempt to contact the subject was made [DD/MMM/YYYY) Can you confirm through any other sources if the subject is alive? No Yes Date of Contact [DD/MMM/YYYY) Was the subject alive based on the contact? No Yes |
| Please describe the type of deviation |
| What was the reason for the deviation? |
| Please specify |
| Please indicate the corrective action taken to prevent further deviations |
| Please specify |

| III E1 . 1.1% .: | | | | <b>-</b> | | _ |
|---|---|---|---|---|---|---|
| Edwards Lifesciences Stud | У | | | Doc# | | |
| Subject ID Site | | Visit Date | | Status | | $\neg$ |
| Visit Name Sub- | event# | CRF Name | | | Blank CRF | |
| | PROTOCOL | DEVIATION | (3 Year) | | Version A | |
| Date of Deviation | (DD/M | IMM/YYYY) | | | | |
| Please select type of deviation | | | | | | |
| Was subject's family or friend No Please indicate to | he date when | | mpt to contact the | subject \ | was made | _ |
| Can you confirm | | | if the subject is | alive? | ONo OYes | |
| O Yes | an ough any c | varier source. | in the subject is t | a | 01.0010 | • |
| Date of Contact | | (DD | /MMM/YYYY) | | | |
| Was the subject | | | | Yes | | |
| Please describe the type of o | deviation | | | | | |
| What was the reason for the devi | ation? | | | | | |
| Please speci | fy | | | | | |
| Please indicate the corrective act | ion taken to p | revent furthe | r deviations | | | |
| Please speci | fy | | | | | |

| 10 | | | | | | _ |
|---|---|---|---|---|---|---|
| Edwards Lifesciences Stuc | У | | | Doc# | | |
| Subject ID Site | | Visit Date | | Status | | $\neg$ |
| Visit Name Sub | event# | CRF Name | | | Blank CRF | |
| | PROTOCOL | DEVIATION | (4 Year) | | Version A | |
| Date of Deviation | (DD/N | IMM/YYYY) | | | | |
| Please select type of deviation | | | | | | |
| Was subject's family or frien No Please indicate t | he date when | | mpt to contact the | e subject v | was made | _ |
| Can you confirm | | | if the subject is | alive? | ○No ○Yes | |
| O Yes | unough any v | outer source. | on the subject is | unve : | O No O Tes | , |
| Date of Contact | | (DD | /MMM/YYYY) | | | |
| Was the subject | | | | Yes | | |
| Please describe the type of | deviation | | | | | |
| What was the reason for the devi | ation? | | | | | |
| Please speci | y | | | | | |
| Please indicate the corrective act | ion taken to p | revent furthe | r deviations | | | |
| Please specif | У | | | | | 7 |

| E Edwards Lifesciences Stud | | | | ⊐ ⊳# Г | | _ |
|---|---|---|---|---|---|---|
| | <u></u> | | | Doc# | | _ |
| Subject ID Site | | Visit Date | | Status | | |
| Visit Name Sube | event# | CRF Name | | | Blank CRF | |
| | PROTOCOL | DEVIATION | (5 Year) | | Version A | |
| Date of Deviation | (DD/M | IMM/YYYY) | | | | |
| Please select type of deviation | | | | | | |
| Was subject's family or friend No Please indicate t | he date when | | mpt to contact the | subject \ | was made | |
| Can you confirm | | | ' /<br>s if the subject is a | alive? | ONo OYes | |
| O Yes | anough any c | | in the subject to t | | 0.10 0.10 | • |
| Date of Contact | | (DD | /MMM/YYYY) | | | |
| Was the subject | | | | Yes | | |
| Please describe the type of o | leviation | | | | | |
| What was the reason for the devi | ation? | | | | | |
| Please specif | У | | | | | |
| Please indicate the corrective act | ion taken to p | revent furthe | r deviations | | | |
| Please speci | fy | | | | | |

| E Edwards Lifesciences Study | | Doc# |
|---|---|---|
| Subject ID Site | Visit Date | Status |
| Visit Name Sube | vent# CRF Name | Blank CRF |
| ı | ROTOCOL DEVIATION (Miscellaneous) | Version A |
| Date of Deviation | (DD/MMM/YYYY) | |
| Please select type of deviation | | |
| Please describe the type of d | | |
| What was the reason for the devia | tion? | |
| Please specif | | |
| Please indicate the corrective acti | on taken to prevent further deviations | |
| Please specify | | |

| Edwards Lifesciences Subject ID Visit Name | Study Doc# Site Visit Date Status Subevent# CRF Name | Blank CRF |
|---|---|---|
| | PROTOCOL DEVIATION (Adverse Event) | Version A |
| Date of Deviation (DD/MMM/YYYY) | | |
| Please select type of deviat | ion | |
| Please describe the type the t | | |
| Please | specify | |
| Please indicate the corrective | ve action taken to prevent further deviations | |
| Please | specify | |

| E Edward | ds Lifesciences | Study GLX_EXT_201 | 0_03 | Doc# |
|---|---|---|---|---|
| Subject ID | | Site | Visit Date | Status |
| Visit Name | AE | Subevent# | CRF Name REOPERATION | ON Blank CRF |
| Data of | REOP_EXP Version A | | | |
| Did the | the study valve remonstrate surgical procedure of procedu | occur at the investig | | (DD/MMM/YYYY) No O Yes |
| | Please indicate the type of procedure that was performed: If Valve-in-valve replacement or Other is the type of procedure that was performed, please answer questions at the bottom of the next page | | | |
| Whe | n was the device expla | ented? | ANT — | |
| | • | | t procedure? | No ∩Yes |
| | Was information collected about the explant procedure? | | | |
| | What type of aorto<br>(Enter Type or Not | tomy was performed?<br>Available) | | |
| | Were study valve l | eaflets removed? | ONo OYes | O Not Available |
| | Was study valve se | ewing ring removed? | O No O Yes | O Not Available |
| | _ | e explant (Rate ease | on a scale of 1-5, 5 bei | ng the best) |
| | Additional commer | nts: | | |
| ١ | Was a replacement va | lve implanted? | ) No O Yes | |
| | Please provide th | e following informat | tion about the replace | ement valve: |
| | Manufacturer an | d model: | | |
| | Size (mm): | | | |

| Edwards Lifesciences | Study GLX_EXT_ | 2010_03 | | Doc# |
|---|---|---|---|---|
| Subject ID | Site | Visit Date | | Status |
| Visit Name AE | Subevent# | CRF Name | REOPERATION | Blank CRF |
| | | 1 | | |
| Was information colle | cted about the appeara | nce of the val | ve prior to or imme | diately following |
| evolant? | No OYes | | | |
| | whether the following<br>Yes Thrombus | conditions | were observed: | |
| 0 0 | | | | |
| | Yes Vegetation Yes Suture interfe | rence | | |
| | Yes Suture interfe<br>Yes Calcification | rence | | |
| | Yes Fibrosis | | | |
| | Yes Dehiscence | | | |
| 0140 | | | | |
| | Other observ | ations | | |
| Did excision of the stu | dy valve require or resu | ılt in structura | l changes? | |
| ONo OYes | S O Not Available | | | |
| Please sp | ecify: | | | |
| Was the explanted stu | idv valve returned? | O № ( | Yes | |
| Trao tiro oxpiamou oto | ay raive retained. | 0110 | ) les | |
| RGA# | | | | |
| | VALVE-IN-V | ALVE REPLA | ACEMENT - | |
| Please provide the | following information | about the re | eplacement valve: | : |
| Manufacto | urer and model: | | | |
| Size (mm | ٠. ــــــــــــــــــــــــــــــــــــ | | <br>1 | |
| Oize (IIIII) | | | | |
| Please specific F | | OTHER - | | |
| Please specify: | | | | |

| E Edwards Lifesciences | Study GLX_EXT_2 | 010_03 | Doc# |
|---|---|---|---|
| Subject ID | Site | Visit Date | Status |
| Visit Name STUDY_EXIT | Subevent# | CRF Name STUDY EXIT | Blank CRF |
| Date of Study Exit: | | UDY EXIT (DD/MMM/YYYY) | Version A |
| Please indicate when the Please indicate the rea | | | |
| r lease indicate the rea | SOITIOI WILIIUIAWAI. | | |
| Date of Death: | | (DD/MMM/YYYY) | |
| Did the subject die intra | aoperatively during th | ne study procedure? | )No OYes |
| Did the subject die prio | r to discharge from th | ne hospital after the study pro | ocedure? O No O Yes |
| Please provide the | | ation about the subject's ho | spitalization |
| Duration of | time in the Intensive | Care Unit (ICU) | |
| Days: | and Hours: | | |
| | time in the Intermed | iate Care / High Dependency | Unit |
| Duration of | time in the General | Ward | |
| Days: | and Hours: | | |
| Cause of Death: | | | |
| Date reported to the sp | onsor: | (DD/MI | MM/YYYY) |
| Was an autopsy perform | med? ONo ( | Yes | |
| Date of autopsy: | | (DD/MMM/YYYY) | |
| Was a study valve r | removed at autopsy? | If Yes, Please | e fill out the Study Valve<br>placement form (REOP_EXP) |
| Please specify: | | | |

| E Edwards Lifesciences | Study GLX_EXT_ | 2010_03 | Doc# | | |
|---|---|---|---|---|---|
| Subject ID | Site | Visit Date | Status | | |
| Visit Name STUDY_EXIT | Subevent# | CRF Name STUDY EX | Т | Blank CRF | |
| | | | | | _ |
| Comments: | | | | | |



## 15.4 PROTOCOL DEVIATION CODES



#### PROTOCOL DEVIATION CODES

| SUBJECTS | SCREENING | 3 13 | MORE THAN 2 STUDY VALVES ATTEMPTED TO BE IMPLANTED |
|---|---|---|---|
| 1.01 | SUBJECT DID NOT MEET INCLUSION CRITERION | | TIME FIST STITCH PLACED ON THE VALVE NOT RECORDED |
| | SUBJECT MET EXCLUSION CRITERION | | COMPLETION TIME OF STUDY PROCEDURE (LAST STITCH TIED DOWN |
| | DATE OF INFORMED CONSENT IS AFTER DATE OF STUDY ENROLLMENT | | ON THE VALVE) NOT RECORDED |
| 1.04 | INFORMED CONSENT WAS IMPROPERLY OBTAINED | 3.16 | POST-IMPLANT ECHOCARDIOGRAM NOT DONE |
| 1.05 | PERSON OBTAINING INFORMED CONSENT DID NOT SIGN/DATE THE | | POST-IMPLANT ECHOCARDIOGRAM NOT DONE WITHIN 1 HOUR OF |
| 1.00 | CONSENT FORM | | REMOVING THE CROSS-CLAMP |
| 1.06 | OTHER SCREENING DEVIATION | 3.18 | OTHER PROCEDURE DEVIATION |
| BASELINE | | DISCHARG | E |
| 2.01 | BASELINE ECHOCARDIOGRAM NOT DONE | 4.01 | DISCHARGE OR 10-DAY ECHOCARDIOGRAM NOT DONE |
| 2.02 | BASELINE ECHOCARDIOGRAM DONE > 30 DAYS PRIOR IMPLANT DATE | | DISCHARGE OR 10-DAY ECHOCARDIOGRAM DONE > 10 DAYS POST |
| 2.03 | BASELINE BLOOD NOT DONE | | IMPLANT DATE |
| 2.04 | BASELINE BLOOD DONE > 30 DAYS BEFORE IMPLANT | 4.03 | DISCHARGE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE |
| | BASELINE BLOOD INCOMPLETE | 4.04 | DISCHARGE ELECTROCARDIOGRAM NOT DONE |
| 2.06 | BASELINE COAGULATION PROFILE NOT DONE | 4.05 | DISCHARGE COAGULATION PROFILE NOT DONE |
| 2.07 | BASELINE COAGULATION PROFILE DONE > 30 DAYS BEFORE IMPLANT | 4.06 | DISCHARGE MEDICATIONS NOT ASSESSED |
| 2.08 | BASELINE NYHA NOT DONE | 4.07 | OTHER DISCHARGE DEVIATION |
| 2.09 | BASELINE ELECTROCARDIOGRAM NOT DONE | | |
| 2.10 | BASELINE ELECTROCARDIOGRAM DONE > 30 DAYS BEFORE IMPLANT | | |
| 2.11 | BASELINE EQ-5D NOT DONE | 3 MONTHS | |
| 2.12 | BASELINE SF-12 NOT DONE | 6.01 | 3 MONTHS - SUBJECT NOT CONTACTED |
| 2.12 | BASELINE SF-12 NOT DONE<br>BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE | 6.01<br>6.02 | 3 MONTHS - SUBJECT NOT CONTACTED 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW |
| 2.12<br>2.13 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE<br>PREGNACY TEST NOT DONE | 6.02<br>6.03 | |
| 2.12<br>2.13<br>2.14 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE | 6.02<br>6.03<br>6.04 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW |
| 2.12<br>2.13<br>2.14 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE<br>PREGNACY TEST NOT DONE | 6.02<br>6.03<br>6.04<br>6.05 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE |
| 2.12<br>2.13<br>2.14<br>2.15 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION | 6.02<br>6.03<br>6.04 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP |
| 2.12<br>2.13<br>2.14 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY | 6.02<br>6.03<br>6.04<br>6.05<br>6.06 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW |
| 2.12<br>2.13<br>2.14<br>2.15<br><u>IMPLANT S</u><br>3.01 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION | 6.02<br>6.03<br>6.04<br>6.05<br>6.06 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE | 6.02<br>6.03<br>6.04<br>6.05<br>6.06 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP |
| 2.12<br>2.13<br>2.14<br>2.15<br><u>IMPLANT S</u><br>3.01 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08<br>6.09<br>6.10 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05<br>3.06 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED START CROSS CLAMP TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE 3 MONTHS - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05<br>3.06<br>3.07 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED START CROSS CLAMP TIME NOT RECORDED START OF SIZING TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08<br>6.09<br>6.10<br>6.11 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE 3 MONTHS - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR PATIENTS ON ANTICOAGULANT THERAPY) |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05<br>3.06<br>3.07<br>3.08 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED START CROSS CLAMP TIME NOT RECORDED START OF SIZING TIME NOT RECORDED REMOVAL CROSS CLAMP TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08<br>6.09<br>6.10<br>6.11 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE 3 MONTHS - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR PATIENTS ON ANTICOAGULANT THERAPY) 3 MONTHS - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05<br>3.06<br>3.07<br>3.08<br>3.09 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED START CROSS CLAMP TIME NOT RECORDED START OF SIZING TIME NOT RECORDED REMOVAL CROSS CLAMP TIME NOT RECORDED END ECC (PUMP) TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08<br>6.09<br>6.10<br>6.11<br>6.12<br>6.13 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE 3 MONTHS - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR PATIENTS ON ANTICOAGULANT THERAPY) 3 MONTHS - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - MEDICATIONS NOT ASSESSED |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05<br>3.06<br>3.07<br>3.08<br>3.09<br>3.10 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED START CROSS CLAMP TIME NOT RECORDED START OF SIZING TIME NOT RECORDED REMOVAL CROSS CLAMP TIME NOT RECORDED END ECC (PUMP) TIME NOT RECORDED SKIN CLOSURE TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08<br>6.09<br>6.10<br>6.11 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE 3 MONTHS - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR PATIENTS ON ANTICOAGULANT THERAPY) 3 MONTHS - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - MEDICATIONS NOT ASSESSED 3 MONTHS - MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP |
| 2.12<br>2.13<br>2.14<br>2.15<br>IMPLANT S<br>3.01<br>3.02<br>3.03<br>3.04<br>3.05<br>3.06<br>3.07<br>3.08<br>3.09<br>3.10<br>3.11 | BASELINE PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE PREGNACY TEST NOT DONE MEDICAL HISTORY NOT COLLECTED OTHER BASELINE DEVIATION SURGERY IMPLANTING SURGEON IS NOT ON APPROVED LIST PROCEDURE DIAGNOSIS NOT DONE INCORRECT SIZER USED SKIN INCISION TIME NOT RECORDED START TIME OF ECC (PUMP) NOT RECORDED START CROSS CLAMP TIME NOT RECORDED START OF SIZING TIME NOT RECORDED REMOVAL CROSS CLAMP TIME NOT RECORDED END ECC (PUMP) TIME NOT RECORDED | 6.02<br>6.03<br>6.04<br>6.05<br>6.06<br>6.07<br>6.08<br>6.09<br>6.10<br>6.11<br>6.12<br>6.13 | 3 MONTHS - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE 3 MONTHS - NYHA NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE 3 MONTHS - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - ECHOCARDIOGRAM NOT DONE 3 MONTHS - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - BLOOD NOT DONE 3 MONTHS - BLOOD INCOMPLETE 3 MONTHS - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR PATIENTS ON ANTICOAGULANT THERAPY) 3 MONTHS - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW 3 MONTHS - MEDICATIONS NOT ASSESSED |

CONFIDENTIAL AND PROPRIETATARY DATA: This document and the information contained herein may not be reproduced, used, or disclosed without written permission from Edwards Lifesciences LLC



| 1-YEAR | | 3 YEAR | |
|---|---|---|---|
| | EAR - SUBJECT NOT CONTACTED | | 3 YEAR - SUBJECT NOT CONTACTED |
| | EAR - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW | 10.02 | 3 YEAR - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW |
| 8.03 1 Y | EAR - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE | 10.03 | 3 YEAR - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE |
| 8.04 1 Y | EAR - NYHA NOT DONE | 10.04 | 3 YEAR - NYHA NOT DONE |
| 8.05 1 Y | EAR - ELECTROCARDIOGRAM NOT DONE | 10.05 | 3 YEAR - ELECTROCARDIOGRAM NOT DONE |
| 8.06 1 Y | EAR - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP | 10.06 | 3 YEAR - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP |
| WIN | IDOW | | WINDOW |
| 8.07 1 Y | EAR - ECHOCARDIOGRAM NOT DONE | 10.07 | 3 YEAR - ECHOCARDIOGRAM NOT DONE |
| 8.08 1 Y | EAR - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW | 10.08 | 3 YEAR - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW |
| 8.09 1 Y | EAR - BLOOD NOT DONE | 10.09 | 3 YEAR - BLOOD NOT DONE |
| 8.10 1 Y | EAR - BLOOD INCOMPLETE | 10.10 | 3 YEAR - BLOOD INCOMPLETE |
| 8.11 1 Y | EAR - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR | 10.11 | 3 YEAR - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR |
| PAT | TIENTS ON ANTICOAGULANT THERAPY) | | PATIENTS ON ANTICOAGULANT THERAPY) |
| | EAR - BLOOD NOT DONE WITHIN FOLLÓW-UP WINDOW | 10.12 | 3 YEAR - BLOOD NOT DONE WITHIN FOLLÓW-UP WINDOW |
| 8.13 1 YE | EAR - MEDICATIONS NOT ASSESSED | 10.13 | 3 YEAR - MEDICATIONS NOT ASSESSED |
| | EAR - MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW | | 3 YEAR - MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW |
| | EAR - EQ-5D NOT DONE | | 3 YEAR - OTHER DEVIATION |
| | EAR - SF-12 NOT DONE | | |
| | EAR - OTHER DEVIATION | 4 YEAR | |
| | | 11 01 | 4 YEAR - SUBJECT NOT CONTACTED |
| 2 YEAR | | | 4 YEAR - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW |
| 9.01 2 Y | EAR - SUBJECT NOT CONTACTED | | 4 YEAR - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE |
| 9.02 2 Y | EAR - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW | | 4 YEAR - NYHA NOT DONE |
| 9.03 2 Y | EAR - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE | 11.05 | 4 YEAR - ELECTROCARDIOGRAM NOT DONE |
| | EAR - NYHA NOT DONE | | 4 YEAR - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP |
| 9.05 2 Y | EAR - ELECTROCARDIOGRAM NOT DONE | | WINDOW |
| | EAR - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP | 11.07 | 4 YEAR - AUSCULTATION NOT DONE |
| | IDOW | | 4 YEAR - ECHOCARDIOGRAM NOT DONE (AUSCULTATION INDICATED |
| 9.07 2 YE | EAR - AUSCULTATION NOT DONE | | AORTIC MURMUR) |
| | EAR - ECHOCARDIOGRAM NOT DONE (AUSCULTATION INDICATED | 11.09 | 4 YEAR - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW |
| | RTIC MURMUR) | | (AUSCULTATION INDICATED AORTIC MURMUR) |
| | EAR - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW | 11.10 | 4 YEAR - BLOOD NOT DONE |
| | SCULTATION INDICATED AORTIC MURMUR) | | 4 YEAR - BLOOD INCOMPLETE |
| | EAR - BLOOD NOT DONE | | 4 YEAR - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW |
| | EAR - BLOOD INCOMPLETE | | 4 YEAR - MEDICATIONS NOT ASSESSED |
| | EAR - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW | | 4 YEAR - MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW |
| | EAR - MEDICATIONS NOT ASSESSED | | 4 YEAR - OTHER DEVIATION |
| | EAR - MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW | | |

Edwards Pericardial Aortic Bioprosthesis, Model 11000

Clinical Trial Number: 2010-03



#### 5 YEAR

12.01 5 YEAR - SUBJECT NOT CONTACTED
12.02 5 YEAR - ASSESSMENT NOT DONE WITHIN FOLLOW-UP WINDOW
12.03 5 YEAR - PHYSICAL ASSESSMENT / VITAL SIGNS NOT DONE
12.04 5 YEAR - NYHA NOT DONE
12.05 5 YEAR - ELECTROCARDIOGRAM NOT DONE
12.06 5 YEAR - ELECTROCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
12.07 5 YEAR - ECHOCARDIOGRAM NOT DONE
12.08 5 YEAR - ECHOCARDIOGRAM NOT DONE WITHIN FOLLOW-UP WINDOW
12.09 5 YEAR - BLOOD NOT DONE
12.10 5 YEAR - BLOOD INCOMPLETE
12.11 5 YEAR - COAGULATION PROFILE NOT DONE (ONLY REQUIRED FOR PATIENTS ON ANTICOAGULANT THERAPY)
12.12 5 YEAR - BLOOD NOT DONE WITHIN FOLLOW-UP WINDOW
12.13 5 YEAR - MEDICATIONS NOT ASSESSED
12.14 5 YEAR - MEDICATIONS NOT ASSESSED WITHIN FOLLOW-UP WINDOW
12.15 5 YEAR - OTHER DEVIATION



## 15.5 DEVICE DEFICIENCY CODES



#### **DEVICE DEFICIENCY CODES**

| Code | Label |
|---|---|
| DD.2 | Valve / Holder |
| DD.2.01 | Device function, packaging not intact |
| DD.2.02 | Device function, component contamination |
| DD.2.03 | Device function, unable to remove from jar |
| DD.2.04 | Device function, unable to place sutures through sewing ring |
| DD.2.05 | Device function, unable to position on the aortic annulus |
| DD.2.06 | Device function, bioprosthesis and holder separate during procedure |
| DD.2.07 | Device function, other, specify |
| DD.2.08 | Device use, sizing technique |
| DD.2.09 | Device use, sterility compromised |
| DD.2.10 | Device use, used expired product |
| DD.2.11 | Device use, component damaged by operator |
| DD.2.12 | Device use, improper positioning |
| DD.2.13 | Device use, other specify |

Edwards Pericardial Aortic Bioprosthesis, Model 11000 Clinical Trial Number: 2010-03

Edwards

#### 15.6 ECHO MANUAL



Clinical Study Number: 2010-03

## **Table of Contents**

| 1 | Purr | oose | 2 |
|---|-------|----------------------------------------------|---|
| | _ | | |
| 2 | Intro | oduction | 2 |
| 3 | Trar | nsthoracic echocardiogram (TTE) | 2 |
| | 3.1 | Performing the exam | |
| | 3.2 | Exam view sequence | |
| | 3.3 | Data collection | |
| | | nsesophageal echocardiogram (TEE) | |
| • | IIai | isesopriagear ecriocardiogram (TEL) | |
| | 4.1 | Performing the exam | 4 |
| | 4.2 | Exam view | 4 |
| | 4.3 | Data collection | |
| | | reviated Transthoracic Echocardiogram (aTTE) | |
| • | ADD | | |
| | 5.1 | Performing the exam | |
| | 5.2 | Exam view sequence | 5 |
| | 5.3 | Data collection | C |



Clinical Study Number: 2010-03

#### 1 Purpose

The purpose of this Echo Manual is to provide instruction on study echocardiograms for clinical sites participating in the #2010-03 clinical study.

#### 2 Introduction

There are three types of echocardiographic exams required in the #2010-03 clinical study protocol:

- Transthoracic echocardiogram (TTE)
- Transesophageal echocardiogram (TEE)
- Abbreviated transthoracic echocardiogram (aTTE)

| Investigation<br>Procedure | Baseline | Implant | Discharge | 3<br>month | 1, 3, 5<br>year | 2 & 4<br>years |
|---|---|---|---|---|---|---|
| TTE | Х | | X | X | X | |
| TEE | | Χ | | | | |
| aTTE | | Χ | | | | X |

#### 3 Transthoracic echocardiogram (TTE)

#### 3.1 Performing the exam

Study subjects are typically examined in the left lateral decubitus or supine position. All views are to be acquired twice for 3 beats.

The sweep speed for all spectral Doppler and M-mode recordings should be 100 mm/sec. Nyquist settings for color Doppler assessment of the cardiac valves should be >50 cm/sec.

#### 3.2 Exam view sequence

| View | <b>2</b> -D | Pulse wave | Continuous wave | Color |
|---|---|---|---|---|
| Parasternal long axis | X | | | AV |
| Parasternal short axis | Χ | AV | | AV |
| Apical 4-chamber | Х | | | |
| Apical 5-chamber | X | LVOT | AV | LVOT / AV |
| Apical 2-chamber | Х | | | |
| Apical 3-chamber | X | AV | AV | LVOT / AV |

#### 3.3 Data collection

The clinical site is to provide the following data for each TTE:



Clinical Study Number: 2010-03

- Study subject identification number
- Heart rate (bpm)
- Height (cm)
- Weight (kg)
- Cardiac rhythm

Data from TTE exams is to include the following measurements/calculations by a Core Lab:

- Aortic bioprosthesis assessment
  - Flow velocities and gradients
    - Mean gradient
    - Peak gradient
    - Effective orifice area
    - Time velocity integral left ventricular outflow tract
    - Time velocity integral aortic valve
    - Maximum velocity aortic valve
    - Maximum velocity left ventricular outflow tract
  - Aortic insufficiency
    - Central leak grade
    - Paravalvular / perivalvular leak grade
  - Aortic stenosis grade
- Left ventricle measurements
  - Dimension
    - Left ventricle end-systolic
    - Left ventricle end-diastolic
    - Septal wall thickness (end-diastolic)
    - Posterior wall thickness (end-diastolic)
  - Volume
    - Left ventricle end-systolic
    - Left ventricle end-diastolic
  - o Ejection fraction
- Calculated cardiac performance parameters
  - o Cardiac Output
  - Stroke Volume



Clinical Study Number: 2010-03

#### 4 Transesophageal echocardiogram (TEE)

#### 4.1 Performing the exam

Study subjects are typically examined within 1 hour after aortic valve replacement with the study device (after the aortic cross clamp is removed).

#### 4.2 Exam view

The exact position of the TEE probe may vary from patient to patient, but should be aligned at the level of the aortic annulus.

Doppler requirements in this view:

- Continuous wave through the aortic valve
- Color of AV

#### 4.3 Data collection

The clinical site is to provide the following data for each TEE:

- Study subject identification number
- Heart rate (bpm)
- Height (cm)
- Weight (kg)
- Cardiac rhythm

Data from TEE exams is to include the following measurements/calculations by a Core Lab:

- Aortic bioprosthesis assessment
  - Aortic insufficiency
    - Central leak grade
    - Paravalvular / perivalvular leak grade

#### 5 Abbreviated transthoracic echocardiogram (aTTE)

#### 5.1 Performing the exam

Study subjects are typically examined in the left lateral decubitus or supine position. This exam may performed while the subject is still in the Operating Room. All views are to be taken with 2 captures, the length of which will vary under the following clinical conditions:

- Sinus rhythm with up to 90bpm: 3 beat capture
- Sinus rhythm with more than 90bpm: 5 beat capture



Clinical Study Number: 2010-03

Frequent atrial or ventricular ectopy: 3 second capture

Atrial fibrillation or atrial flutter: 5 second capture

Paced rhythm: 5 second capture

The sweep speed for all spectral Doppler and M-mode recordings should be 100 mm/sec. Nyquist settings for color Doppler assessment of the aortic valve should be >50 cm/sec.

#### 5.2 Exam view sequence

| View | 2-D | Pulse wave | Continuous wave | Color |
|------------------------|-----|------------|-----------------|-----------|
| Parasternal short axis | X | AV | | AV |
| Apical 4-chamber | Х | | | |
| Apical 3-chamber | X | AV | AV | LVOT / AV |

#### 5.3 Data collection

The clinical site is to provide the following data for each aTTE:

- Study subject identification number
- Heart rate (bpm)
- Height (cm)
- Weight (kg)
- Cardiac rhythm

Data from aTTE exams is to include the following measurements/calculations by a Core Lab:

- Aortic bioprosthesis assessment
  - Aortic insufficiency
    - Central leak grade
    - Paravalvular / perivalvular leak grade
  - Aortic stenosis grade



# 15.7 EQ-5D QUESTIONNAIRE



Kwestionariusz Dotyczący Zdrowia

wesja polska do użytku w Polsce

(Polish version for Poland)

Poprzez zaznaczenie symbolem (☑) jednego kwadratu w każdej grupie podanej poniżej, proszę wybrać zdanie najlepiej określające stan Pana/Pani zdrowia dzisiaj.

| Zdolność poruszania się | |
|---|---|
| Nie mam problemów z chodzeniem | |
| Mam trochę problemów z chodzeniem | |
| Jestem zmuszony/a pozostawać w łóżku | |
| Samoopieka | |
| Nie mam żadnych problemów z samoopieką | |
| Mam trochę problemów z myciem i ubieraniem się | |
| Nie mogę sam/a się umyć ani ubrać | |
| Zwykła działalność (np. praca, nauka, zajęcia domowe, aktywności rodzinne, zajęcia w czasie wolnym) Nie mam problemów z wykonywaniem moich zwykłych czynności Mam trochę problemów z wykonywaniem moich zwykłych czynności Nie mogę wykonywać moich zwykłych czynności | <u> </u> |
| Nie odczuwam bólu ani dyskomfortu | |
| Odczuwam umiarkowany ból lub dyskomfort | |
| Odczuwam krańcowy ból lub dyskomfort | |
| Niepokój/Przygnębienie | |
| Nie jestem niespokojny/a ani przygnębiony/a | |
| Jestem umiarkowanie niespokojny/a lub przygnębiony/a | |
| lestem krańcowo niespokojny/a lub przygnebiony/a | |

Aby umożliwić badanym ocenę jak dobry lub zły jest ich stan zdrowia przygotowaliśmy skalę (podobną do skali termometru), na której najlepszy stan zdrowia jaki można sobie wyobrazić jest oznaczony liczbą 100, a najgorszy stan zdrowia jaki można sobie wyobrazić jest oznaczony jako 0.

Prosimy o wskazanie na skali, jak dobry lub zły jest w państwa opinii stan Pana/Pani zdrowia dzisiaj. Proszę zrobić to rysując linię z kostki poniżej do jakiegokolwiek punktu na skali, określającego jak dobry lub zły jest Pana/Pani dzisiejszy stan zdrowia.

Twój stan zdrowia dzisiaj





# 15.8 SF-12 V2 QUESTIONNAIRE



## STUDY NUMBER 2010-03

QUALITY OF LIFE PAGE 1 OF 3

# CLINICAL STUDY OF THE EDWARDS PERICARDIAL AORTIC BIOPROSTHESIS, **MODEL 11000**

| S | ubject Study ID# | 2 | 0 | 1 | 0 | 0 | 3 | • | | | | | 5 | | | Site# | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| qu<br>mi | QualityMetric's SF-12v2® Health Survey¹ is a shorter version of the SF-36v2® Health Survey that uses just 12 questions to measure functional health and well-being from the subject's point of view. It takes only 2-3 minutes to complete. The SF-12v2 is a practical, reliable, and valid measure of physical and mental health and covers the same eight health domains as the SF-36v2 with one or two questions per domain. | | | | | | | | | | | | | | | | | | |
| VIS | BIT INTERVAL: | | SCR | EENIN | IG □ | ] 1 YI | EAR | | | | | | | | | | | | |
| Da | Date of Assessment: | | | | | | | | | | | | | | | | | | |
| 1. | 1. In general, would you say your health is: | | | | | | | | | | | | | | | | | | |
| | Excellent 1 | Very good Goo | | | | | | | | | | | | | Poor<br>D <sub>5</sub> | | | | |
| 2. | The following questions are about activities you might do during a typical day. Does <u>your health now limit</u> <u>you</u> in these activities? If so, how much? | | | | | | | | | | | | | | | | | | |
| | | | | Ye | Yes, limited a Yes, lim | | | | | | I | | | | | | | | |
| a. | Moderate activit<br>table, pushing a<br>or playing golf. | _ | | | | | | | <b>]</b> , | | | | | | 3 | | | | |
| b. | Climbing <u>several</u> | flight | s of s | tairs. | | | | | <b>]</b> 1 | | | | | □₃ | | | | | |
| 3. | During the <u>past</u><br>other regular da | | | | | | | | _ | | | y of th | he follo | owing | prol | blems w | ith yo | ur wo | rk or |
| | | | | Al | ll of th | | | st of<br>time | | me of | | little of<br>e time | | one o | | | | | |
| | a. Accomplishe would like. | d les | s tha | n you | 1 | | | | <b>]</b> 2 | , | <b>]</b> ₃ | | $\square_4$ | | <b>]</b> 5 | | | | |

<sup>&</sup>lt;sup>1</sup>SF-12v2<sup>3t</sup> Health Survey<sup>6t</sup> 1994, 2002 by QualityMetric incorporated and Medical Outcomes Trust. SF-12<sup>3th</sup> a registered trademark of Medical Outcomes Trust. (SF12v2 Standard, US version 2.0).



# STUDY NUMBER 2010-03

CLINICAL STUDY OF THE EDWARDS PERICARDIAL AORTIC BIOPROSTHESIS, MODEL 11000

| QUALITYO | F | LIF | Б |
|----------|---|-----|---|
| PAGE | 2 | OF | 3 |

| s | ubject Study ID# | 2 | 0 | 1 | 0 | 0 | 3 | - | | | | | | | Site | # | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| b. Were limited in the <u>kind</u> of work or other activities. | | | | | | | | ]2 | | <b>l</b> <sub>3</sub> | | <b>1</b> <sub>4</sub> | | <b>1</b> 5 | | | |
| 4. | other regular da | ily ac | tiviti | es <u>as</u> | a re | | of an | y em<br>Mos | | | blems<br>e of | | h as t<br>le of | eeling<br>Nor | | | |
| | <ul> <li>a. <u>Accomplishe</u><br/>would like.</li> </ul> | u iess | <u>s</u> ulai | ii yot | | | | | ]2 | | <b>1</b> <sub>3</sub> | | 14 | | <b>]</b> 5 | | |
| | b. Did work o | | | <u>les</u> | <u>s</u> | | | | ]2 | | <b>l</b> <sub>3</sub> | | <b>1</b> <sub>4</sub> | | <b>1</b> <sub>5</sub> | | |
| 5. | 5. During the <u>past 4 weeks</u> , how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)? | | | | | | | | | | | | | | | | |
| | Not at all | | ittle b | oit | | | derate | ely | | Quite | | | Ex | treme | У | | |
| 6. | 5. These questions are about how you feel and how things have been with you during the <u>past 4</u> <u>weeks.</u> For each question, please give one answer that comes closest to the way you have been feeling. How much of the time during the <u>past 4 weeks</u> All of the Most of Some of A little of None of | | | | | | | | | | | | | | | | |
| | a. Have you feltopeaceful? | t calm | and | | | time | | | time | the t | | the t | | | time<br>] <sub>5</sub> | | |
| | b. Did you have | a lot | of en | ergy | ? | | | | ]2 | | <b>1</b> <sub>3</sub> | | 14 | | <b>]</b> 5 | | |
| | c. Have you felt | | nhear | ted | | <b>□</b> ₁ | | | ]2 | | 3 | | 1, | | <b>1</b> <sub>5</sub> | | |
| _ | Danis a Alexander | | | | | | - 6 41 | | F | | | | l In a - | 141 | | | <br>I |

7. During the <u>past 4 weeks</u>, how much of the time has your <u>physical health or emotional problems</u> interfered with your social activities (like visiting friends, relatives, etc.)?



# STUDY NUMBER 2010-03

QUALITY OF LIFE PAGE 3 OF 3

# CLINICAL STUDY OF THE EDWARDS PERICARDIAL AORTIC BIOPROSTHESIS, **MODEL 11000**

| Subject Study ID # | 2 | 0 | 1 | 0 | 0 | 3 | - | | | | | | | | Sit | e# | | | | _ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| All of the time | Мо | | | | | ne of time | the | he A little of the time | | | | | None of the time ☐ 5 | | | | | | | |
| I HAVE REVIEWED AND AGREE WITH ALL DATA ENTERED ON THIS FORM | | | | | | | | | | | | | | | | | | | | |
| INVESTIGATOR SIGNATURE | <u> </u> | | | | | | | | DATE | SIGN | IED | D | D | M | M | M | Y | Y | Y | ] |